CLINICAL TRIAL: NCT00805389
Title: Comparison of the Immunogenicity and Safety of Various Investigational and Licensed Formulations of Hepatitis B Surface Antigen (HBsAg) Vaccines.
Brief Title: Study to Compare the Efficacy of GSK Biologicals' Adjuvants in Combination With the Antigen of the Hepatitis B Vaccine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 112115
Record Dates: First submitted 2008-12-05; First posted 2008-12-09 (Estimated); Results first posted 2013-01-25 (Estimated); Last update posted 2018-08-20 (Actual); Status verified 2018-06

CONDITIONS: Hepatitis B
Keywords: Adjuvant Systems; Hepatitis B
MeSH Terms: conditions — Hepatitis B | interventions — Engerix-B; Fendrix; Hepatitis B Surface Antigens; Immunization, Secondary

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (5):
- GSK223192A 1 Group (Experimental): Subjects aged between, and including, 18 and 45 years at the time of first vaccination received 2 doses of GSK223192A vaccine, lot 1, at Days 0 and 30. 2 subsets of subjects within the group - subjects identified with either a pre-defined Human Leukocytes Antigen (HLA) Class I subtype (Subset 1) or a pre-defined HLA Class II subtype (Subset 2) - additionally received 1 booster dose of Hepatitis B surface antigens (HBsAg) at Day 360. The GSK223192A vaccine and HBsAg antigens were administered intramuscularly into the deltoid muscle of the non-dominant arm.
  Interventions: Biological: GSK Biologicals' Hepatitis B vaccines (GSK223192A); Biological: HBsAg (Booster injection)
- GSK223192A 2 Group (Experimental): Subjects aged between, and including, 18 and 45 years at the time of first vaccination received 2 doses of GSK223192A vaccine, lot 2, at Days 0 and 30. 2 subsets of subjects within the group - subjects identified with either a pre-defined Human Leukocytes Antigen (HLA) Class I subtype (Subset 1) or a pre-defined HLA Class II subtype (Subset 2) - additionally received 1 booster dose of Hepatitis B surface antigens (HBsAg) at Day 360. The GSK223192A vaccine and HBsAg antigens were administered intramuscularly into the deltoid muscle of the non-dominant arm.
  Interventions: Biological: GSK Biologicals' Hepatitis B vaccines (GSK223192A); Biological: HBsAg (Booster injection)
- GSK223192A 3 Group (Experimental): Subjects aged between, and including, 18 and 45 years at the time of first vaccination received 2 doses of GSK223192A vaccine, lot 3, at Days 0 and 30. 2 subsets of subjects within the group - subjects identified with either a pre-defined Human Leukocytes Antigen (HLA) Class I subtype (Subset 1) or a pre-defined HLA Class II subtype (Subset 2) - additionally received 1 booster dose of Hepatitis B surface antigens (HBsAg) at Day 360. The GSK223192A vaccine and HBsAg antigens were administered intramuscularly into the deltoid muscle of the non-dominant arm.
  Interventions: Biological: GSK Biologicals' Hepatitis B vaccines (GSK223192A); Biological: HBsAg (Booster injection)
- Fendrix Group (Experimental): Subjects aged between, and including, 18 and 45 years at the time of first vaccination received 2 doses of Fendrix™ vaccine at Days 0 and 30. 2 subsets of subjects within the group - subjects identified with either a pre-defined Human Leukocytes Antigen (HLA) Class I subtype (Subset 1) or a pre-defined HLA Class II subtype (Subset 2) - additionally received 1 booster dose of Hepatitis B surface antigens (HBsAg) at Day 360. The Fendrix™ vaccine and HBsAg antigens were administered intramuscularly into the deltoid muscle of the non-dominant arm.
  Interventions: Biological: Fendrix™; Biological: HBsAg (Booster injection)
- Engerix-B Group (Active Comparator): Subjects aged between, and including, 18 and 45 years at the time of first vaccination received 2 doses of Engerix-B™ vaccine at Days 0 and 30. 2 subsets of subjects within the group - subjects identified with either a pre-defined Human Leukocytes Antigen (HLA) Class I subtype (Subset 1) or a pre-defined HLA Class II subtype (Subset 2) - additionally received 1 booster dose of Hepatitis B surface antigens (HBsAg) at Day 360. The Engerix-B™ vaccine and HBsAg antigens were administered intramuscularly into the deltoid muscle of the non-dominant arm.
  Interventions: Biological: Engerix-B™; Biological: HBsAg (Booster injection)

INTERVENTIONS:
Biological: Engerix-B™ — 2 doses intramuscular injections
  Arms: Engerix-B Group
Biological: Fendrix™ — 2 doses intramuscular injections
  Arms: Fendrix Group
Biological: GSK Biologicals' Hepatitis B vaccines (GSK223192A) — 2 doses intramuscular injections 3 different formulations of (GSK223192A), each administered to 1 group
  Arms: GSK223192A 1 Group; GSK223192A 2 Group; GSK223192A 3 Group
Biological: HBsAg (Booster injection) — Single dose intramuscular injection

SUMMARY:
The aim of this Observer-blind study is to compare different Adjuvant Systems with the same, well-known antigen (HBsAg) already used in the GSK marketed vaccines against Hepatitis B (Engerix-BTM and FendrixTM), in order to better understand the immune response induced by each of the Adjuvant System.

This Protocol Posting has been updated following Protocol amendment 6, October 2009. The section impacted is Eligibility Criteria

ELIGIBILITY:
Inclusion Criteria:

All subjects must satisfy the following criteria at study entry :

* Subjects who the investigator believes that they can and will comply with the requirements of the protocol.
* A male or female between, and including, 18 and 45 years at the time of the first vaccination.
* Written informed consent obtained from the subject.
* Healthy subjects as established by medical history, clinical examination and clinical laboratory assessment before entering into the study.
* If the subject is female, she must be of non-childbearing potential, or if she is of childbearing potential, she must practice adequate contraception for 30 days prior to vaccination, have a negative pregnancy test and continue such precautions for 2 months after completion of the vaccination series.

Exclusion criteria:

The following criteria should be checked at the time of study entry. If any apply, the subject must not be included in the study:

* Previous vaccination against Hepatitis B.
* Positive for anti-HBs antibodies, antiHBc antibodies, HBsAg, HCV antibodies and/or HIV.
* Any previous administration of specific adjuvant components.
* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period or participation to another pharmaceutical/vaccine study.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose.
* Planned administration/ administration of a vaccine not foreseen by the study protocol within 30 days of the first dose of vaccine with the exception of the influenza vaccine (pandemic or seasonal) which can be administered > 21 days preceding or > 21 days following each primary vaccine dose (Doses 1 and 2) AND > 7 days preceding or > 7 days following the booster dose.
* Administration of immunoglobulins and/or any blood products within the last 3 months.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine(s).
* Current serious neurologic or mental disease.
* Any past or current malignancies and lymphoproliferative disorders.
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic, renal functional abnormality, autoimmune disease or anemia, as determined by physical examination or laboratory screening tests at the discretion of the investigator.
* Acute disease at the time of enrolment.
* Pregnant or lactating female.
* History of chronic alcohol consumption and/or drug abuse.
* Other conditions that the principal investigator judges may interfere with study findings.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 713 (Actual)
Dates: Start 2008-12-15 (Actual); Primary Completion 2010-09-29 (Actual); Study Completion 2011-07-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (12):
- Belgium (4):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, La Louvière
  - GSK Investigational Site, Wilrijk
- Germany (8):
  - GSK Investigational Site, Tübingen, Baden-Wurttemberg
  - GSK Investigational Site, Haag, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Regensburg, Bavaria
  - GSK Investigational Site, Würzburg, Bavaria
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Tasdighian S, Bechtold V, Essaghir A, Saeys Y, Burny W. An innate immune signature induced by AS01- or AS03-adjuvanted vaccines predicts the antibody response magnitude and quality consistently over time. Front Immunol. 2024 Aug 14;15:1412732. doi: 10.3389/fimmu.2024.1412732. eCollection 2024. PMID 39206189
- [Derived] Moris P, Bellanger A, Ofori-Anyinam O, Jongert E, Yarzabal Rodriguez JP, Janssens M. Whole blood can be used as an alternative to isolated peripheral blood mononuclear cells to measure in vitro specific T-cell responses in human samples. J Immunol Methods. 2021 May;492:112940. doi: 10.1016/j.jim.2020.112940. Epub 2021 Jan 23. PMID 33493551
- [Derived] De Mot L, Bechtold V, Bol V, Callegaro A, Coccia M, Essaghir A, Hasdemir D, Ulloa-Montoya F, Siena E, Smilde A, van den Berg RA, Didierlaurent AM, Burny W, van der Most RG. Transcriptional profiles of adjuvanted hepatitis B vaccines display variable interindividual homogeneity but a shared core signature. Sci Transl Med. 2020 Nov 11;12(569):eaay8618. doi: 10.1126/scitranslmed.aay8618. PMID 33177181
- [Derived] Hasdemir D, van den Berg RA, van Kampen A, Smilde AK. Modeling adaptive response profiles in a vaccine clinical trial. BMC Med Res Methodol. 2020 Jul 16;20(1):191. doi: 10.1186/s12874-020-01070-3. PMID 32677968
- [Derived] Burny W, Marchant A, Herve C, Callegaro A, Caubet M, Fissette L, Gheyle L, Legrand C, Ndour C, Tavares Da Silva F, van der Most R, Willems F, Didierlaurent AM, Yarzabal J; ECR-008 study group. Inflammatory parameters associated with systemic reactogenicity following vaccination with adjuvanted hepatitis B vaccines in humans. Vaccine. 2019 Mar 28;37(14):2004-2015. doi: 10.1016/j.vaccine.2019.02.015. Epub 2019 Mar 5. PMID 30850240
- [Derived] Burny W, Callegaro A, Bechtold V, Clement F, Delhaye S, Fissette L, Janssens M, Leroux-Roels G, Marchant A, van den Berg RA, Garcon N, van der Most R, Didierlaurent AM; ECR-002 Study Group. Different Adjuvants Induce Common Innate Pathways That Are Associated with Enhanced Adaptive Responses against a Model Antigen in Humans. Front Immunol. 2017 Aug 14;8:943. doi: 10.3389/fimmu.2017.00943. eCollection 2017. PMID 28855902
- See also: IPD for this study will be made available via the Clinical Study Data Request site. — https://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Approximately 75 subjects in each group, approximately 23 and 52 subjects/group identified with a pre-defined Human Leukocytes Antigen (HLA) Class I and II subtypes [Subset 1 and 2, respectively], received a booster dose of HBsAg at Day 360.
Pre-assignment Details: Study duration was of 390 days for subjects in Subsets 1 and 2 (subjects identified with a pre-defined Human Leukocytes Antigen (HLA) Class I subtype (Subset 1) or a pre-defined HLA Class II subtype (Subset 2) vaccinated with an additional dose of Hepatitis B surface antigens (HBsAg)) and of 360 days for subjects not receiving this dose of HBsAg.
Period: Overall Study
Arm/Group | GSK223192A 1 Group | GSK223192A 2 Group | GSK223192A 3 Group | Fendrix Group | Engerix-B Group
Started | 143 | 142 | 141 | 145 | 142
Completed | 136 | 137 | 129 | 128 | 129
Not Completed | 7 | 5 | 12 | 17 | 13
Not completed — Adverse Event | 0 | 0 | 1 | 2 | 0
Not completed — Lost to Follow-up | 4 | 3 | 6 | 10 | 9
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 2 | 4 | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK223192A 1 Group | GSK223192A 2 Group | GSK223192A 3 Group | Fendrix Group | Engerix-B Group | Total
Number analyzed (Participants) | 143 | 142 | 141 | 145 | 142 | 713
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.7 (6.94) | 33.7 (7.28) | 32.9 (7.58) | 33.5 (7.41) | 32.9 (7.50) | 33.5 (7.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 66 | 64 | 66 | 65 | 327
  Male | 77 | 76 | 77 | 79 | 77 | 386
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — White - Caucasian / European heritage
  Participants
    White - Caucasian / European heritage | 135 | 138 | 138 | 142 | 136 | 689

OUTCOME MEASURES:

1. Primary Outcome: Number of Hepatitis B (HB)-Specific Cluster of Differentiation 4 (CD4+) T Cells .
Description: The number of HB-CD4+ T cells (per million cells) producing 2 or more markers amongst Cluster Differentiation 40 Ligand (CD40L), Interleukin (IL)-2, Interferon-gamma (IFN-g), Tumor Necrosis Factor-alpha (TNF-a), IL-13 and IL-17 was measured by Intracellular Cytokine Staining (ICS), using frozen Peripheral Blood Mononuclear Cells (PBMCs). Results for the Day 44 time point are the primary results among the outcome measure results presented.
Time Frame: At Day 44
Population: Analyses were performed on the According-to-Protocol (ATP) cohort for adaptive immunogenicity up to Day 60, which included all evaluable subjects who complied with the vaccination schedule and for whom T cell, antibody and memory B cell response data were available for at least one amongst the Day 44 time point.
Measure: Median (Inter-Quartile Range); unit: HB-CD4+ T cells (per million cells)
Arm/Group | GSK223192A 1 Group | GSK223192A 2 Group | GSK223192A 3 Group | Fendrix Group | Engerix-B Group
Number analyzed (Participants) | 114 | 112 | 109 | 112 | 107
HB-CD4+ T cells (per million cells) | 1345 [626 to 3100] | 1257 [540 to 2168] | 647 [436 to 1284] | 391 [242 to 557] | 299 [202 to 486]

2. Secondary Outcome: Number of Hepatitis B (HB)-Specific Cluster of Differentiation 4 (CD4+) T Cells
Description: The number of HB-CD4+ T cells (per million cells) producing 2 or more markers amongst Cluster Differentiation 40 Ligand (CD-40L), Interleukin(IL)-2, Interferon-gamma (IFN-g), Tumor Necrosis Factor-alpha (TNF-a), IL-13 and IL-17 was measured by Intracellular Cytokine Staining (ICS), using frozen Peripheral Blood Mononuclear Cells (PBMCs).
Time Frame: At Days 0, 14, 30 and 60
Population: Analyses were performed on the According-to-Protocol (ATP) cohort for adaptive immunogenicity up to Day 60, which included all evaluable subjects who complied with the vaccination schedule and for whom T cell, antibody and memory B cell response data were available for at least one amongst the Day 0, 14, 30 or 60 time points.
Measure: Median (Inter-Quartile Range); unit: HB-CD4+ T cells (per million cells)
Arm/Group | GSK223192A 1 Group | GSK223192A 2 Group | GSK223192A 3 Group | Fendrix Group | Engerix-B Group
Number analyzed (Participants) | 114 | 112 | 109 | 112 | 107
HB-CD4+ T cells (per million cells)
  HB-CD4+, at Day 0: number analyzed (Participants) | 111 | 110 | 107 | 109 | 106
  HB-CD4+, at Day 0 | 228 [163 to 332] | 230 [166 to 326] | 234 [171 to 312] | 234 [172 to 362] | 235 [176 to 353]
  HB-CD4+, at Day 14: number analyzed (Participants) | 114 | 110 | 106 | 112 | 107
  HB-CD4+, at Day 14 | 408 [225 to 656] | 447 [248 to 752] | 460 [309 to 819] | 289 [208 to 434] | 245 [173 to 412]
  HB-CD4+, at Day 30: number analyzed (Participants) | 108 | 107 | 109 | 109 | 101
  HB-CD4+, at Day 30 | 277 [190 to 430] | 333 [233 to 482] | 314 [249 to 496] | 255 [189 to 362] | 249 [178 to 376]
  HB-CD4+, at Day 60: number analyzed (Participants) | 108 | 112 | 108 | 112 | 104
  HB-CD4+, at Day 60 | 965 [560 to 1925] | 958 [450 to 1777] | 587 [360 to 1031] | 393 [250 to 582] | 308 [201 to 555]

3. Secondary Outcome: Number of Hepatitis B (HB) - Specific Cluster of Differentiation 8 (CD8+) T Cells.
Description: The number of HB-CD8+ T cells (per million cells) producing 2 or more markers amongst Cluster Differentiation 40 Ligand (CD40L), Interleukin (IL)-2, Interferon-gamma (IFN-g), Tumor Necrosis Factor-alpha (TNF-a), IL-13 and IL-17 was measured by Intracellular Cytokine Staining (ICS), using frozen Peripheral Blood Mononuclear Cells (PBMCs).
Time Frame: At Days 0, 14, 30, 44, and 60
Population: Analysis was done on the According-to-Protocol (ATP) cohort for adaptive immunogenicity to Day 60, which included all evaluable subjects for whom T cell, antibody and memory B cell response data were available for at least one amongst the Day 0, 14, 30, 44, or 60 time points.
Measure: Median (Inter-Quartile Range); unit: HB-CD8+ T cells (per million cells)
Arm/Group | GSK223192A 1 Group | GSK223192A 2 Group | GSK223192A 3 Group | Fendrix Group | Engerix-B Group
Number analyzed (Participants) | 112 | 112 | 107 | 109 | 105
HB-CD8+ T cells (per million cells)
  HB-CD8+, at Day 0: number analyzed (Participants) | 107 | 108 | 105 | 104 | 104
  HB-CD8+, at Day 0 | 176 [107 to 286] | 174 [112 to 312] | 172 [123 to 236] | 201 [109 to 300] | 184 [108 to 236]
  HB-CD8+, at Day 14: number analyzed (Participants) | 112 | 110 | 104 | 108 | 105
  HB-CD8+, at Day 14 | 174 [121 to 290] | 160 [106 to 273] | 174 [121 to 234] | 193 [129 to 296] | 177 [129 to 274]
  HB-CD8+, at Day 30: number analyzed (Participants) | 105 | 103 | 107 | 107 | 100
  HB-CD8+, at Day 30 | 185 [109 to 276] | 173 [118 to 255] | 160 [113 to 248] | 191 [132 to 254] | 173 [133 to 259]
  HB-CD8+, at Day 44: number analyzed (Participants) | 107 | 106 | 102 | 105 | 98
  HB-CD8+, at Day 44 | 212 [129 to 300] | 213 [148 to 338] | 177 [116 to 272] | 157 [106 to 274] | 169 [118 to 246]
  HB-CD8+, at Day 60: number analyzed (Participants) | 108 | 112 | 107 | 109 | 104
  HB-CD8+, at Day 60 | 209 [129 to 308] | 228 [144 to 339] | 171 [123 to 281] | 184 [115 to 298] | 166 [124 to 266]

4. Secondary Outcome: Number of HB Specific CD4+ T Cells .
Description: as for outcome 2
Time Frame: At Days 0, 180 and 360
Population: Analysis was done on the According-to-Protocol (ATP) cohort for persistence which included all subjects from the ATP cohort for adaptive immunogenicity up to Day 60 for whom adaptive immunogenicity data were available for at least one post-vaccination time point (Day 180 or Day 360).
Measure: Median (Inter-Quartile Range); unit: HB-CD4+ T cells (per million cells)
Arm/Group | GSK223192A 1 Group | GSK223192A 2 Group | GSK223192A 3 Group | Fendrix Group | Engerix-B Group
Number analyzed (Participants) | 108 | 107 | 101 | 106 | 101
HB-CD4+ T cells (per million cells)
  HB-CD4+, at Day 0: number analyzed (Participants) | 106 | 102 | 98 | 99 | 97
  HB-CD4+, at Day 0 | 230 [163 to 333] | 231 [166 to 331] | 248 [179 to 313] | 223 [171 to 348] | 240 [172 to 347]
  HB-CD4+, at Day 180: number analyzed (Participants) | 104 | 107 | 97 | 106 | 101
  HB-CD4+, at Day 180 | 1090 [573 to 1827] | 954 [508 to 1504] | 546 [382 to 911] | 360 [259 to 666] | 334 [256 to 493]
  HB-CD4+, at Day 360: number analyzed (Participants) | 108 | 105 | 101 | 100 | 95
  HB-CD4+, at Day 360 | 960 [564 to 1566] | 829 [388 to 1509] | 564 [340 to 887] | 388 [217 to 627] | 350 [246 to 499]

5. Secondary Outcome: Number of HB - Specific CD8+ T Cells.
Description: The number of HB-CD8+ T cells (per million cells) producing 2 or more markers amongst Cluster Differentiation 40 Ligand (CD-40L), Interleukin(IL)-2, Interferon-gamma (IFN-g), Tumor Necrosis Factor-alpha (TNF-a), IL-13 and IL-17 was measured by Intracellular Cytokine Staining (ICS), using frozen Peripheral Blood Mononuclear Cells (PBMCs).
Time Frame: At Days 0, 180 and 360
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: HB-CD8+ T cells (per million cells)
Arm/Group | GSK223192A 1 Group | GSK223192A 2 Group | GSK223192A 3 Group | Fendrix Group | Engerix-B Group
Number analyzed (Participants) | 108 | 107 | 99 | 105 | 101
HB-CD8+ T cells (per million cells)
  HB-CD8+, at Day 0: number analyzed (Participants) | 102 | 100 | 96 | 96 | 95
  HB-CD8+, at Day 0 | 175 [107 to 284] | 169 [110 to 312] | 176 [125 to 261] | 191 [107 to 286] | 184 [107 to 237]
  HB-CD8+, at Day 180: number analyzed (Participants) | 104 | 107 | 96 | 105 | 101
  HB-CD8+, at Day 180 | 120 [81 to 170] | 124 [81 to 187] | 92 [57 to 133] | 102 [57 to 153] | 110 [64 to 171]
  HB-CD8+, at Day 360: number analyzed (Participants) | 108 | 104 | 99 | 98 | 94
  HB-CD8+, at Day 360 | 114 [57 to 163] | 115 [57 to 163] | 112 [78 to 160] | 104 [57 to 154] | 90 [57 to 159]

6. Secondary Outcome: Number of HB - Specific CD4+ T Cells.
Description: as for outcome 2
Time Frame: At Days 0, 360 and 374
Population: Analysis was done on the Booster According-to-Protocol (ATP) cohort for immunogenicity which included all subjects from subsets 1 and 2 who received a booster vaccination at Day 360 for whom adaptive immunogenicity data were available for at least one post-booster time point.
Measure: Median (Inter-Quartile Range); unit: HB-CD4+ T cells (per million cells)
Arm/Group | GSK223192A 1 Group | GSK223192A 2 Group | GSK223192A 3 Group | Fendrix Group | Engerix-B Group
Number analyzed (Participants) | 54 | 51 | 53 | 52 | 48
HB-CD4+ T cells (per million cells)
  HB-CD4+, at Day 0 | 228 [175 to 346] | 233 [172 to 307] | 254 [177 to 347] | 234 [183 to 293] | 266 [194 to 362]
  HB-CD4+, at Day 360 | 1029 [601 to 1781] | 770 [388 to 1511] | 538 [301 to 974] | 300 [199 to 590] | 360 [273 to 506]
  HB-CD4+, at Day 374: number analyzed (Participants) | 50 | 48 | 49 | 52 | 48
  HB-CD4+, at Day 374 | 1006 [725 to 1907] | 1037 [580 to 1882] | 688 [456 to 1129] | 401 [250 to 750] | 353 [271 to 599]

7. Secondary Outcome: Number of HB - Specific CD8+ T Cells
Description: as for outcome 5
Time Frame: At Days 0, 360 and 374
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: HB-CD8+ T cells (per million cells)
Arm/Group | GSK223192A 1 Group | GSK223192A 2 Group | GSK223192A 3 Group | Fendrix Group | Engerix-B Group
Number analyzed (Participants) | 54 | 51 | 51 | 52 | 48
HB-CD8+ T cells (per million cells)
  HB-CD8+, at Day 0: number analyzed (Participants) | 51 | 45 | 49 | 46 | 42
  HB-CD8+, at Day 0 | 187 [111 to 304] | 161 [100 to 256] | 196 [138 to 271] | 244 [120 to 316] | 168 [125 to 234]
  HB-CD8+, at Day 360: number analyzed (Participants) | 54 | 51 | 51 | 50 | 47
  HB-CD8+, at Day 360 | 109 [57 to 151] | 118 [57 to 161] | 121 [77 to 183] | 99 [57 to 130] | 90 [57 to 169]
  HB-CD8+, at Day 374: number analyzed (Participants) | 50 | 48 | 49 | 52 | 48
  HB-CD8+, at Day 374 | 107 [57 to 133] | 111 [57 to 166] | 122 [57 to 174] | 121 [75 to 185] | 111 [85 to 212]

8. Secondary Outcome: Number of HB - Specific CD4+ T Cells
Description: The number of HB-CD4+ T cells (per million cells) producing 2 or more markers amongst Cluster Differentiation 40 Ligand (CD-40L), Interleukin(IL)-2, Interferon-gamma (IFN-g), and Tumor Necrosis Factor-alpha (TNF-a) was measured by Intracellular Cytokine Staining (ICS), using whole blood. This analysis was performed solely on eligible subjects enrolled at the Centre for Vaccinology (CEVAC) in Ghent, Belgium.
Time Frame: At Days 0, 14, 30, 33, 37, 44 and 60
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: HB-CD4+ T cells (per million cells)
Arm/Group | GSK223192A 1 Group | GSK223192A 2 Group | GSK223192A 3 Group | Fendrix Group | Engerix-B Group
Number analyzed (Participants) | 17 | 14 | 15 | 19 | 14
HB-CD4+ T cells (per million cells)
  HB-CD4+, at Day 0: number analyzed (Participants) | 13 | 11 | 13 | 16 | 12
  HB-CD4+, at Day 0 | 68 [11 to 104] | 98 [11 to 159] | 25 [11 to 144] | 48 [11 to 106] | 31 [11 to 94]
  HB-CD4+, at Day 14: number analyzed (Participants) | 16 | 14 | 10 | 19 | 11
  HB-CD4+, at Day 14 | 425 [199 to 687] | 498 [184 to 1204] | 149 [71 to 503] | 75 [11 to 125] | 85 [46 to 139]
  HB-CD4+, at Day 30: number analyzed (Participants) | 15 | 14 | 13 | 17 | 14
  HB-CD4+, at Day 30 | 313 [161 to 424] | 314 [170 to 562] | 243 [87 to 344] | 67 [20 to 102] | 110 [47 to 172]
  HB-CD4+, at Day 33: number analyzed (Participants) | 16 | 12 | 13 | 15 | 13
  HB-CD4+, at Day 33 | 114 [80 to 242] | 270 [160 to 445] | 110 [54 to 188] | 63 [14 to 91] | 126 [37 to 166]
  HB-CD4+, at Day 37: number analyzed (Participants) | 17 | 13 | 14 | 19 | 14
  HB-CD4+, at Day 37 | 844 [598 to 1679] | 869 [473 to 3559] | 486 [223 to 1740] | 67 [32 to 178] | 174 [119 to 271]
  HB-CD4+, at Day 44: number analyzed (Participants) | 14 | 13 | 14 | 17 | 12
  HB-CD4+, at Day 44 | 2021 [1187 to 3686] | 2890 [1232 to 4337] | 1253 [647 to 2197] | 271 [95 to 515] | 265 [127 to 716]
  HB-CD4+, at Day 60: number analyzed (Participants) | 11 | 12 | 15 | 16 | 14
  HB-CD4+, at Day 60 | 1291 [396 to 2265] | 1477 [763 to 3920] | 768 [317 to 1458] | 200 [110 to 459] | 247 [107 to 398]

9. Secondary Outcome: Number of HB - Specific CD8+ T Cells
Description: The number of HB-CD8+ T cells (per million cells) producing 2 or more markers amongst Cluster Differentiation 40 Ligand (CD-40L), Interleukin(IL)-2, Interferon-gamma (IFN-g), and Tumor Necrosis Factor-alpha (TNF-a) was measured by Intracellular Cytokine Staining (ICS), using whole blood. This analysis was performed solely on eligible subjects enrolled at the Centre for Vaccinology (CEVAC) in Ghent, Belgium.
Time Frame: At Days 0, 14, 30, 44, 60 and 180
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: HB-CD8+ T cells (per million cells)
Arm/Group | GSK223192A 1 Group | GSK223192A 2 Group | GSK223192A 3 Group | Fendrix Group | Engerix-B Group
Number analyzed (Participants) | 16 | 13 | 16 | 15 | 14
HB-CD8+ T cells (per million cells)
  HB-CD4+, at Day 0: number analyzed (Participants) | 13 | 10 | 13 | 14 | 11
  HB-CD4+, at Day 0 | 11 [11 to 11] | 11 [11 to 64] | 11 [11 to 11] | 11 [11 to 40] | 11 [11 to 11]
  HB-CD4+, at Day 14: number analyzed (Participants) | 13 | 10 | 10 | 15 | 11
  HB-CD4+, at Day 14 | 12 [11 to 91] | 11 [11 to 123] | 11 [11 to 67] | 11 [11 to 121] | 11 [11 to 205]
  HB-CD4+, at Day 30: number analyzed (Participants) | 14 | 12 | 13 | 15 | 14
  HB-CD4+, at Day 30 | 64 [11 to 100] | 11 [11 to 11] | 11 [11 to 68] | 11 [11 to 52] | 11 [11 to 92]
  HB-CD4+, at Day 33: number analyzed (Participants) | 16 | 12 | 10 | 12 | 13
  HB-CD4+, at Day 33 | 11 [11 to 106] | 11 [11 to 68] | 41 [11 to 82] | 11 [11 to 11] | 11 [11 to 68]
  HB-CD4+, at Day 37: number analyzed (Participants) | 16 | 13 | 14 | 15 | 14
  HB-CD4+, at Day 37 | 11 [11 to 108] | 103 [11 to 207] | 11 [11 to 84] | 11 [11 to 11] | 42 [11 to 98]
  HB-CD4+, at Day 44: number analyzed (Participants) | 13 | 13 | 13 | 14 | 11
  HB-CD4+, at Day 44 | 11 [11 to 97] | 99 [11 to 184] | 11 [11 to 130] | 11 [11 to 89] | 11 [11 to 178]
  HB-CD4+, at Day 60: number analyzed (Participants) | 11 | 9 | 16 | 13 | 13
  HB-CD4+, at Day 60 | 37 [11 to 109] | 102 [11 to 229] | 11 [11 to 73] | 11 [11 to 64] | 11 [11 to 69]

10. Secondary Outcome: Number of Hepatitis B (HB)-Specific Cluster of Differentiation 4 (CD4+) T Cells Expressing T Helper Cell Type 1 Response/T Helper Cell Type 2 Response (Th1/Th2) Cytokine Profile
Description: The number of HB-specific CD4+ T cells (per million cells) expressing Th1 and/or Th2 cytokine profile was measured by Intracellular Cytokine Staining (ICS), using frozen Peripheral Blood Mononuclear Cells (PBMCs).
Time Frame: At Days 0, 14, 30, 44 and 60
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: HB-CD4+ T cells (per million cells)
Arm/Group | GSK223192A 1 Group | GSK223192A 2 Group | GSK223192A 3 Group | Fendrix Group | Engerix-B Group
Number analyzed (Participants) | 114 | 112 | 109 | 112 | 107
HB-CD4+ T cells (per million cells)
  HB-CD4+, Th1, at Day 0: number analyzed (Participants) | 111 | 110 | 107 | 109 | 106
  HB-CD4+, Th1, at Day 0 | 65 [38 to 113] | 62 [40 to 111] | 53 [29 to 101] | 70 [41 to 117] | 67 [38 to 119]
  HB-CD4+, Th1, at Day 14: number analyzed (Participants) | 114 | 110 | 106 | 112 | 107
  HB-CD4+, Th1, at Day 14 | 64 [40 to 103] | 75 [44 to 124] | 68 [40 to 102] | 81 [48 to 132] | 66 [38 to 102]
  HB-CD4+, Th1, at Day 30: number analyzed (Participants) | 108 | 107 | 109 | 109 | 101
  HB-CD4+, Th1, at Day 30 | 61 [36 to 91] | 66 [42 to 109] | 75 [45 to 120] | 64 [35 to 113] | 72 [40 to 119]
  HB-CD4+, Th1, at Day 44: number analyzed (Participants) | 112 | 109 | 103 | 108 | 101
  HB-CD4+, Th1, at Day 44 | 155 [78 to 382] | 174 [72 to 354] | 95 [46 to 184] | 74 [46 to 140] | 64 [40 to 115]
  HB-CD4+, Th1, at Day 60: number analyzed (Participants) | 108 | 112 | 108 | 112 | 104
  HB-CD4+, Th1, at Day 60 | 119 [63 to 244] | 141 [71 to 270] | 90 [53 to 146] | 94 [52 to 144] | 61 [40 to 129]
  HB-CD4+, Th2, at Day 0: number analyzed (Participants) | 111 | 110 | 107 | 109 | 106
  HB-CD4+, Th2, at Day 0 | 50 [26 to 95] | 63 [35 to 119] | 55 [17 to 102] | 53 [27 to 118] | 52 [28 to 100]
  HB-CD4+, Th2, at Day 14: number analyzed (Participants) | 114 | 110 | 106 | 112 | 107
  HB-CD4+, Th2, at Day 14 | 52 [28 to 99] | 58 [29 to 124] | 60 [28 to 105] | 42 [21 to 90] | 57 [28 to 125]
  HB-CD4+, Th2, at Day 30: number analyzed (Participants) | 108 | 107 | 109 | 109 | 101
  HB-CD4+, Th2, at Day 30 | 39 [16 to 91] | 52 [28 to 96] | 56 [25 to 100] | 45 [25 to 95] | 47 [28 to 92]
  HB-CD4+, Th2, at Day 44: number analyzed (Participants) | 112 | 109 | 103 | 108 | 101
  HB-CD4+, Th2, at Day 44 | 85 [33 to 133] | 77 [34 to 158] | 87 [37 to 155] | 55 [29 to 109] | 74 [29 to 141]
  HB-CD4+, Th2, at Day 60: number analyzed (Participants) | 108 | 112 | 108 | 112 | 104
  HB-CD4+, Th2, at Day 60 | 78 [41 to 125] | 58 [29 to 127] | 71 [38 to 127] | 53 [29 to 123] | 59 [28 to 153]

11. Secondary Outcome: Number of HB Specific Cluster of Differentiation 4 (CD4+) T Cells Expressing Th1/Th2 Cytokine Profile
Description: as for outcome 10
Time Frame: At Days 0 and 180
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: HB-CD4+ T cells (per million cells)
Arm/Group | GSK223192A 1 Group | GSK223192A 2 Group | GSK223192A 3 Group | Fendrix Group | Engerix-B Group
Number analyzed (Participants) | 106 | 107 | 98 | 106 | 101
HB-CD4+ T cells (per million cells)
  HB-CD4+, Th1, at Day 0: number analyzed (Participants) | 106 | 102 | 98 | 99 | 97
  HB-CD4+, Th1, at Day 0 | 66 [40 to 106] | 63 [44 to 123] | 53 [29 to 101] | 65 [41 to 114] | 64 [38 to 117]
  HB-CD4+, Th1, at Day 180: number analyzed (Participants) | 104 | 107 | 97 | 106 | 101
  HB-CD4+, Th1, at Day 180 | 129 [71 to 215] | 137 [73 to 244] | 76 [49 to 129] | 68 [40 to 122] | 70 [40 to 108]
  HB-CD4+, Th2, at Day 0: number analyzed (Participants) | 106 | 102 | 98 | 99 | 97
  HB-CD4+, Th2, at Day 0 | 51 [27 to 95] | 64 [35 to 119] | 57 [25 to 105] | 50 [27 to 102] | 48 [28 to 100]
  HB-CD4+, Th2, at Day 180: number analyzed (Participants) | 104 | 107 | 97 | 106 | 101
  HB-CD4+, Th2, at Day 180 | 54 [20 to 106] | 63 [28 to 106] | 46 [20 to 85] | 54 [31 to 101] | 49 [16 to 96]

12. Secondary Outcome: Anti-Hepatitis B (Anti-HB) Antibody Concentrations in Serum, as Measured by Chemi Luminescence Immuno Assay (CLIA)
Description: Anti-HBs antibody concentrations in serum were measured by CLIA Assay. Concentrations were presented as geometric mean concentrations, in milli-International Units per milliliter (mIU/mL). Analysis was initially planned to be performed by Enzyme-Linked Immunosorbent Assay (ELISA). A decrease in the specificity of the anti-HB ELISA assay had been observed in some studies for low levels of antibody (10-100 mIU/mL). Following these laboratory quality issues, GSB Biologicals decided to stop testing with the HBs in-house ELISA and to have the anti-HB analysis performed using the new validated CLIA assay. This outcome measure concerns solely subjects part of the HLA Subsets 1 & 2 who received the Day 360 booster dose of HBsAg.
Time Frame: At Days 0, 30, 44, and 60
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Groups:
- GSK223192A 1 - HLA Subsets Group: This group consisted in the subset of subjects in the GSK223192A 1 Group identified with a pre-defined Human Leukocytes Antigen (HLA) Class I or II subtype aged between, and including, 18 and 45 years at the time of first vaccination received 2 doses of GSK223192A vaccine, lot 1, at Days 0 and 30, followed by one booster dose of Hepatitis B surface antigens (HBsAg) at Day 360. The GSK223192A vaccine and HBsAg antigens were administered intramuscularly into the deltoid muscle of the non-dominant arm.
- GSK223192A 2 - HLA Subsets Group: This group consisted in the subset of subjects in the GSK223192A 2 Group identified with a pre-defined Human Leukocytes Antigen (HLA) Class II subtype aged between, and including, 18 and 45 years at the time of first vaccination received 2 doses of GSK223192A vaccine, lot 2, at Days 0 and 30, followed by one booster dose of Hepatitis B surface antigens (HBsAg) at Day 360. The GSK223192A vaccine and HBsAg antigens were administered intramuscularly into the deltoid muscle of the non-dominant arm.
- GSK223192A 3 - HLA Subsets Group: This group consisted in the subset of subjects in the GSK223192A 3 Group identified with a pre-defined Human Leukocytes Antigen (HLA) Class I or II subtype aged between, and including, 18 and 45 years at the time of first vaccination received 2 doses of GSK223192A vaccine, lot 3, at Days 0 and 30, followed by one booster dose of Hepatitis B surface antigens (HBsAg) at Day 360. The GSK223192A vaccine and HBsAg antigens were administered intramuscularly into the deltoid muscle of the non-dominant arm.
- Fendrix - HLA Subsets Group: This group consisted in the subset of subjects in the Fendrix Group identified with a pre-defined Human Leukocytes Antigen (HLA) Class I or II subtype aged between, and including, 18 and 45 years at the time of first vaccination received 2 doses of Fendrix™, at Days 0 and 30, followed by one booster dose of Hepatitis B surface antigens (HBsAg) at Day 360. The Fendrix™ vaccine and HBsAg antigens were administered intramuscularly into the deltoid muscle of the non-dominant arm.
- Engerix-B - HLA Subsets Group: This group consisted in the subset of subjects in the Engerix-B Group identified with a pre-defined Human Leukocytes Antigen (HLA) Class I or II subtype aged between, and including, 18 and 45 years at the time of first vaccination received 2 doses of Engerix-B™, at Days 0 and 30, followed by one booster dose of Hepatitis B surface antigens (HBsAg) at Day 360. The Engerix-B™ vaccine and HBsAg antigens were administered intramuscularly into the deltoid muscle of the non-dominant arm.
Arm/Group | GSK223192A 1 - HLA Subsets Group | GSK223192A 2 - HLA Subsets Group | GSK223192A 3 - HLA Subsets Group | Fendrix - HLA Subsets Group | Engerix-B - HLA Subsets Group
Number analyzed (Participants) | 59 | 57 | 58 | 62 | 57
mIU/mL
  Anti HBs, Day 0 | 3.1 [3.1 to 3.2] | 0 [0 to 0] | 3.3 [3.1 to 3.6] | 0 [0 to 0] | 0 [0 to 0]
  Anti HBs, Day 30: number analyzed (Participants) | 59 | 57 | 58 | 60 | 55
  Anti HBs, Day 30 | 108.0 [65.0 to 179.6] | 59.6 [31.9 to 111.5] | 66.3 [35.7 to 123.0] | 6.1 [4.2 to 9.1] | 3.5 [2.9 to 4.2]
  Anti HBs, Day 44: number analyzed (Participants) | 59 | 56 | 57 | 60 | 53
  Anti HBs, Day 44 | 11986.2 [8676.4 to 16558.7] | 7942.6 [5288.7 to 11928.2] | 5525.4 [3639.3 to 8389.2] | 220.2 [126.5 to 383.3] | 19.2 [11.1 to 33.2]
  Anti HBs, Day 60: number analyzed (Participants) | 59 | 57 | 58 | 59 | 55
  Anti HBs, Day 60 | 7454.3 [5603.6 to 9916.2] | 5030.9 [3396.4 to 7452.1] | 4194.3 [2805.4 to 6270.8] | 251.9 [150.6 to 421.5] | 21.5 [12.7 to 36.4]

13. Secondary Outcome: Anti-HB Antibody Concentrations in Serum, as Measured by Chemi Luminescence Immuno Assay (CLIA)
Description: as for outcome 12
Time Frame: At Days 0, 180 and 360
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | GSK223192A 1 - HLA Subsets Group | GSK223192A 2 - HLA Subsets Group | GSK223192A 3 - HLA Subsets Group | Fendrix - HLA Subsets Group | Engerix-B - HLA Subsets Group
Number analyzed (Participants) | 58 | 54 | 55 | 56 | 54
mIU/mL
  Anti HBs, Day 0 | 3.1 [3.1 to 3.2] | 3.1 [3.1 to 3.1] | 3.3 [3.1 to 3.6] | 3.1 [3.1 to 3.1] | 3.1 [3.1 to 3.1]
  Anti HBs, Day 180: number analyzed (Participants) | 57 | 54 | 55 | 55 | 53
  Anti HBs, Day 180 | 3840.7 [2953.4 to 4994.6] | 2657.5 [1972.1 to 3581.0] | 3330.2 [2502.2 to 4432.1] | 254.5 [169.9 to 381.2] | 39.0 [23.3 to 65.2]
  Anti HBs, Day 360: number analyzed (Participants) | 58 | 53 | 54 | 54 | 51
  Anti HBs, Day 360 | 2150.7 [1602.7 to 2885.9] | 1650.6 [1159.7 to 2349.4] | 2122.5 [1542.3 to 2921.1] | 94.5 [59.6 to 149.8] | 19.8 [12.5 to 31.3]

14. Secondary Outcome: Anti-HB Antibody Concentrations in Serum, as Measured by CLIA
Description: as for outcome 12
Time Frame: At Days 0, 374 and 390
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | GSK223192A 1 - HLA Subsets Group | GSK223192A 2 - HLA Subsets Group | GSK223192A 3 - HLA Subsets Group | Fendrix - HLA Subsets Group | Engerix-B - HLA Subsets Group
Number analyzed (Participants) | 55 | 52 | 54 | 54 | 50
mIU/mL
  Anti HBs, Day 0 | 3.1 [3.1 to 3.2] | 3.1 [3.1 to 3.1] | 3.3 [3.1 to 3.6] | 3.1 [3.1 to 3.1] | 3.1 [3.1 to 3.1]
  Anti HBs, Day 374: number analyzed (Participants) | 52 | 50 | 53 | 54 | 50
  Anti HBs, Day 374 | 51509.0 [35731.5 to 74253.1] | 31985.9 [22628.6 to 45212.7] | 27135.3 [19376.8 to 38000.5] | 3788.4 [2047.8 to 7008.6] | 341.3 [143.7 to 810.4]
  Anti HBs, Day 390: number analyzed (Participants) | 52 | 48 | 53 | 51 | 50
  Anti HBs, Day 390 | 43674.6 [29975.7 to 63633.8] | 27035.7 [18737.0 to 39009.7] | 25105.7 [17730.1 to 35549.4] | 3352.2 [1756.0 to 6399.1] | 351.1 [147.0 to 838.5]

15. Secondary Outcome: Number of Hepatitis B (HB)-Specific Memory B Cells
Description: The number of HB-specific memory B-cells (HB mem-B cells), per million cells - expressed through tabulation of interquartile range data - was measured by B-cell Enzyme-Linked Immunosorbent Spot (ELISPOT) using Peripheral Blood Mononuclear Cells (PBMCs). This outcome measure concerns solely subjects part of the HLA Subsets 1 & 2 who received the Day 360 booster dose of HBsAg.
Time Frame: At Days 0, 30, 37, 44 and 60.
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: HB mem-B cells (per million cells)
Arm/Group | GSK223192A 1 - HLA Subsets Group | GSK223192A 2 - HLA Subsets Group | GSK223192A 3 - HLA Subsets Group | Fendrix - HLA Subsets Group | Engerix-B - HLA Subsets Group
Number analyzed (Participants) | 54 | 53 | 55 | 54 | 52
HB mem-B cells (per million cells)
  HB-mem B cells, at Day 0: number analyzed (Participants) | 50 | 51 | 53 | 53 | 51
  HB-mem B cells, at Day 0 | 14 [1 to 64] | 1 [1 to 44] | 1 [1 to 39] | 1 [1 to 38] | 1 [1 to 55]
  HB-mem B cells, at Day 30: number analyzed (Participants) | 54 | 51 | 55 | 53 | 52
  HB-mem B cells, at Day 30 | 296 [38 to 1161] | 186 [35 to 776] | 265 [48 to 759] | 28 [1 to 86] | 1 [1 to 54]
  HB-mem B cells, at Day 37: number analyzed (Participants) | 52 | 53 | 48 | 53 | 52
  HB-mem B cells, at Day 37 | 3817 [1440 to 9196] | 3577 [1486 to 9753] | 2597 [1028 to 8770] | 71 [1 to 167] | 19 [1 to 85]
  HB-mem B cells, at Day 44: number analyzed (Participants) | 54 | 52 | 50 | 51 | 48
  HB-mem B cells, at Day 44 | 4656 [1430 to 7808] | 4808 [1845 to 11274] | 2498 [672 to 7782] | 51 [1 to 299] | 28 [1 to 114]
  HB-mem B cells, at Day 60: number analyzed (Participants) | 52 | 51 | 54 | 53 | 47
  HB-mem B cells, at Day 60 | 3742 [835 to 7997] | 3383 [1467 to 8145] | 1806 [599 to 5833] | 47 [1 to 152] | 44 [1 to 161]

16. Secondary Outcome: Number of HB-specific Memory B Cells
Description: as for outcome 15
Time Frame: At Days 180 and 360
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: HB mem-B cells (per million cells)
Arm/Group | GSK223192A 1 - HLA Subsets Group | GSK223192A 2 - HLA Subsets Group | GSK223192A 3 - HLA Subsets Group | Fendrix - HLA Subsets Group | Engerix-B - HLA Subsets Group
Number analyzed (Participants) | 53 | 51 | 52 | 50 | 51
HB mem-B cells (per million cells)
  HB-mem B cells, at Day 180: number analyzed (Participants) | 49 | 48 | 49 | 45 | 50
  HB-mem B cells, at Day 180 | 1454 [395 to 2486] | 1013 [227 to 2164] | 1410 [567 to 2671] | 24 [1 to 128] | 1 [1 to 67]
  HB-mem B cells, at Day 360: number analyzed (Participants) | 52 | 46 | 50 | 49 | 49
  HB-mem B cells, at Day 360 | 1070 [747 to 2616] | 1437 [306 to 2770] | 1473 [463 to 2430] | 66 [1 to 255] | 21 [1 to 104]

17. Secondary Outcome: Concentrations of the Interferon-gamma (IFN-g), Interleukin (IL)-1beta, IL-5, IL-6, IL-10, Tumor Necrosis Factor-alpha, IFN-g-inducible Protein-10 and Monocyte Chemotactic Protein-1 Cytokines in Serum
Description: Concentrations of IFN-g, IL-1 beta (IL-1B), IL-5, IL-6, IL-10, Tumor Necrosis Factor-alpha (TNF-a), IFN-g-inducible protein-10 (IP-10) and monocyte chemotactic protein (MCP)-1 Concentrations of the IFN-g, IL-1B, IL-5, IL-6, IL-10, TNF-a, IP-10 and MCP-1 cytokines in serum were measured by Cytokine bead assay (CBA) and expressed in picograms per milliliter (pg/mL). This outcome measure concerns solely subjects part of the HLA Subsets 1 & 2 who received the Day 360 booster dose of HBsAg.
Time Frame: At Days 0, 0+ (Day 0 + 3 to 6 hours), 1, 30,30+ (Day 30 + 3 to 6 hours), 31, 33 and 37.
Population: Analysis was done on the According-to-Protocol (ATP) cohort for innate immunogenicity to Day 60, which included all evaluable subjects with immunogenicity and innate response (=early immune response [i.e. cytokines in serum, gene expression signature, white blood cells counts]) results available for at least one post-vaccination time point.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | GSK223192A 1 - HLA Subsets Group | GSK223192A 2 - HLA Subsets Group | GSK223192A 3 - HLA Subsets Group | Fendrix - HLA Subsets Group | Engerix-B - HLA Subsets Group
Number analyzed (Participants) | 59 | 57 | 61 | 61 | 55
pg/mL
  IFN-g; Day 0: number analyzed (Participants) | 59 | 57 | 59 | 60 | 55
  IFN-g; Day 0 | 3.704 [3.704 to 3.704] | 3.704 [3.704 to 3.704] | 3.704 [3.704 to 3.704] | 3.704 [3.704 to 3.704] | 3.704 [3.704 to 3.704]
  IFN-g; Day 0+: number analyzed (Participants) | 59 | 57 | 59 | 61 | 55
  IFN-g; Day 0+ | 3.704 [3.704 to 3.704] | 3.704 [3.704 to 3.704] | 3.704 [3.704 to 3.704] | 3.704 [3.704 to 3.704] | 3.704 [3.704 to 3.704]
  IFN-g; Day 1: number analyzed (Participants) | 58 | 57 | 58 | 61 | 55
  IFN-g; Day 1 | 3.704 [3.704 to 3.704] | 3.704 [3.704 to 3.704] | 3.704 [3.704 to 3.704] | 3.704 [3.704 to 3.704] | 3.704 [3.704 to 3.704]
  IFN-g; Day 30: number analyzed (Participants) | 59 | 57 | 57 | 59 | 55
  IFN-g; Day 30 | 3.704 [3.704 to 3.704] | 3.704 [3.704 to 3.704] | 3.704 [3.704 to 3.704] | 3.704 [3.704 to 3.704] | 3.704 [3.704 to 3.704]
  IFN-g; Day 30+: number analyzed (Participants) | 59 | 57 | 57 | 59 | 54
  IFN-g; Day 30+ | 3.704 [3.704 to 3.704] | 3.704 [3.704 to 3.704] | 3.704 [3.704 to 3.704] | 3.704 [3.704 to 3.704] | 3.704 [3.704 to 3.704]
  IFN-g; Day 31: number analyzed (Participants) | 58 | 57 | 56 | 57 | 55
  IFN-g; Day 31 | 5.568 [3.704 to 57.695] | 3.704 [3.704 to 21.747] | 3.704 [3.704 to 5.575] | 3.704 [3.704 to 3.704] | 3.704 [3.704 to 3.704]
  IFN-g; Day 33: number analyzed (Participants) | 59 | 57 | 57 | 59 | 55
  IFN-g; Day 33 | 3.704 [3.704 to 3.704] | 3.704 [3.704 to 3.704] | 3.704 [3.704 to 3.704] | 3.704 [3.704 to 3.704] | 3.704 [3.704 to 3.704]
  IFN-g; Day 37: number analyzed (Participants) | 59 | 56 | 57 | 58 | 55
  IFN-g; Day 37 | 3.704 [3.704 to 3.704] | 3.704 [3.704 to 3.704] | 3.704 [3.704 to 3.704] | 3.704 [3.704 to 3.704] | 3.704 [3.704 to 3.704]
  IL-1B; Day 0: number analyzed (Participants) | 59 | 57 | 59 | 60 | 55
  IL-1B; Day 0 | 0.411 [0.411 to 1.837] | 1.379 [0.411 to 3.046] | 0.411 [0.411 to 1.937] | 0.411 [0.411 to 2.516] | 0.411 [0.411 to 2.06]
  IL-1B; Day 0+: number analyzed (Participants) | 59 | 57 | 59 | 61 | 55
  IL-1B; Day 0+ | 1.636 [0.411 to 2.087] | 1.873 [0.411 to 2.742] | 0.856 [0.411 to 2.535] | 0.947 [0.411 to 2.394] | 1.146 [0.411 to 2.674]
  IL-1B; Day 1: number analyzed (Participants) | 58 | 57 | 58 | 61 | 55
  IL-1B; Day 1 | 2.024 [0.852 to 3.406] | 2.237 [1.302 to 4.214] | 1.912 [0.411 to 3.07] | 1.628 [0.856 to 2.449] | 1.885 [1.094 to 3.819]
  IL-1B; Day 30: number analyzed (Participants) | 59 | 57 | 57 | 59 | 55
  IL-1B; Day 30 | 1.232 [0.411 to 2.385] | 0.879 [0.411 to 2.26] | 1.017 [0.411 to 2.631] | 0.925 [0.411 to 2.516] | 0.411 [0.411 to 2.326]
  IL-1B; Day 30+: number analyzed (Participants) | 59 | 57 | 57 | 59 | 54
  IL-1B; Day 30+ | 1.292 [0.411 to 2.333] | 1.099 [0.411 to 2.28] | 0.856 [0.411 to 2.332] | 1.214 [0.411 to 1.981] | 1.349 [0.411 to 2.384]
  IL-1B; Day 31: number analyzed (Participants) | 58 | 57 | 56 | 57 | 55
  IL-1B; Day 31 | 0.991 [0.411 to 2.577] | 1.263 [0.411 to 2.528] | 1.117 [0.411 to 3.164] | 1.159 [0.411 to 2.581] | 1.135 [0.411 to 2.775]
  IL-1B; Day 33: number analyzed (Participants) | 59 | 57 | 57 | 59 | 55
  IL-1B; Day 33 | 0.411 [0.411 to 1.432] | 0.411 [0.411 to 1.886] | 0.411 [0.411 to 2.182] | 0.411 [0.411 to 1.77] | 0.86 [0.411 to 1.88]
  IL-1B; Day 37: number analyzed (Participants) | 59 | 56 | 57 | 58 | 55
  IL-1B; Day 37 | 0.411 [0.411 to 1.585] | 0.411 [0.411 to 2.41] | 0.411 [0.411 to 1.506] | 0.411 [0.411 to 2.122] | 0.411 [0.411 to 2.764]
  IL-10; Day 0: number analyzed (Participants) | 59 | 57 | 59 | 60 | 55
  IL-10; Day 0 | 0.411 [0.411 to 0.411] | 0.411 [0.411 to 1.051] | 0.411 [0.411 to 1.13] | 0.411 [0.411 to 0.411] | 0.411 [0.411 to 0.411]
  IL-10; Day 0+: number analyzed (Participants) | 59 | 57 | 59 | 61 | 55
  IL-10; Day 0+ | 0.411 [0.411 to 1.597] | 0.411 [0.411 to 1.516] | 0.411 [0.411 to 1.31] | 0.411 [0.411 to 0.904] | 0.411 [0.411 to 1.46]
  IL-10; Day 1: number analyzed (Participants) | 58 | 57 | 58 | 61 | 55
  IL-10; Day 1 | 0.977 [0.411 to 2.135] | 1.08 [0.411 to 2.323] | 1.055 [0.411 to 2.518] | 0.893 [0.411 to 1.813] | 0.916 [0.411 to 2.593]
  IL-10; Day 30: number analyzed (Participants) | 59 | 57 | 57 | 59 | 55
  IL-10; Day 30 | 0.411 [0.411 to 1.409] | 0.411 [0.411 to 1.165] | 0.411 [0.411 to 1.799] | 0.411 [0.411 to 1.289] | 0.411 [0.411 to 0.967]
  IL-10; Day 30+: number analyzed (Participants) | 59 | 57 | 57 | 59 | 54
  IL-10; Day 30+ | 0.411 [0.411 to 1.113] | 0.411 [0.411 to 1.027] | 0.411 [0.411 to 1.082] | 0.411 [0.411 to 0.867] | 0.411 [0.411 to 0.908]
  IL-10; Day 31: number analyzed (Participants) | 58 | 57 | 56 | 57 | 55
  IL-10; Day 31 | 0.705 [0.411 to 2.233] | 0.411 [0.411 to 1.961] | 0.411 [0.411 to 2.046] | 0.411 [0.411 to 1.392] | 0.411 [0.411 to 1.303]
  IL-10; Day 33: number analyzed (Participants) | 59 | 57 | 57 | 59 | 55
  IL-10; Day 33 | 0.411 [0.411 to 0.411] | 0.411 [0.411 to 1.165] | 0.411 [0.411 to 1.208] | 0.411 [0.411 to 0.989] | 0.411 [0.411 to 0.411]
  IL-10; Day 37: number analyzed (Participants) | 59 | 56 | 57 | 58 | 55
  IL-10; Day 37 | 0.411 [0.411 to 0.844] | 0.411 [0.411 to 0.906] | 0.411 [0.411 to 0.984] | 0.411 [0.411 to 1.425] | 0.411 [0.411 to 1.052]
  IL-5; Day 0: number analyzed (Participants) | 59 | 57 | 59 | 60 | 55
  IL-5; Day 0 | 0.411 [0.411 to 1.662] | 0.411 [0.411 to 2.413] | 0.905 [0.411 to 1.677] | 0.867 [0.411 to 1.917] | 0.411 [0.411 to 1.619]
  IL-5; Day 0+: number analyzed (Participants) | 59 | 57 | 59 | 61 | 55
  IL-5; Day 0+ | 1.161 [0.411 to 2.094] | 1.37 [0.411 to 2.089] | 0.905 [0.411 to 2.017] | 0.411 [0.411 to 1.77] | 1.092 [0.411 to 2.105]
  IL-5; Day 1: number analyzed (Participants) | 58 | 57 | 58 | 61 | 55
  IL-5; Day 1 | 2.004 [0.932 to 2.758] | 2.089 [1.092 to 3.095] | 1.83 [0.411 to 3.049] | 1.77 [1.023 to 2.73] | 1.942 [1.23 to 3.143]
  IL-5; Day 30: number analyzed (Participants) | 59 | 57 | 57 | 59 | 55
  IL-5; Day 30 | 1.202 [0.411 to 1.972] | 0.411 [0.411 to 1.663] | 1.011 [0.411 to 2.733] | 0.89 [0.411 to 2.403] | 0.411 [0.411 to 2.381]
  IL-5; Day 30+: number analyzed (Participants) | 59 | 57 | 57 | 59 | 54
  IL-5; Day 30+ | 0.884 [0.411 to 2.024] | 0.916 [0.411 to 2.028] | 0.411 [0.411 to 2.15] | 0.992 [0.411 to 1.89] | 0.411 [0.411 to 2.273]
  IL-5; Day 31: number analyzed (Participants) | 58 | 57 | 56 | 57 | 55
  IL-5; Day 31 | 1.119 [0.411 to 2.719] | 0.951 [0.411 to 2.664] | 1.289 [0.411 to 2.901] | 1.113 [0.411 to 2.367] | 0.99 [0.411 to 2.501]
  IL-5; Day 33: number analyzed (Participants) | 59 | 57 | 57 | 59 | 55
  IL-5; Day 33 | 0.411 [0.411 to 1.599] | 0.411 [0.411 to 2.134] | 1.192 [0.411 to 2.948] | 0.411 [0.411 to 2.047] | 0.411 [0.411 to 2.221]
  IL-5; Day 37: number analyzed (Participants) | 59 | 56 | 57 | 58 | 55
  IL-5; Day 37 | 0.411 [0.411 to 1.509] | 0.411 [0.411 to 2.015] | 0.411 [0.411 to 1.43] | 0.411 [0.411 to 2.262] | 0.411 [0.411 to 2.661]
  IL-6; Day 0: number analyzed (Participants) | 59 | 57 | 59 | 60 | 55
  IL-6; Day 0 | 1.291 [0.411 to 1.984] | 1.19 [0.411 to 2.783] | 1.291 [0.411 to 1.946] | 1.26 [0.411 to 2.176] | 1.055 [0.411 to 1.768]
  IL-6; Day 0+: number analyzed (Participants) | 59 | 57 | 59 | 61 | 55
  IL-6; Day 0+ | 2.882 [2.018 to 4.57] | 2.523 [1.55 to 3.977] | 1.605 [0.411 to 2.652] | 1.579 [1.174 to 2.278] | 1.418 [0.411 to 2.049]
  IL-6; Day 1: number analyzed (Participants) | 58 | 57 | 58 | 61 | 55
  IL-6; Day 1 | 4.07 [2.707 to 5.621] | 2.578 [1.748 to 3.807] | 2.223 [1.435 to 3.637] | 2.147 [1.658 to 3.273] | 1.739 [1.159 to 2.819]
  IL-6; Day 30: number analyzed (Participants) | 59 | 57 | 57 | 59 | 55
  IL-6; Day 30 | 1.641 [0.92 to 2.839] | 1.377 [0.411 to 1.982] | 1.79 [0.411 to 2.564] | 1.653 [0.411 to 2.368] | 1.218 [0.411 to 2.229]
  IL-6; Day 30+: number analyzed (Participants) | 59 | 57 | 57 | 59 | 54
  IL-6; Day 30+ | 3.195 [2.056 to 5.288] | 2.53 [1.589 to 3.87] | 1.664 [1.074 to 2.223] | 1.753 [1.273 to 2.341] | 1.394 [0.411 to 2.272]
  IL-6; Day 31: number analyzed (Participants) | 58 | 57 | 56 | 57 | 55
  IL-6; Day 31 | 7.459 [5.284 to 10.345] | 4.174 [2.925 to 7.202] | 3.457 [1.971 to 5.488] | 2.538 [1.521 to 4.016] | 1.567 [0.861 to 2.316]
  IL-6; Day 33: number analyzed (Participants) | 59 | 57 | 57 | 59 | 55
  IL-6; Day 33 | 1.644 [1.1 to 3.287] | 1.253 [0.411 to 2.538] | 1.435 [0.411 to 2.405] | 1.676 [0.937 to 2.456] | 1.389 [0.411 to 2.001]
  IL-6; Day 37: number analyzed (Participants) | 59 | 56 | 57 | 58 | 55
  IL-6; Day 37 | 1.003 [0.411 to 1.982] | 0.976 [0.411 to 1.875] | 0.95 [0.411 to 1.938] | 1.321 [0.411 to 1.946] | 1.158 [0.411 to 2.17]
  IP-10; Day 0: number analyzed (Participants) | 59 | 57 | 58 | 60 | 55
  IP-10; Day 0 | 94 [70 to 162] | 92 [68 to 141] | 101.5 [62 to 136] | 102 [64.5 to 154.5] | 91 [61 to 136]
  IP-10; Day 0+: number analyzed (Participants) | 57 | 57 | 59 | 61 | 54
  IP-10; Day 0+ | 80 [53 to 117] | 81 [54 to 113] | 78 [46 to 113] | 80 [52 to 109] | 75.5 [55 to 100]
  IP-10; Day 1: number analyzed (Participants) | 58 | 57 | 58 | 60 | 55
  IP-10; Day 1 | 147 [99 to 252] | 111 [71 to 154] | 92.5 [61 to 144] | 85.5 [71.5 to 106] | 85 [52 to 140]
  IP-10; Day 30: number analyzed (Participants) | 59 | 57 | 57 | 59 | 55
  IP-10; Day 30 | 103 [72 to 154] | 109 [72 to 160] | 106 [77 to 180] | 104 [75 to 173] | 107 [77 to 173]
  IP-10; Day 30+: number analyzed (Participants) | 59 | 57 | 56 | 59 | 54
  IP-10; Day 30+ | 75 [49 to 101] | 63 [41 to 103] | 70.5 [30.5 to 105] | 68 [42 to 100] | 70 [49 to 108]
  IP-10; Day 31: number analyzed (Participants) | 58 | 57 | 56 | 57 | 55
  IP-10; Day 31 | 295 [130 to 465] | 211 [129 to 377] | 176.5 [83.5 to 304] | 63 [51 to 100] | 76 [48 to 117]
  IP-10; Day 33: number analyzed (Participants) | 59 | 57 | 57 | 59 | 55
  IP-10; Day 33 | 232 [163 to 393] | 170 [111 to 269] | 156 [99 to 274] | 86 [53 to 119] | 84 [52 to 127]
  IP-10; Day 37: number analyzed (Participants) | 59 | 56 | 57 | 58 | 55
  IP-10; Day 37 | 119 [88 to 185] | 100.5 [62.5 to 151.5] | 90 [71 to 138] | 83.5 [54 to 123] | 85 [54 to 144]
  MCP-1; Day 0: number analyzed (Participants) | 59 | 57 | 58 | 60 | 55
  MCP-1; Day 0 | 130 [92 to 205] | 168 [100 to 211] | 148.5 [104 to 194] | 143 [93.5 to 219.5] | 120 [83 to 182]
  MCP-1; Day 0+: number analyzed (Participants) | 57 | 57 | 59 | 61 | 54
  MCP-1; Day 0+ | 112 [73 to 183] | 141 [99 to 175] | 114 [83 to 175] | 131 [91 to 181] | 95 [68 to 167]
  MCP-1; Day 1: number analyzed (Participants) | 58 | 57 | 58 | 60 | 55
  MCP-1; Day 1 | 144 [97 to 198] | 139 [88 to 208] | 111.5 [88 to 170] | 133.5 [92.5 to 193] | 133 [80 to 187]
  MCP-1; Day 30: number analyzed (Participants) | 59 | 57 | 57 | 59 | 55
  MCP-1; Day 30 | 151 [70 to 245] | 179 [111 to 233] | 164 [119 to 213] | 165 [109 to 275] | 161 [94 to 227]
  MCP-1; Day 30+: number analyzed (Participants) | 59 | 57 | 56 | 59 | 54
  MCP-1; Day 30+ | 140 [72 to 193] | 114 [84 to 176] | 121.5 [80.5 to 185] | 121 [74 to 195] | 114.5 [80 to 162]
  MCP-1; Day 31: number analyzed (Participants) | 58 | 57 | 56 | 57 | 55
  MCP-1; Day 31 | 171 [112 to 283] | 155 [82 to 248] | 114.5 [91.5 to 186.5] | 120 [68 to 161] | 105 [61 to 175]
  MCP-1; Day 33: number analyzed (Participants) | 59 | 57 | 57 | 59 | 55
  MCP-1; Day 33 | 83 [48 to 134] | 92 [59 to 139] | 79 [50 to 136] | 122 [72 to 180] | 88 [56 to 151]
  MCP-1; Day 37: number analyzed (Participants) | 59 | 56 | 57 | 58 | 55
  MCP-1; Day 37 | 129 [75 to 182] | 138.5 [102 to 176] | 150 [111 to 196] | 140.5 [87 to 201] | 133 [74 to 170]
  TNF-a; Day 0: number analyzed (Participants) | 59 | 57 | 59 | 60 | 55
  TNF-a; Day 0 | 0.411 [0.411 to 1.348] | 1.262 [0.411 to 2.484] | 0.411 [0.411 to 1.707] | 0.651 [0.411 to 1.893] | 0.411 [0.411 to 1.455]
  TNF-a; Day 0+: number analyzed (Participants) | 59 | 57 | 59 | 61 | 55
  TNF-a; Day 0+ | 1.482 [0.411 to 2.309] | 1.641 [0.411 to 2.276] | 0.411 [0.411 to 2.128] | 0.411 [0.411 to 1.889] | 0.911 [0.411 to 2.274]
  TNF-a; Day 1: number analyzed (Participants) | 58 | 57 | 58 | 61 | 55
  TNF-a; Day 1 | 1.902 [0.411 to 2.346] | 1.909 [1.079 to 3.135] | 1.727 [0.411 to 3.277] | 1.579 [0.411 to 2.274] | 1.701 [0.411 to 2.907]
  TNF-a; Day 30: number analyzed (Participants) | 59 | 57 | 57 | 59 | 55
  TNF-a; Day 30 | 0.969 [0.411 to 2.192] | 1.023 [0.411 to 1.809] | 1.203 [0.411 to 2.568] | 0.411 [0.411 to 2.298] | 0.411 [0.411 to 2.032]
  TNF-a; Day 30+: number analyzed (Participants) | 59 | 57 | 57 | 59 | 54
  TNF-a; Day 30+ | 1.069 [0.411 to 1.796] | 1.08 [0.411 to 2.196] | 1.321 [0.411 to 2.204] | 1.243 [0.411 to 1.853] | 1.323 [0.411 to 2.124]
  TNF-a; Day 31: number analyzed (Participants) | 58 | 57 | 56 | 57 | 55
  TNF-a; Day 31 | 0.881 [0.411 to 2.507] | 1.151 [0.411 to 2.399] | 1.081 [0.411 to 3.366] | 1.091 [0.411 to 2.257] | 1.375 [0.411 to 2.249]
  TNF-a; Day 33: number analyzed (Participants) | 59 | 57 | 57 | 59 | 55
  TNF-a; Day 33 | 0.411 [0.411 to 1.568] | 0.981 [0.411 to 1.853] | 1.129 [0.411 to 2.486] | 0.411 [0.411 to 2.084] | 0.411 [0.411 to 2.204]
  TNF-a; Day 37: number analyzed (Participants) | 59 | 56 | 57 | 58 | 55
  TNF-a; Day 37 | 0.411 [0.411 to 1.879] | 0.934 [0.411 to 2.158] | 0.411 [0.411 to 1.826] | 0.411 [0.411 to 2.483] | 0.841 [0.411 to 2.399]

18. Secondary Outcome: Normalized Levels of White Blood Cells (WBC) and Creatine Phosphokinases (CPK)
Description: Analysis of levels of CPK and WBC was performed with reference to the range observed at the Immune Health (IH) Centre in La Louvière, Belgium. Levels are presented as normalized levels vs. the IH center. Normalization was performed as follows: (Raw result - lower limit normal (LLN) at the IH center) divided by (Upper Limit Normal (ULN) at the IH center minus LLN at the IH center). This outcome measure concerns solely subjects part of the HLA Subsets 1 & 2 who received the Day 360 booster dose of HBsAg.
Time Frame: At Days 0, 0+ (Day 0 + 3 to 6 hours), 1, 30, 30+ (Day 30 + 3 to 6 hours), 31, 33, 37 and 60.
Population: as for outcome 17
Measure: Median (Inter-Quartile Range); unit: IH Center normalized ratio
Arm/Group | GSK223192A 1 - HLA Subsets Group | GSK223192A 2 - HLA Subsets Group | GSK223192A 3 - HLA Subsets Group | Fendrix - HLA Subsets Group | Engerix-B - HLA Subsets Group
Number analyzed (Participants) | 59 | 57 | 59 | 61 | 55
IH Center normalized ratio
  WBC; Day 0 | 6840 [5520 to 7647.619] | 6090 [5230 to 7680] | 6650 [5130 to 8210] | 6523.81 [5542.857 to 7350] | 6480 [5320 to 7540]
  WBC; Day 0+ | 7729.231 [6340 to 9157.895] | 7670 [6111.111 to 9368.421] | 7520 [6460 to 9290] | 7620 [6860 to 8421.053] | 7210 [6300 to 9063.655]
  WBC; Day 1: number analyzed (Participants) | 58 | 57 | 58 | 61 | 55
  WBC; Day 1 | 8265 [7000 to 9838.095] | 7850 [6400 to 9066.667] | 7610 [6540 to 9530] | 8400 [7200 to 9200] | 7130 [5750 to 8110]
  WBC; Day 30: number analyzed (Participants) | 59 | 57 | 57 | 59 | 55
  WBC; Day 30 | 5960 [5260 to 7866.667] | 6090 [5230 to 7500] | 6290 [5152.381 to 7797.342] | 6421.053 [5570 to 7680] | 6076.923 [5430 to 7580.952]
  WBC; Day 30+: number analyzed (Participants) | 59 | 57 | 57 | 59 | 54
  WBC; Day 30+ | 7570 [6430 to 8838.095] | 7350 [5894.737 to 8620] | 7120 [5980 to 8720] | 7371.429 [6133.333 to 8680] | 7625 [6270 to 8520]
  WBC; Day 31: number analyzed (Participants) | 59 | 57 | 56 | 59 | 55
  WBC; Day 31 | 8160 [7110 to 10170] | 7533.333 [6759.754 to 8920] | 7422.222 [6405 to 8352.641] | 7980 [6950 to 9090] | 6550 [5580 to 7410]
  WBC; Day 33: number analyzed (Participants) | 59 | 57 | 57 | 59 | 55
  WBC; Day 33 | 6450 [5010 to 7971.429] | 6080 [4990 to 7360] | 6290 [5650 to 7560] | 7150 [6210 to 8130] | 6170 [5314.286 to 8150]
  WBC; Day 37: number analyzed (Participants) | 59 | 56 | 57 | 58 | 55
  WBC; Day 37 | 6219.048 [5520 to 7790.476] | 6464.341 [5455 to 8130] | 6760 [5530 to 8000] | 6740 [5685.714 to 7560] | 6870 [5470 to 8333.333]
  WBC; Day 60: number analyzed (Participants) | 59 | 57 | 57 | 58 | 55
  WBC; Day 60 | 6400 [5280 to 8230] | 6320 [5466.667 to 7420] | 6090 [5320 to 8430] | 6540 [5257.143 to 7378.738] | 5970 [5100 to 7980.952]
  CPK; Day 0 | 113 [91 to 139.263] | 93 [73 to 121] | 110 [74.216 to 157.789] | 114 [85 to 175] | 84.108 [70 to 121.579]
  CPK; Day 0+ | 117 [90 to 156] | 99.297 [77 to 120.054] | 112 [73.351 to 159] | 114.842 [89.784 to 170.941] | 94 [74 to 114.842]
  CPK; Day 1: number analyzed (Participants) | 58 | 57 | 57 | 61 | 55
  CPK; Day 1 | 109 [81.135 to 136.947] | 89.784 [73 to 115] | 104 [76.443 to 141] | 102 [78.541 to 163.297] | 86 [70 to 123.514]
  CPK, at Day 30: number analyzed (Participants) | 59 | 57 | 57 | 59 | 55
  CPK, at Day 30 | 123.263 [93 to 172.444] | 90 [72 to 114.842] | 115.73 [73.569 to 163] | 99 [71.653 to 158.973] | 93 [74 to 137]
  CPK; Day 30+: number analyzed (Participants) | 59 | 57 | 57 | 59 | 54
  CPK; Day 30+ | 120 [96 to 174.541] | 91.772 [75 to 118.741] | 115.73 [74.216 to 158.108] | 106 [78 to 144.27] | 93 [75.081 to 143]
  CPK; Day 31: number analyzed (Participants) | 59 | 57 | 56 | 59 | 55
  CPK; Day 31 | 109 [83 to 153.529] | 90 [70.211 to 105] | 106.973 [74.5 to 141.973] | 103.614 [76 to 153.784] | 98 [75.081 to 142.541]
  CPK; Day 33: number analyzed (Participants) | 59 | 57 | 57 | 59 | 55
  CPK; Day 33 | 107 [80.316 to 149.459] | 87 [71.053 to 113.135] | 104 [69 to 147] | 101 [75.485 to 136.588] | 91.772 [75.485 to 119]
  CPK; Day 37: number analyzed (Participants) | 59 | 56 | 57 | 58 | 55
  CPK; Day 37 | 112.118 [81 to 153.529] | 93.986 [67.921 to 116.395] | 118 [78.359 to 172.811] | 106.311 [77 to 170.216] | 93.689 [69 to 126]
  CPK; Day 60: number analyzed (Participants) | 59 | 57 | 57 | 58 | 55
  CPK; Day 60 | 120 [85 to 174.632] | 85 [70 to 108.811] | 114 [85 to 157] | 110.647 [79.405 to 149.765] | 96 [76 to 131]

19. Secondary Outcome: Normalized Levels of C-reactive Protein (CRP)
Description: Analysis of levels of CRP was performed with reference to the range observed at the Immune Health (IH) Centre in La Louvière, Belgium. Levels are presented as normalized levels vs. the IH center. Normalization was performed as follows: (Raw result - lower limit normal (LLN) at the IH center) divided by (Upper Limit Normal (ULN) at the IH center minus LLN at the IH center). This outcome measure concerns solely subjects part of the HLA Subsets 1 & 2 who received the Day 360 booster dose of HBsAg.
Time Frame: At Days 0, 0+ (Day 0 + 3 to 6 hours), 1, 30, 30+ (Day 30 + 3 to 6 hours), 31, 33 and 37.
Population: as for outcome 17
Measure: Median (Inter-Quartile Range); unit: IH Center normlized ratio
Arm/Group | GSK223192A 1 - HLA Subsets Group | GSK223192A 2 - HLA Subsets Group | GSK223192A 3 - HLA Subsets Group | Fendrix - HLA Subsets Group | Engerix-B - HLA Subsets Group
Number analyzed (Participants) | 59 | 57 | 59 | 61 | 55
IH Center normlized ratio
  CRP; Day 0: number analyzed (Participants) | 59 | 57 | 59 | 61 | 54
  CRP; Day 0 | 0.248 [0.18 to 0.326] | 0.248 [0.15 to 0.51] | 0.248 [0.13 to 0.55] | 0.248 [0.17 to 0.486] | 0.248 [0.09 to 0.486]
  CRP; Day 0+: number analyzed (Participants) | 59 | 57 | 59 | 61 | 54
  CRP; Day 0+ | 0.248 [0.14 to 0.391] | 0.248 [0.12 to 0.5] | 0.248 [0.14 to 0.52] | 0.248 [0.17 to 0.486] | 0.248 [0.1 to 0.462]
  CRP; Day 1: number analyzed (Participants) | 58 | 57 | 58 | 61 | 55
  CRP; Day 1 | 1.97 [0.795 to 3.342] | 0.962 [0.486 to 1.661] | 0.486 [0.25 to 0.94] | 0.462 [0.248 to 0.724] | 0.248 [0.11 to 0.462]
  CRP; Day 30: number analyzed (Participants) | 58 | 57 | 57 | 57 | 53
  CRP; Day 30 | 0.248 [0.187 to 0.486] | 0.248 [0.17 to 0.34] | 0.248 [0.129 to 0.486] | 0.248 [0.2 to 0.486] | 0.248 [0.15 to 0.486]
  CRP; Day 30+: number analyzed (Participants) | 59 | 57 | 57 | 59 | 54
  CRP; Day 30+ | 0.248 [0.192 to 0.53] | 0.248 [0.18 to 0.34] | 0.248 [0.13 to 0.486] | 0.248 [0.2 to 0.52] | 0.248 [0.15 to 0.486]
  CRP; Day 31: number analyzed (Participants) | 59 | 56 | 55 | 59 | 55
  CRP; Day 31 | 1.521 [0.87 to 2.39] | 1.047 [0.498 to 1.518] | 0.61 [0.248 to 1.224] | 0.486 [0.248 to 0.724] | 0.248 [0.129 to 0.486]
  CRP; Day 33: number analyzed (Participants) | 58 | 56 | 56 | 59 | 55
  CRP; Day 33 | 2.6 [1.438 to 4.333] | 1.2 [0.637 to 2.186] | 0.707 [0.46 to 1.365] | 0.486 [0.248 to 0.962] | 0.248 [0.129 to 0.486]
  CRP; Day 37: number analyzed (Participants) | 59 | 55 | 55 | 56 | 53
  CRP; Day 37 | 0.319 [0.229 to 0.641] | 0.248 [0.17 to 0.486] | 0.248 [0.13 to 0.41] | 0.248 [0.229 to 0.478] | 0.248 [0.12 to 0.468]

20. Secondary Outcome: Normalized Levels of WBC and of CPK
Description: Analysis of levels of CPK and WBC was performed with reference to the range observed at the Immune Health (IH) Centre in La Louvière, Belgium. Levels are presented as normalized levels vs. the IH center. Normalization was performed as follows: (Raw result - lower limit normal (LLN) at the IH center) divided by (Upper Limit Normal (ULN) at the IH center minus LLN at the IH center). This outcome measure concerns all subjects except subjects part of the HLA Subsets 1 and 2.
Time Frame: At Days 0, 30, 37 and 60.
Population: Analysis was done on the Total Vaccinated cohort which included all vaccinated subjects, on subjects for whom results were available for the timepoint/outcome analyzed.
Measure: Median (Inter-Quartile Range); unit: IH Center normalized ratio
Groups:
- GSK223192A 1 - Non-HLA Subsets Group: This group consisted in the subjects in the GSK223192A 1 Group who were not identified with a pre-defined Human Leukocytes Antigen (HLA) Class I or II subtype. Subjects in this group were aged between, and including, 18 and 45 years at the time of first vaccination and received 2 doses of GSK223192A vaccine, lot 1, at Days 0 and 30. The GSK223192A vaccine antigens were administered intramuscularly into the deltoid muscle of the non-dominant arm.
- GSK223192A 2 - Non-HLA Subsets Group: This group consisted in the subjects in the GSK223192A 2 Group who were not identified with a pre-defined Human Leukocytes Antigen (HLA) Class I or II subtype. Subjects in this group were aged between, and including, 18 and 45 years at the time of first vaccination and received 2 doses of GSK223192A vaccine, lot 2, at Days 0 and 30. The GSK223192A vaccine antigens were administered intramuscularly into the deltoid muscle of the non-dominant arm.
- GSK223192A 3 - Non-HLA Subsets Group: This group consisted in the subjects in the GSK223192A 3 Group who were not identified with a pre-defined Human Leukocytes Antigen (HLA) Class I or II subtype. Subjects in this group were aged between, and including, 18 and 45 years at the time of first vaccination and received 2 doses of GSK223192A vaccine, lot 3, at Days 0 and 30. The GSK223192A vaccine was administered intramuscularly into the deltoid muscle of the non-dominant arm.
- Fendrix - Non-HLA Subsets Group: This group consisted in the subjects in the Fendrix Group who were not identified with a pre-defined Human Leukocytes Antigen (HLA) Class I or II subtype. Subjects in this group were aged between, and including, 18 and 45 years at the time of first vaccination and received 2 doses of Fendrix™, at Days 0 and 30. The Fendrix™ vaccine was administered intramuscularly into the deltoid muscle of the non-dominant arm.
- Engerix-B - Non-HLA Subsets Group: This group consisted in the subjects in the Engerix-B Group who were not identified with a pre-defined Human Leukocytes Antigen (HLA) Class I or II subtype. Subjects in this group were aged between, and including, 18 and 45 years at the time of first vaccination and received 2 doses of Engerix-B™, at Days 0 and 30. The Engerix-B™ vaccine was administered intramuscularly into the deltoid muscle of the non-dominant arm.
Arm/Group | GSK223192A 1 - Non-HLA Subsets Group | GSK223192A 2 - Non-HLA Subsets Group | GSK223192A 3 - Non-HLA Subsets Group | Fendrix - Non-HLA Subsets Group | Engerix-B - Non-HLA Subsets Group
Number analyzed (Participants) | 68 | 68 | 66 | 71 | 67
IH Center normalized ratio
  WBC; Day 0 | 6627.764 [5719.286 to 8273.819] | 6748.689 [5403.462 to 8568.018] | 6782.414 [5578.947 to 8350] | 7590 [5810 to 8550] | 6810 [5573.77 to 8020]
  WBC; Day 30: number analyzed (Participants) | 68 | 65 | 65 | 69 | 66
  WBC; Day 30 | 6870.05 [5643.182 to 7705] | 6454.545 [5735.385 to 7888.889] | 6600 [5555.556 to 7900] | 6950.82 [5475.41 to 8777.778] | 6590 [5720 to 8272.727]
  WBC; Day 37: number analyzed (Participants) | 65 | 66 | 61 | 66 | 63
  WBC; Day 37 | 6736.842 [5772.308 to 7960] | 7196.579 [6113.846 to 8454.545] | 6550 [5672.131 to 8622.951] | 6673.182 [5550 to 8264.615] | 6440 [5770 to 8650]
  WBC; Day 60: number analyzed (Participants) | 68 | 66 | 60 | 68 | 65
  WBC; Day 60 | 6738.636 [5999.933 to 8061.393] | 6330 [5333.333 to 8181.818] | 6625.789 [5265 to 8110.526] | 7175.909 [5420 to 9099.817] | 6740 [5530 to 8090]
  CPK; Day 0 | 105.529 [76 to 140.279] | 102.696 [82.842 to 135.314] | 109.756 [86.706 to 184.919] | 114 [87 to 159.474] | 120.857 [71.622 to 184.4]
  CPK; Day 30: number analyzed (Participants) | 68 | 65 | 65 | 68 | 66
  CPK; Day 30 | 108.617 [79.697 to 148.105] | 103.647 [81 to 128.316] | 114 [88.4 to 172.947] | 102.1 [87.885 to 135.311] | 113.079 [79 to 151.333]
  CPK; Day 37: number analyzed (Participants) | 65 | 66 | 61 | 66 | 63
  CPK; Day 37 | 105.351 [84.824 to 141.676] | 99.399 [77.294 to 132.891] | 109.294 [88.054 to 147.655] | 122.66 [88.919 to 161.059] | 124.667 [82 to 203.081]
  CPK; Day 60: number analyzed (Participants) | 68 | 66 | 61 | 68 | 65
  CPK; Day 60 | 112.842 [84.5 to 187.354] | 104 [75.6 to 140.105] | 107.6 [78.541 to 152.919] | 102.4 [84.333 to 146.793] | 120.989 [84.526 to 178]

21. Secondary Outcome: Normalized Levels of CRP
Description: Analysis of levels of CRP was performed with reference to the range observed at the Immune Health (IH) Centre in La Louvière, Belgium. Levels are presented as normalized levels vs. the IH center. Normalization was performed as follows: (Raw result - lower limit normal (LLN) at the IH center) divided by (Upper Limit Normal (ULN) at the IH center minus LLN at the IH center). This outcome measure concerns all subjects except subjects part of the HLA Subsets 1 and 2.
Time Frame: At Days 0, 30 and 37.
Population: as for outcome 20
Measure: Median (Inter-Quartile Range); unit: IH Center normalized levels
Arm/Group | GSK223192A 1 - Non-HLA Subsets Group | GSK223192A 2 - Non-HLA Subsets Group | GSK223192A 3 - Non-HLA Subsets Group | Fendrix - Non-HLA Subsets Group | Engerix-B - Non-HLA Subsets Group
Number analyzed (Participants) | 66 | 66 | 64 | 69 | 66
IH Center normalized levels
  CRP; Day 0: number analyzed (Participants) | 65 | 65 | 64 | 69 | 66
  CRP; Day 0 | 0.33 [0.153 to 0.755] | 0.486 [0.248 to 0.739] | 0.253 [0.229 to 0.739] | 0.296 [0.224 to 0.739] | 0.365 [0.178 to 0.739]
  CRP; Day 30 | 0.248 [0.129 to 0.724] | 0.371 [0.208 to 0.739] | 0.38 [0.248 to 0.739] | 0.277 [0.19 to 0.739] | 0.319 [0.105 to 0.739]
  CRP; Day 37: number analyzed (Participants) | 64 | 65 | 59 | 66 | 59
  CRP; Day 37 | 0.486 [0.272 to 0.807] | 0.523 [0.248 to 1.224] | 0.486 [0.248 to 1.152] | 0.363 [0.229 to 0.836] | 0.248 [0.114 to 0.739]

22. Secondary Outcome: Levels of White Blood Cells, Neutrophils, Lymphocytes, Monocytes, Eosinophils and Basophils
Description: Levels of white blood cells (WBC) as absolute counts, neutrophils (NEU), lymphocytes (LYM), monocytes (MON), eosinophils (EOS) and basophils (BAS) were assessed with reference to the range observed at the Immune Health (IH) Centre in La Louvière, Belgium. This outcome measure presents the raw data collected in percent (%), expressed in IH Center normalized levels based on raw data in % (IH normalized %), and concerns solely subjects part of the HLA Subsets 1 & 2 who received the Day 360 booster dose of HBsAg.
Time Frame: At Days 0, 0+ (Day 0 + 3 to 6 hours), 1, 30, 30+ (Day 30 + 3 to 6 hours), 31, 33, 37 and 60.
Population: as for outcome 17
Measure: Median (Inter-Quartile Range); unit: IH normalized ratio
Arm/Group | GSK223192A 1 - HLA Subsets Group | GSK223192A 2 - HLA Subsets Group | GSK223192A 3 - HLA Subsets Group | Fendrix - HLA Subsets Group | Engerix-B - HLA Subsets Group
Number analyzed (Participants) | 21 | 17 | 14 | 22 | 14
IH normalized ratio
  WBC; Day 0 | 0.498 [0.323 to 0.608] | 0.509 [0.422 to 0.93] | 0.341 [0.143 to 0.756] | 0.43 [0.246 to 0.517] | 0.479 [0.329 to 0.608]
  WBC; Day 0+ | 0.702 [0.427 to 0.886] | 1.123 [0.476 to 1.205] | 0.578 [0.395 to 1.051] | 0.647 [0.518 to 0.926] | 0.662 [0.498 to 0.927]
  WBC; Day 1: number analyzed (Participants) | 20 | 17 | 14 | 22 | 14
  WBC; Day 1 | 0.76 [0.485 to 0.969] | 0.756 [0.459 to 0.971] | 0.54 [0.351 to 1.154] | 0.698 [0.593 to 0.895] | 0.607 [0.448 to 0.84]
  WBC; Day 30: number analyzed (Participants) | 21 | 17 | 13 | 22 | 14
  WBC; Day 30 | 0.456 [0.246 to 0.644] | 0.596 [0.219 to 0.878] | 0.263 [0.193 to 0.549] | 0.385 [0.249 to 0.479] | 0.517 [0.392 to 0.684]
  WBC; Day 30+: number analyzed (Participants) | 21 | 17 | 13 | 22 | 14
  WBC; Day 30+ | 0.69 [0.546 to 0.844] | 0.789 [0.479 to 1.098] | 0.574 [0.371 to 0.814] | 0.556 [0.356 to 0.737] | 0.76 [0.479 to 0.86]
  WBC; Day 31: number analyzed (Participants) | 21 | 17 | 12 | 22 | 14
  WBC; Day 31 | 0.79 [0.617 to 1.018] | 0.737 [0.46 to 0.938] | 0.629 [0.476 to 0.763] | 0.633 [0.562 to 0.789] | 0.536 [0.443 to 0.772]
  WBC; Day 33: number analyzed (Participants) | 21 | 17 | 13 | 22 | 14
  WBC; Day 33 | 0.441 [0.229 to 0.662] | 0.491 [0.222 to 0.719] | 0.404 [0.303 to 0.646] | 0.441 [0.299 to 0.579] | 0.537 [0.219 to 0.772]
  WBC; Day 37: number analyzed (Participants) | 21 | 17 | 13 | 22 | 14
  WBC; Day 37 | 0.379 [0.298 to 0.646] | 0.525 [0.335 to 0.781] | 0.468 [0.31 to 0.544] | 0.354 [0.263 to 0.537] | 0.49 [0.251 to 0.983]
  WBC; Day 60: number analyzed (Participants) | 21 | 17 | 13 | 22 | 14
  WBC; Day 60 | 0.41 [0.213 to 0.634] | 0.557 [0.244 to 0.737] | 0.271 [0.123 to 0.584] | 0.42 [0.21 to 0.563] | 0.446 [0.222 to 0.665]
  NEU; Day 0 | 0.648 [0.422 to 0.83] | 0.53 [0.478 to 0.894] | 0.58 [0.3 to 0.837] | 0.663 [0.343 to 0.85] | 0.445 [0.41 to 0.541]
  NEU; Day 0+ | 0.84 [0.652 to 0.957] | 0.752 [0.627 to 0.993] | 0.693 [0.47 to 0.797] | 0.767 [0.581 to 0.87] | 0.654 [0.443 to 0.713]
  NEU; Day 1: number analyzed (Participants) | 20 | 17 | 14 | 22 | 14
  NEU; Day 1 | 0.93 [0.727 to 1.15] | 0.817 [0.653 to 0.903] | 0.727 [0.67 to 0.927] | 0.769 [0.635 to 0.923] | 0.654 [0.53 to 0.8]
  NEU; Day 30: number analyzed (Participants) | 21 | 17 | 13 | 22 | 14
  NEU; Day 30 | 0.604 [0.46 to 0.757] | 0.6 [0.387 to 0.791] | 0.387 [0.322 to 0.757] | 0.578 [0.35 to 0.719] | 0.581 [0.46 to 0.699]
  NEU; Day 30+: number analyzed (Participants) | 21 | 17 | 13 | 22 | 14
  NEU; Day 30+ | 0.9 [0.497 to 1.107] | 0.717 [0.583 to 0.887] | 0.609 [0.377 to 0.84] | 0.663 [0.521 to 0.95] | 0.642 [0.465 to 0.717]
  NEU; Day 31: number analyzed (Participants) | 21 | 17 | 12 | 22 | 14
  NEU; Day 31 | 1.161 [1.067 to 1.373] | 0.959 [0.797 to 1.135] | 0.921 [0.478 to 1.118] | 0.78 [0.672 to 0.943] | 0.589 [0.357 to 0.684]
  NEU; Day 33: number analyzed (Participants) | 21 | 17 | 13 | 22 | 14
  NEU; Day 33 | 0.591 [0.447 to 0.787] | 0.509 [0.275 to 0.69] | 0.539 [0.34 to 0.657] | 0.587 [0.426 to 0.819] | 0.567 [0.457 to 0.653]
  NEU; Day 37: number analyzed (Participants) | 21 | 17 | 13 | 22 | 14
  NEU; Day 37 | 0.63 [0.459 to 0.726] | 0.652 [0.503 to 0.77] | 0.443 [0.313 to 0.553] | 0.569 [0.365 to 0.823] | 0.542 [0.373 to 0.67]
  NEU; Day 60: number analyzed (Participants) | 21 | 17 | 13 | 22 | 14
  NEU; Day 60 | 0.656 [0.537 to 0.807] | 0.543 [0.391 to 0.667] | 0.54 [0.375 to 0.684] | 0.61 [0.363 to 0.843] | 0.561 [0.422 to 0.733]
  LYM; Day 0 | 0.474 [0.345 to 0.607] | 0.366 [0.341 to 0.524] | 0.531 [0.359 to 0.839] | 0.403 [0.235 to 0.557] | 0.68 [0.459 to 0.779]
  LYM; Day 0+ | 0.328 [0.045 to 0.438] | 0.407 [0.048 to 0.552] | 0.543 [0.41 to 0.679] | 0.361 [0.148 to 0.479] | 0.609 [0.354 to 0.745]
  LYM; Day 1: number analyzed (Participants) | 20 | 17 | 14 | 22 | 14
  LYM; Day 1 | 0.178 [-0.136 to 0.316] | 0.272 [0.093 to 0.341] | 0.412 [0.19 to 0.521] | 0.283 [0.059 to 0.472] | 0.478 [0.324 to 0.597]
  LYM; Day 30: number analyzed (Participants) | 21 | 17 | 13 | 22 | 14
  LYM; Day 30 | 0.452 [0.274 to 0.552] | 0.51 [0.221 to 0.538] | 0.528 [0.336 to 0.745] | 0.433 [0.207 to 0.634] | 0.536 [0.335 to 0.838]
  LYM; Day 30+: number analyzed (Participants) | 21 | 17 | 13 | 22 | 14
  LYM; Day 30+ | 0.3 [0.026 to 0.513] | 0.386 [0.222 to 0.5] | 0.497 [0.345 to 0.831] | 0.413 [0.266 to 0.479] | 0.54 [0.313 to 0.628]
  LYM; Day 31: number analyzed (Participants) | 21 | 17 | 12 | 22 | 14
  LYM; Day 31 | -0.086 [-0.2 to 0] | -0.003 [-0.179 to 0.269] | 0.15 [-0.11 to 0.526] | 0.302 [0.034 to 0.372] | 0.54 [0.348 to 0.776]
  LYM; Day 33: number analyzed (Participants) | 21 | 17 | 13 | 22 | 14
  LYM; Day 33 | 0.309 [0.231 to 0.531] | 0.407 [0.269 to 0.683] | 0.445 [0.31 to 0.552] | 0.405 [0.196 to 0.552] | 0.622 [0.314 to 0.731]
  LYM; Day 37: number analyzed (Participants) | 21 | 17 | 13 | 22 | 14
  LYM; Day 37 | 0.503 [0.279 to 0.57] | 0.357 [0.225 to 0.561] | 0.555 [0.493 to 0.683] | 0.423 [0.224 to 0.593] | 0.572 [0.27 to 0.779]
  LYM; Day 60: number analyzed (Participants) | 21 | 17 | 13 | 22 | 14
  LYM; Day 60 | 0.452 [0.257 to 0.645] | 0.376 [0.3 to 0.63] | 0.534 [0.441 to 0.731] | 0.402 [0.178 to 0.579] | 0.538 [0.4 to 0.779]
  MON; Day 0 | 0.5 [0.356 to 0.589] | 0.311 [0.222 to 0.489] | 0.439 [0.389 to 0.522] | 0.51 [0.4 to 0.64] | 0.489 [0.356 to 0.58]
  MON; Day 0+ | 0.422 [0.311 to 0.533] | 0.367 [0.32 to 0.4] | 0.367 [0.3 to 0.567] | 0.439 [0.321 to 0.54] | 0.389 [0.322 to 0.456]
  MON; Day 1: number analyzed (Participants) | 20 | 17 | 14 | 22 | 14
  MON; Day 1 | 0.594 [0.367 to 0.834] | 0.522 [0.422 to 0.622] | 0.522 [0.44 to 0.611] | 0.477 [0.359 to 0.622] | 0.45 [0.333 to 0.5]
  MON; Day 30: number analyzed (Participants) | 21 | 17 | 13 | 22 | 14
  MON; Day 30 | 0.533 [0.411 to 0.644] | 0.411 [0.322 to 0.522] | 0.5 [0.344 to 0.533] | 0.472 [0.378 to 0.551] | 0.422 [0.289 to 0.478]
  MON; Day 30+: number analyzed (Participants) | 21 | 17 | 13 | 22 | 14
  MON; Day 30+ | 0.456 [0.333 to 0.533] | 0.422 [0.302 to 0.544] | 0.433 [0.3 to 0.478] | 0.443 [0.367 to 0.589] | 0.363 [0.311 to 0.46]
  MON; Day 31: number analyzed (Participants) | 21 | 17 | 12 | 22 | 14
  MON; Day 31 | 0.533 [0.333 to 0.667] | 0.544 [0.444 to 0.756] | 0.632 [0.4 to 0.833] | 0.427 [0.333 to 0.6] | 0.478 [0.278 to 0.611]
  MON; Day 33: number analyzed (Participants) | 21 | 17 | 13 | 22 | 14
  MON; Day 33 | 0.767 [0.533 to 1.056] | 0.578 [0.378 to 0.711] | 0.656 [0.389 to 0.733] | 0.549 [0.389 to 0.656] | 0.472 [0.278 to 0.578]
  MON; Day 37: number analyzed (Participants) | 21 | 17 | 13 | 22 | 14
  MON; Day 37 | 0.478 [0.4 to 0.544] | 0.433 [0.311 to 0.5] | 0.433 [0.289 to 0.533] | 0.472 [0.311 to 0.567] | 0.394 [0.256 to 0.522]
  MON; Day 60: number analyzed (Participants) | 21 | 17 | 13 | 22 | 14
  MON; Day 60 | 0.5 [0.367 to 0.567] | 0.467 [0.378 to 0.556] | 0.456 [0.333 to 0.511] | 0.461 [0.356 to 0.6] | 0.344 [0.256 to 0.556]
  EOS; Day 0 | 0.5 [0.34 to 0.594] | 0.594 [0.475 to 0.875] | 0.37 [0.24 to 0.54] | 0.596 [0.4 to 1.1] | 0.495 [0.42 to 0.82]
  EOS; Day 0+ | 0.3 [0.225 to 0.4] | 0.429 [0.32 to 0.575] | 0.25 [0.125 to 0.44] | 0.423 [0.29 to 0.58] | 0.42 [0.375 to 0.58]
  EOS; Day 1: number analyzed (Participants) | 20 | 17 | 14 | 22 | 14
  EOS; Day 1 | 0.291 [0.194 to 0.478] | 0.48 [0.36 to 0.754] | 0.313 [0.24 to 0.531] | 0.464 [0.28 to 0.775] | 0.41 [0.26 to 0.66]
  EOS; Day 30: number analyzed (Participants) | 21 | 17 | 13 | 22 | 14
  EOS; Day 30 | 0.45 [0.3 to 0.6] | 0.673 [0.362 to 0.9] | 0.42 [0.26 to 0.878] | 0.693 [0.42 to 1.08] | 0.53 [0.32 to 0.75]
  EOS; Day 30+: number analyzed (Participants) | 21 | 17 | 13 | 22 | 14
  EOS; Day 30+ | 0.32 [0.25 to 0.348] | 0.475 [0.375 to 0.696] | 0.34 [0.174 to 0.6] | 0.496 [0.355 to 0.7] | 0.38 [0.348 to 0.56]
  EOS; Day 31: number analyzed (Participants) | 21 | 17 | 12 | 22 | 14
  EOS; Day 31 | 0.145 [0.1 to 0.275] | 0.38 [0.3 to 0.62] | 0.25 [0.167 to 0.493] | 0.505 [0.26 to 0.85] | 0.43 [0.3 to 0.525]
  EOS; Day 33: number analyzed (Participants) | 21 | 17 | 13 | 22 | 14
  EOS; Day 33 | 0.6 [0.36 to 0.7] | 0.667 [0.52 to 0.825] | 0.58 [0.26 to 1.02] | 0.645 [0.377 to 0.825] | 0.443 [0.36 to 0.64]
  EOS; Day 37: number analyzed (Participants) | 21 | 17 | 13 | 22 | 14
  EOS; Day 37 | 0.46 [0.325 to 0.625] | 0.64 [0.42 to 0.768] | 0.44 [0.3 to 0.939] | 0.69 [0.452 to 1.188] | 0.52 [0.28 to 0.78]
  EOS; Day 60: number analyzed (Participants) | 21 | 17 | 13 | 22 | 14
  EOS; Day 60 | 0.45 [0.36 to 0.575] | 0.652 [0.32 to 1.1] | 0.38 [0.3 to 0.653] | 0.709 [0.44 to 1.058] | 0.465 [0.28 to 0.623]
  BAS; Day 0 | 0.25 [0.158 to 0.35] | 0.35 [0.143 to 0.5] | 0.325 [0.214 to 0.421] | 0.25 [0.15 to 0.455] | 0.375 [0.25 to 0.5]
  BAS; Day 0+ | 0.25 [0.2 to 0.35] | 0.3 [0.2 to 0.4] | 0.232 [0.158 to 0.4] | 0.25 [0.1 to 0.3] | 0.225 [0.15 to 0.4]
  BAS; Day 1: number analyzed (Participants) | 20 | 17 | 14 | 22 | 14
  BAS; Day 1 | 0.232 [0.105 to 0.35] | 0.25 [0.2 to 0.35] | 0.286 [0.15 to 0.4] | 0.179 [0.1 to 0.3] | 0.25 [0.15 to 0.421]
  BAS; Day 30: number analyzed (Participants) | 21 | 17 | 13 | 22 | 14
  BAS; Day 30 | 0.4 [0.25 to 0.5] | 0.35 [0.25 to 0.5] | 0.35 [0.182 to 0.45] | 0.333 [0.2 to 0.5] | 0.3 [0.25 to 0.4]
  BAS; Day 30+: number analyzed (Participants) | 21 | 17 | 13 | 22 | 14
  BAS; Day 30+ | 0.25 [0.2 to 0.368] | 0.25 [0.214 to 0.45] | 0.25 [0.15 to 0.4] | 0.211 [0.15 to 0.45] | 0.333 [0.25 to 0.4]
  BAS; Day 31: number analyzed (Participants) | 21 | 17 | 12 | 22 | 14
  BAS; Day 31 | 0.2 [0.15 to 0.3] | 0.3 [0.211 to 0.4] | 0.3 [0.146 to 0.325] | 0.25 [0.158 to 0.364] | 0.325 [0.211 to 0.5]
  BAS; Day 33: number analyzed (Participants) | 21 | 17 | 13 | 22 | 14
  BAS; Day 33 | 0.35 [0.3 to 0.526] | 0.4 [0.25 to 0.65] | 0.35 [0.2 to 0.5] | 0.3 [0.182 to 0.5] | 0.3 [0.263 to 0.5]
  BAS; Day 37: number analyzed (Participants) | 21 | 17 | 13 | 22 | 14
  BAS; Day 37 | 0.316 [0.25 to 0.45] | 0.421 [0.3 to 0.55] | 0.286 [0.2 to 0.4] | 0.286 [0.15 to 0.5] | 0.3 [0.2 to 0.4]
  BAS; Day 60: number analyzed (Participants) | 21 | 17 | 13 | 22 | 14
  BAS; Day 60 | 0.3 [0.2 to 0.4] | 0.4 [0.3 to 0.6] | 0.4 [0.182 to 0.55] | 0.25 [0.15 to 0.421] | 0.308 [0.25 to 0.4]

23. Secondary Outcome: Levels of WBC, NEU, LYM, MON, EOS and BAS
Description: Levels of white blood cells (WBC) as absolute counts, neutrophils (NEU), lymphocytes (LYM), monocytes (MON), eosinophils (EOS) and basophils (BAS) were assessed with reference to the range observed at the Immune Health (IH) Centre in La Louvière, Belgium. This outcome measure presents the raw data collected in percent (%), expressed in IH Center normalized levels based on raw data in % (IH normalized %), and concerns all subjects except subjects part of the HLA Subsets 1 and 2.
Time Frame: At Days 0, 30, 37 and 60.
Population: as for outcome 20
Measure: Median (Inter-Quartile Range); unit: IH normalized ratio
Arm/Group | GSK223192A 1 - Non-HLA Subsets Group | GSK223192A 2 - Non-HLA Subsets Group | GSK223192A 3 - Non-HLA Subsets Group | Fendrix - Non-HLA Subsets Group | Engerix-B - Non-HLA Subsets Group
Number analyzed (Participants) | 47 | 47 | 42 | 43 | 47
IH normalized ratio
  WBC; Day 0 | 0.426 [0.262 to 0.79] | 0.413 [0.246 to 0.857] | 0.497 [0.273 to 0.722] | 0.672 [0.344 to 0.912] | 0.465 [0.258 to 0.722]
  WBC; Day 30: number analyzed (Participants) | 47 | 47 | 41 | 41 | 46
  WBC; Day 30 | 0.492 [0.262 to 0.618] | 0.426 [0.289 to 0.704] | 0.428 [0.258 to 0.697] | 0.573 [0.221 to 0.963] | 0.455 [0.332 to 0.786]
  WBC; Day 37: number analyzed (Participants) | 44 | 47 | 38 | 40 | 43
  WBC; Day 37 | 0.455 [0.293 to 0.644] | 0.574 [0.328 to 0.784] | 0.405 [0.243 to 0.77] | 0.523 [0.284 to 0.81] | 0.426 [0.275 to 0.826]
  WBC; Day 60: number analyzed (Participants) | 47 | 46 | 37 | 41 | 45
  WBC; Day 60 | 0.44 [0.311 to 0.718] | 0.44 [0.222 to 0.697] | 0.439 [0.166 to 0.754] | 0.607 [0.426 to 0.967] | 0.478 [0.28 to 0.832]
  NEU; Day 0: number analyzed (Participants) | 47 | 46 | 42 | 43 | 47
  NEU; Day 0 | 0.534 [0.291 to 0.752] | 0.559 [0.224 to 0.838] | 0.426 [0.297 to 0.633] | 0.503 [0.3 to 0.788] | 0.458 [0.256 to 0.705]
  NEU; Day 30: number analyzed (Participants) | 47 | 47 | 41 | 41 | 46
  NEU; Day 30 | 0.457 [0.17 to 0.703] | 0.524 [0.26 to 0.686] | 0.491 [0.075 to 0.726] | 0.5 [0.291 to 0.714] | 0.532 [0.326 to 0.796]
  NEU; Day 37: number analyzed (Participants) | 44 | 47 | 38 | 40 | 43
  NEU; Day 37 | 0.417 [0.225 to 0.698] | 0.5 [0.292 to 0.703] | 0.436 [0.125 to 0.708] | 0.458 [0.083 to 0.603] | 0.491 [0.334 to 0.726]
  NEU; Day 60: number analyzed (Participants) | 47 | 46 | 37 | 41 | 45
  NEU; Day 60 | 0.47 [0.333 to 0.715] | 0.496 [0.3 to 0.772] | 0.389 [0.167 to 0.57] | 0.471 [0.194 to 0.671] | 0.474 [0.294 to 0.731]
  LYM; Day 0: number analyzed (Participants) | 47 | 46 | 42 | 43 | 47
  LYM; Day 0 | 0.408 [0.183 to 0.6] | 0.388 [0.128 to 0.646] | 0.552 [0.248 to 0.757] | 0.37 [-0.05 to 0.613] | 0.45 [0.15 to 0.66]
  LYM; Day 30: number analyzed (Participants) | 47 | 47 | 41 | 41 | 46
  LYM; Day 30 | 0.45 [0.24 to 0.7] | 0.404 [0.26 to 0.69] | 0.55 [0.228 to 0.893] | 0.373 [0.15 to 0.69] | 0.43 [0.111 to 0.6]
  LYM; Day 37: number analyzed (Participants) | 44 | 47 | 38 | 40 | 43
  LYM; Day 37 | 0.514 [0.263 to 0.713] | 0.433 [0.183 to 0.62] | 0.605 [0.291 to 0.791] | 0.492 [0.334 to 0.7] | 0.43 [0.122 to 0.62]
  LYM; Day 60: number analyzed (Participants) | 47 | 46 | 37 | 41 | 45
  LYM; Day 60 | 0.45 [0.177 to 0.634] | 0.388 [0.168 to 0.65] | 0.578 [0.38 to 0.9] | 0.426 [0.25 to 0.683] | 0.417 [0.233 to 0.593]
  MON; Day 0: number analyzed (Participants) | 47 | 46 | 42 | 43 | 47
  MON; Day 0 | 0.52 [0.256 to 0.675] | 0.473 [0.333 to 0.64] | 0.5 [0.325 to 0.656] | 0.438 [0.3 to 0.611] | 0.55 [0.288 to 0.7]
  MON; Day 30: number analyzed (Participants) | 47 | 47 | 41 | 41 | 46
  MON; Day 30 | 0.556 [0.367 to 0.765] | 0.471 [0.267 to 0.783] | 0.538 [0.311 to 0.667] | 0.431 [0.319 to 0.733] | 0.506 [0.3 to 0.667]
  MON; Day 37: number analyzed (Participants) | 44 | 47 | 38 | 40 | 43
  MON; Day 37 | 0.471 [0.298 to 0.673] | 0.456 [0.333 to 0.738] | 0.465 [0.233 to 0.66] | 0.465 [0.261 to 0.744] | 0.5 [0.349 to 0.667]
  MON; Day 60: number analyzed (Participants) | 47 | 46 | 37 | 41 | 45
  MON; Day 60 | 0.463 [0.333 to 0.625] | 0.41 [0.256 to 0.8] | 0.444 [0.222 to 0.688] | 0.456 [0.322 to 0.733] | 0.5 [0.363 to 0.738]
  EOS; Day 0: number analyzed (Participants) | 47 | 46 | 42 | 43 | 47
  EOS; Day 0 | 0.304 [0.12 to 0.582] | 0.29 [0.164 to 0.775] | 0.275 [0.149 to 0.575] | 0.299 [0.15 to 0.667] | 0.319 [0.149 to 0.612]
  EOS; Day 30: number analyzed (Participants) | 47 | 47 | 41 | 41 | 46
  EOS; Day 30 | 0.4 [0.16 to 0.851] | 0.4 [0.179 to 0.806] | 0.35 [0.225 to 0.49] | 0.375 [0.269 to 0.716] | 0.333 [0.174 to 0.612]
  EOS; Day 37: number analyzed (Participants) | 44 | 47 | 38 | 40 | 43
  EOS; Day 37 | 0.409 [0.239 to 0.7] | 0.35 [0.179 to 0.667] | 0.329 [0.225 to 0.475] | 0.496 [0.308 to 1] | 0.522 [0.224 to 0.716]
  EOS; Day 60: number analyzed (Participants) | 47 | 46 | 37 | 41 | 45
  EOS; Day 60 | 0.429 [0.209 to 0.696] | 0.324 [0.164 to 0.661] | 0.299 [0.104 to 0.44] | 0.347 [0.209 to 0.68] | 0.388 [0.164 to 0.625]
  BAS; Day 0: number analyzed (Participants) | 47 | 46 | 42 | 43 | 47
  BAS; Day 0 | 0.263 [0.118 to 0.4] | 0.286 [0.176 to 0.5] | 0.3 [0.171 to 0.4] | 0.353 [0.229 to 0.6] | 0.353 [0.118 to 0.471]
  BAS; Day 30: number analyzed (Participants) | 47 | 47 | 41 | 41 | 46
  BAS; Day 30 | 0.3 [0.171 to 0.471] | 0.294 [0.171 to 0.5] | 0.316 [0.176 to 0.4] | 0.294 [0.2 to 0.474] | 0.316 [0.176 to 0.6]
  BAS; Day 37: number analyzed (Participants) | 44 | 47 | 38 | 40 | 43
  BAS; Day 37 | 0.351 [0.249 to 0.536] | 0.294 [0.114 to 0.4] | 0.377 [0.211 to 0.6] | 0.353 [0.174 to 0.5] | 0.3 [0.176 to 0.5]
  BAS; Day 60: number analyzed (Participants) | 47 | 46 | 37 | 41 | 45
  BAS; Day 60 | 0.3 [0.143 to 0.5] | 0.2 [0.118 to 0.4] | 0.4 [0.176 to 0.5] | 0.343 [0.286 to 0.5] | 0.286 [0.171 to 0.4]

24. Secondary Outcome: Normalized Levels of Red Blood Cells and Platelets
Description: Analysis of levels of red blood cells (RBC) and platelets (PLA) were assessed with reference to the range observed at the Immune Health (IH) Centre in La Louvière, Belgium. Levels are presented as normalized levels vs. the IH center. Normalization was performed as follows: (Raw result - lower limit normal (LLN) at the IH center) divided by (Upper Limit Normal (ULN) at the IH center minus LLN at the IH center). This outcome measure presents the raw data collected in absolute count, expressed in IH Center normalized levels based on absolute count data (IH normalized abs. count).
Time Frame: At Days 0, 30, 37 and 60.
Population: as for outcome 20
Measure: Median (Inter-Quartile Range); unit: cells/mL
Arm/Group | GSK223192A 1 Group | GSK223192A 2 Group | GSK223192A 3 Group | Fendrix Group | Engerix-B Group
Number analyzed (Participants) | 143 | 142 | 141 | 145 | 142
cells/mL
  RBC; Day 0 | 4.45 [4.269 to 4.618] | 4.433 [4.265 to 4.657] | 4.464 [4.26 to 4.662] | 4.38 [4.243 to 4.6] | 4.456 [4.293 to 4.65]
  RBC; Day 30: number analyzed (Participants) | 141 | 139 | 138 | 140 | 139
  RBC; Day 30 | 4.461 [4.278 to 4.584] | 4.382 [4.24 to 4.569] | 4.423 [4.257 to 4.65] | 4.388 [4.225 to 4.57] | 4.486 [4.243 to 4.651]
  RBC; Day 37: number analyzed (Participants) | 128 | 124 | 120 | 126 | 121
  RBC; Day 37 | 4.372 [4.23 to 4.534] | 4.346 [4.162 to 4.514] | 4.395 [4.2 to 4.583] | 4.37 [4.206 to 4.521] | 4.388 [4.23 to 4.61]
  RBC; Day 60: number analyzed (Participants) | 141 | 140 | 133 | 137 | 138
  RBC; Day 60 | 4.421 [4.243 to 4.555] | 4.393 [4.23 to 4.57] | 4.364 [4.214 to 4.579] | 4.371 [4.219 to 4.56] | 4.4 [4.231 to 4.579]
  PLA; Day 0 | 269318.18 [237500 to 309000] | 270833.33 [229000 to 313000] | 270000 [223333.33 to 309000] | 267187.5 [232000 to 325000] | 259000 [232000 to 308333.33]
  PLA; Day 30: number analyzed (Participants) | 141 | 139 | 138 | 140 | 139
  PLA; Day 30 | 261363.64 [229166.67 to 305000] | 262000 [228000 to 304000] | 260470.78 [222183.1 to 317410.71] | 274431.82 [232071.43 to 322206.9] | 258333.33 [218661.97 to 302288.73]
  PLA; Day 37: number analyzed (Participants) | 128 | 124 | 120 | 126 | 121
  PLA; Day 37 | 295000 [249166.67 to 338690.14] | 274431.82 [245596.15 to 333173.08] | 269000 [230403.85 to 321333.33] | 282477.27 [242500 to 335000] | 268622.45 [228000 to 322000]
  PLA; Day 60: number analyzed (Participants) | 141 | 140 | 133 | 137 | 138
  PLA; Day 60 | 263333.33 [230952.38 to 307954.55] | 267045.46 [221666.67 to 307477.27] | 259000 [224038.46 to 309000] | 273239.44 [243181.82 to 328409.09] | 262588.03 [228000 to 307000]

25. Secondary Outcome: Normalized Levels of Haemoglobin, Alanine Aminotransferase and Aspartate Aminotransferase
Description: Analysis of levels of haemoglobin (Hgb), alanine aminotransferase (ALT) and aspartate aminotransferase (AST) were assessed with reference to the range observed at the Immune Health (IH) Centre in La Louvière, Belgium. Levels are presented as normalized levels vs. the IH center. Normalization was performed as follows: (Raw result - lower limit normal (LLN) at the IH center) divided by (Upper Limit Normal (ULN) at the IH center minus LLN at the IH center). This outcome measure presents the raw data collected in absolute count, expressed in IH Center normalized levels based on absolute count data (IH normalized abs. count).
Time Frame: At Days 0, 30, 37 and 60.
Population: as for outcome 20
Measure: Median (Inter-Quartile Range); unit: cells/mL
Arm/Group | GSK223192A 1 Group | GSK223192A 2 Group | GSK223192A 3 Group | Fendrix Group | Engerix-B Group
Number analyzed (Participants) | 143 | 142 | 141 | 145 | 142
cells/mL
  Hgb; Day 0 | 13.4 [12.825 to 13.875] | 13.35 [12.75 to 13.9] | 13.4 [12.9 to 13.725] | 13.275 [12.7 to 13.725] | 13.35 [12.825 to 13.909]
  Hgb; Day 30: number analyzed (Participants) | 141 | 139 | 138 | 140 | 139
  Hgb; Day 30 | 13.35 [12.886 to 13.725] | 13.186 [12.7 to 13.725] | 13.275 [12.7 to 13.575] | 13.121 [12.501 to 13.715] | 13.35 [12.73 to 13.875]
  Hgb; Day 37: number analyzed (Participants) | 128 | 124 | 120 | 126 | 121
  Hgb; Day 37 | 13.05 [12.434 to 13.575] | 12.957 [12.513 to 13.382] | 13.025 [12.6 to 13.463] | 13.05 [12.525 to 13.568] | 13.05 [12.5 to 13.705]
  Hgb; Day 60: number analyzed (Participants) | 141 | 140 | 133 | 137 | 138
  Hgb; Day 60 | 13.275 [12.75 to 13.725] | 13.136 [12.468 to 13.675] | 13.1 [12.6 to 13.575] | 12.975 [12.467 to 13.568] | 13.163 [12.545 to 13.7]
  ALT; Day 0 | 21.086 [15.5 to 31.061] | 18.792 [13.968 to 27.675] | 18.636 [14.9 to 25.42] | 21.8 [15.6 to 29.294] | 21.32 [16 to 31.16]
  ALT; Day 30: number analyzed (Participants) | 141 | 139 | 138 | 140 | 139
  ALT; Day 30 | 21.32 [15.375 to 32.303] | 18.743 [13.12 to 26.2] | 19.897 [14.548 to 26.9] | 20.5 [15.375 to 27.89] | 18.743 [14.9 to 26.8]
  ALT; Day 37: number analyzed (Participants) | 128 | 124 | 120 | 126 | 121
  ALT; Day 37 | 21.221 [15.623 to 33.061] | 18.767 [13.021 to 25.574] | 18.596 [13.999 to 26.917] | 20.7 [15.229 to 27.06] | 19.8 [14.76 to 27.88]
  ALT; Day 60: number analyzed (Participants) | 141 | 140 | 134 | 137 | 138
  ALT; Day 60 | 21.161 [14.909 to 29.042] | 17.447 [13.16 to 24.848] | 18.07 [13.146 to 27.333] | 20.541 [15.58 to 28.576] | 18.518 [13.94 to 28.7]
  AST; Day 0 | 21 [18 to 25.065] | 20 [16.28 to 24.9] | 20 [17 to 23.727] | 21 [16.71 to 24.8] | 20.478 [17.8 to 24.8]
  AST; Day 30: number analyzed (Participants) | 141 | 139 | 138 | 140 | 139
  AST; Day 30 | 20.72 [18 to 27] | 19.24 [16.28 to 23.7] | 20.188 [17.76 to 24.314] | 20 [16.555 to 25.032] | 19.097 [16.71 to 23.871]
  AST; Day 37: number analyzed (Participants) | 128 | 124 | 120 | 126 | 121
  AST; Day 37 | 20.881 [17.01 to 25.371] | 19.097 [15.35 to 23.433] | 20.043 [17.267 to 22.97] | 20 [16.5 to 25.065] | 20 [16.28 to 23.68]
  AST; Day 60: number analyzed (Participants) | 141 | 140 | 134 | 137 | 138
  AST; Day 60 | 20.72 [17.02 to 24.667] | 17.986 [14.971 to 22.45] | 20.76 [16.313 to 23.871] | 21 [17 to 24.314] | 19.339 [16.6 to 24.314]

26. Secondary Outcome: Normalized Levels of Serum Creatinine, Urea and Lactate Dehydrogenase
Description: Analysis of levels of serum creatinine (S-CREA), urea and lactate dehydrogenase (LDH) were assessed with reference to the range observed at the Immune Health (IH) Centre in La Louvière, Belgium. Levels are presented as normalized levels vs. the IH center. Normalization was performed as follows: (Raw result - lower limit normal (LLN) at the IH center) divided by (Upper Limit Normal (ULN) at the IH center minus LLN at the IH center). This outcome measure presents the raw data collected in absolute count, expressed in IH Center normalized levels based on absolute count data (IH normalized abs. count).
Time Frame: At Days 0, 30, 37 and 60.
Population: as for outcome 20
Measure: Median (Inter-Quartile Range); unit: cells/mL
Arm/Group | GSK223192A 1 Group | GSK223192A 2 Group | GSK223192A 3 Group | Fendrix Group | Engerix-B Group
Number analyzed (Participants) | 143 | 142 | 141 | 145 | 142
cells/mL
  S-CREA; Day 0 | 0.893 [0.745 to 1.046] | 0.841 [0.705 to 0.982] | 0.889 [0.76 to 1.02] | 0.86 [0.722 to 1.025] | 0.85 [0.718 to 1.043]
  S-CREA, at Day 30: number analyzed (Participants) | 141 | 140 | 138 | 140 | 139
  S-CREA, at Day 30 | 0.9 [0.764 to 1.044] | 0.84 [0.7 to 0.983] | 0.874 [0.74 to 1.03] | 0.888 [0.718 to 1.046] | 0.87 [0.73 to 1.05]
  S-CREA; Day 37: number analyzed (Participants) | 128 | 124 | 120 | 126 | 120
  S-CREA; Day 37 | 0.906 [0.737 to 1.037] | 0.83 [0.701 to 0.98] | 0.883 [0.719 to 1.042] | 0.92 [0.74 to 1.043] | 0.909 [0.741 to 1.034]
  S-CREA; Day 60: number analyzed (Participants) | 141 | 140 | 134 | 137 | 138
  S-CREA; Day 60 | 0.92 [0.75 to 1.063] | 0.84 [0.727 to 1.003] | 0.873 [0.757 to 1.043] | 0.934 [0.76 to 1.052] | 0.915 [0.77 to 1.05]
  UREA; Day 0 | 29.5 [25.333 to 33.5] | 28.667 [24.895 to 32.833] | 30.095 [25.7 to 34.5] | 30 [26.167 to 34.5] | 29.202 [25.11 to 33.6]
  UREA; Day 30: number analyzed (Participants) | 141 | 140 | 138 | 140 | 139
  UREA; Day 30 | 30.127 [25.946 to 33.667] | 28.667 [25.333 to 32.988] | 30.462 [26.524 to 34.5] | 30.048 [26.293 to 34.404] | 30.095 [24.692 to 34.5]
  UREA; Day 37: number analyzed (Participants) | 128 | 124 | 120 | 126 | 121
  UREA; Day 37 | 29.5 [25.1 to 33.533] | 27.833 [23.623 to 31.183] | 30.333 [25.791 to 34.5] | 31 [26.9 to 34.5] | 28.667 [25.11 to 33.7]
  UREA; Day 60: number analyzed (Participants) | 141 | 140 | 134 | 137 | 138
  UREA; Day 60 | 29.8 [24.692 to 33.875] | 28.905 [24.895 to 33.35] | 29.5 [26 to 34.5] | 30.095 [26.6 to 34.308] | 29.65 [25.4 to 33.5]
  LHD; Day 0: number analyzed (Participants) | 143 | 141 | 141 | 145 | 142
  LHD; Day 0 | 336.364 [281.169 to 381.973] | 335.281 [283.1 to 372] | 328.3 [278.231 to 368.831] | 336.054 [291.991 to 384.156] | 325.85 [285 to 372.069]
  LHD; Day 30: number analyzed (Participants) | 141 | 139 | 138 | 140 | 138
  LHD; Day 30 | 343.75 [298.9 to 389.063] | 329.6 [283.333 to 375] | 330.32 [290.6 to 364.966] | 337.428 [289.068 to 385.753] | 320.671 [285.498 to 374.479]
  LHD; Day 37: number analyzed (Participants) | 128 | 124 | 120 | 126 | 121
  LHD; Day 37 | 348.894 [297.246 to 388.037] | 342.857 [288.8 to 380] | 331.967 [293.45 to 373.089] | 340.606 [289.5 to 378] | 319.048 [282.251 to 375]
  LHD; Day 60: number analyzed (Participants) | 141 | 140 | 134 | 137 | 138
  LHD; Day 60 | 341.975 [296.32 to 391] | 335.141 [270.7 to 376.435] | 324.675 [278.2 to 366.146] | 348.438 [295.2 to 378.571] | 320.927 [285.526 to 382.9]

27. Secondary Outcome: Number of Subjects With Normal and Abnormal Levels of White Blood Cells, Neutrophils, Lymphocytes, Monocytes, Eosinophils, Basophils, C-reactive Protein, and Creatine Phosphokinase.
Description: Subjects were assessed with regard to their normal (Nor.) and abnormal (Abn.) levels for the above parameters of white blood cells (WBC), neutrophils (NEU), lymphocytes (LYM), monocytes (MON), eosinophils (EOS), basophils (BAS), C-reactive protein (CRP) and creatine phosphokinase (CPK) at the Day 0 baseline versus their status post vaccination (Day 60). This outcome measure concerns solely subjects part of the HLA Subsets 1 & 2 who received the Day 360 booster dose of HBsAg.
Time Frame: At Day 0 and up to Day 60.
Population: as for outcome 20
Measure: Count of Participants; unit: Participants
Arm/Group | GSK223192A 1 - HLA Subsets Group | GSK223192A 2 - HLA Subsets Group | GSK223192A 3 - HLA Subsets Group | Fendrix - HLA Subsets Group | Engerix-B - HLA Subsets Group
Number analyzed (Participants) | 75 | 74 | 75 | 74 | 75
Participants
  BAS Abn. Day 0 - Abn. Day 60: number analyzed (Participants) | 3 | 2 | 4 | 5 | 4
  BAS Abn. Day 0 - Abn. Day 60 | 3 | 2 | 2 | 3 | 4
  BAS Abn. Day 0 - Nor. Day 60: number analyzed (Participants) | 3 | 2 | 4 | 5 | 4
  BAS Abn. Day 0 - Nor. Day 60 | 0 | 0 | 2 | 2 | 0
  BAS Nor. Day 0 - Abn. Day 60: number analyzed (Participants) | 72 | 72 | 71 | 69 | 71
  BAS Nor. Day 0 - Abn. Day 60 | 11 | 10 | 9 | 5 | 7
  BAS Nor. Day 0 - Nor. Day 60: number analyzed (Participants) | 72 | 72 | 71 | 69 | 71
  BAS Nor. Day 0 - Nor. Day 60 | 61 | 62 | 62 | 64 | 64
  CPK Abn. Day 0 - Abn. Day 60: number analyzed (Participants) | 12 | 11 | 13 | 14 | 10
  CPK Abn. Day 0 - Abn. Day 60 | 12 | 11 | 13 | 12 | 8
  CPK Abn. Day 0 - Nor. Day 60: number analyzed (Participants) | 12 | 11 | 13 | 14 | 10
  CPK Abn. Day 0 - Nor. Day 60 | 0 | 0 | 0 | 2 | 2
  CPK Nor. Day 0 - Abn. Day 60: number analyzed (Participants) | 63 | 63 | 62 | 60 | 65
  CPK Nor. Day 0 - Abn. Day 60 | 21 | 9 | 18 | 20 | 14
  CPK Nor. Day 0 - Nor. Day 60: number analyzed (Participants) | 63 | 63 | 62 | 60 | 65
  CPK Nor. Day 0 - Nor. Day 60 | 42 | 54 | 44 | 40 | 51
  CRP Abn. Day 0 - Abn. Day 60: number analyzed (Participants) | 3 | 8 | 5 | 4 | 4
  CRP Abn. Day 0 - Abn. Day 60 | 3 | 8 | 5 | 4 | 3
  CRP Abn. Day 0 - Nor. Day 60: number analyzed (Participants) | 3 | 8 | 5 | 4 | 4
  CRP Abn. Day 0 - Nor. Day 60 | 0 | 0 | 0 | 0 | 1
  CRP Nor. Day 0 - Abn. Day 60: number analyzed (Participants) | 72 | 66 | 70 | 70 | 70
  CRP Nor. Day 0 - Abn. Day 60 | 56 | 33 | 22 | 14 | 8
  CRP Nor. Day 0 - Nor. Day 60: number analyzed (Participants) | 72 | 66 | 70 | 70 | 70
  CRP Nor. Day 0 - Nor. Day 60 | 16 | 33 | 48 | 56 | 62
  EOS Abn. Day 0 - Abn. Day 60]: number analyzed (Participants) | 4 | 6 | 4 | 8 | 4
  EOS Abn. Day 0 - Abn. Day 60] | 3 | 6 | 3 | 7 | 3
  EOS Abn. Day 0 - Nor. Day 60: number analyzed (Participants) | 4 | 6 | 4 | 8 | 4
  EOS Abn. Day 0 - Nor. Day 60 | 1 | 0 | 1 | 1 | 1
  EOS Nor. Day 0 - Abn. Day 60: number analyzed (Participants) | 71 | 68 | 71 | 66 | 71
  EOS Nor. Day 0 - Abn. Day 60 | 13 | 9 | 6 | 6 | 6
  EOS Nor. Day 0 - Nor. Day 60: number analyzed (Participants) | 71 | 68 | 71 | 66 | 71
  EOS Nor. Day 0 - Nor. Day 60 | 58 | 59 | 65 | 60 | 65
  LYM Abn. Day 0 - Abn. Day 60: number analyzed (Participants) | 10 | 6 | 8 | 7 | 6
  LYM Abn. Day 0 - Abn. Day 60 | 10 | 6 | 7 | 6 | 5
  LYM Abn. Day 0 - Nor. Day 60: number analyzed (Participants) | 10 | 6 | 8 | 7 | 6
  LYM Abn. Day 0 - Nor. Day 60 | 0 | 0 | 1 | 1 | 1
  LYM Nor. Day 0 - Abn. Day 60: number analyzed (Participants) | 65 | 68 | 67 | 67 | 69
  LYM Nor. Day 0 - Abn. Day 60 | 30 | 29 | 16 | 11 | 10
  LYM Nor. Day 0 - Nor. Day 60: number analyzed (Participants) | 65 | 68 | 67 | 67 | 69
  LYM Nor. Day 0 - Nor. Day 60 | 35 | 39 | 51 | 56 | 59
  MON Abn. Day 0 - Abn. Day 60: number analyzed (Participants) | 1 | 5 | 7 | 4 | 0
  MON Abn. Day 0 - Abn. Day 60 | 1 | 3 | 4 | 4 | 0
  MON Abn. Day 0 - Nor. Day 60: number analyzed (Participants) | 1 | 5 | 7 | 4 | 0
  MON Abn. Day 0 - Nor. Day 60 | 0 | 2 | 3 | 0 | 0
  MON Nor. Day 0 - Abn. Day 60: number analyzed (Participants) | 74 | 69 | 68 | 70 | 75
  MON Nor. Day 0 - Abn. Day 60 | 29 | 15 | 12 | 8 | 6
  MON Nor. Day 0 - Nor. Day 60: number analyzed (Participants) | 74 | 69 | 68 | 70 | 75
  MON Nor. Day 0 - Nor. Day 60 | 45 | 54 | 56 | 62 | 69
  NEU Abn. Day 0 - Abn. Day 60: number analyzed (Participants) | 7 | 3 | 3 | 4 | 0
  NEU Abn. Day 0 - Abn. Day 60 | 7 | 2 | 3 | 3 | 0
  NEU Abn. Day 0 - Nor. Day 60: number analyzed (Participants) | 7 | 3 | 3 | 4 | 0
  NEU Abn. Day 0 - Nor. Day 60 | 0 | 1 | 0 | 1 | 0
  NEU Nor. Day 0 - Abn. Day 60: number analyzed (Participants) | 68 | 71 | 72 | 70 | 75
  NEU Nor. Day 0 - Abn. Day 60 | 32 | 27 | 19 | 13 | 8
  NEU Nor. Day 0 - Nor. Day 60: number analyzed (Participants) | 68 | 71 | 72 | 70 | 75
  NEU Nor. Day 0 - Nor. Day 60 | 36 | 44 | 53 | 57 | 67
  WBC Abn. Day 0 - Abn. Day 60: number analyzed (Participants) | 6 | 6 | 10 | 3 | 7
  WBC Abn. Day 0 - Abn. Day 60 | 6 | 5 | 9 | 2 | 6
  WBC Abn. Day 0 - Nor. Day 60: number analyzed (Participants) | 6 | 6 | 10 | 3 | 7
  WBC Abn. Day 0 - Nor. Day 60 | 0 | 1 | 1 | 1 | 1
  WBC Nor. Day 0 - Abn. Day 60: number analyzed (Participants) | 69 | 68 | 65 | 71 | 68
  WBC Nor. Day 0 - Abn. Day 60 | 30 | 26 | 19 | 19 | 14
  WBC Nor. Day 0 - Nor. Day 60: number analyzed (Participants) | 69 | 68 | 65 | 71 | 68
  WBC Nor. Day 0 - Nor. Day 60 | 39 | 42 | 46 | 52 | 54

28. Secondary Outcome: Number of Subjects With Normal and Abnormal Levels of WBC, NEU, LYM, MON, EOS, BAS, CRP, and CPK.
Description: Subjects were assessed with regard to their normal (Nor.) and abnormal (Abn.) levels for the above parameters of white blood cells (WBC), neutrophils (NEU), lymphocytes (LYM), monocytes (MON), eosinophils (EOS), basophils (BAS), C-reactive protein (CRP) and creatine phosphokinase (CPK) at the Day 0 baseline versus their status post vaccination (Day 60). This outcome measure concerns all subjects except subjects part of the HLA Subsets 1 and 2.
Time Frame: At Day 0 and up to Day 60.
Population: as for outcome 20
Measure: Count of Participants; unit: Participants
Arm/Group | GSK223192A 1 - Non-HLA Subsets Group | GSK223192A 2 - Non-HLA Subsets Group | GSK223192A 3 - Non-HLA Subsets Group | Fendrix - Non-HLA Subsets Group | Engerix-B - Non-HLA Subsets Group
Number analyzed (Participants) | 68 | 67 | 65 | 70 | 66
Participants
  BAS Abn. Day 0 - Abn. Day 60: number analyzed (Participants) | 4 | 4 | 2 | 6 | 3
  BAS Abn. Day 0 - Abn. Day 60 | 1 | 4 | 1 | 3 | 1
  BAS Abn. Day 0 - Nor. Day 60: number analyzed (Participants) | 4 | 4 | 2 | 6 | 3
  BAS Abn. Day 0 - Nor. Day 60 | 3 | 0 | 1 | 3 | 2
  BAS Nor. Day 0 - Abn. Day 60: number analyzed (Participants) | 64 | 62 | 63 | 64 | 63
  BAS Nor. Day 0 - Abn. Day 60 | 5 | 6 | 3 | 6 | 3
  BAS Nor. Day 0 - Nor. Day 60: number analyzed (Participants) | 64 | 62 | 63 | 64 | 63
  BAS Nor. Day 0 - Nor. Day 60 | 59 | 56 | 60 | 58 | 60
  CPK Abn. Day 0 - Abn. Day 60: number analyzed (Participants) | 12 | 7 | 18 | 13 | 17
  CPK Abn. Day 0 - Abn. Day 60 | 10 | 6 | 12 | 8 | 11
  CPK Abn. Day 0 - Nor. Day 60: number analyzed (Participants) | 12 | 7 | 18 | 13 | 17
  CPK Abn. Day 0 - Nor. Day 60 | 2 | 1 | 6 | 5 | 6
  CPK Nor. Day 0 - Abn. Day 60: number analyzed (Participants) | 56 | 60 | 47 | 57 | 49
  CPK Nor. Day 0 - Abn. Day 60 | 14 | 9 | 9 | 12 | 12
  CPK Nor. Day 0 - Nor. Day 60: number analyzed (Participants) | 56 | 60 | 47 | 57 | 49
  CPK Nor. Day 0 - Nor. Day 60 | 42 | 51 | 38 | 45 | 37
  CRP Abn. Day 0 - Abn. Day 60: number analyzed (Participants) | 8 | 12 | 9 | 5 | 8
  CRP Abn. Day 0 - Abn. Day 60 | 5 | 11 | 8 | 4 | 5
  CRP Abn. Day 0 - Nor. Day 60: number analyzed (Participants) | 8 | 12 | 9 | 5 | 8
  CRP Abn. Day 0 - Nor. Day 60 | 3 | 1 | 1 | 1 | 3
  CRP Nor. Day 0 - Abn. Day 60: number analyzed (Participants) | 57 | 51 | 54 | 62 | 56
  CRP Nor. Day 0 - Abn. Day 60 | 6 | 9 | 9 | 4 | 6
  CRP Nor. Day 0 - Nor. Day 60: number analyzed (Participants) | 57 | 51 | 54 | 62 | 56
  CRP Nor. Day 0 - Nor. Day 60 | 51 | 42 | 45 | 58 | 50
  EOS Abn. Day 0 - Abn. Day 60: number analyzed (Participants) | 9 | 9 | 5 | 6 | 7
  EOS Abn. Day 0 - Abn. Day 60 | 8 | 6 | 5 | 4 | 5
  EOS Abn. Day 0 - Nor. Day 60: number analyzed (Participants) | 9 | 9 | 5 | 6 | 7
  EOS Abn. Day 0 - Nor. Day 60 | 1 | 3 | 0 | 2 | 2
  EOS Nor. Day 0 - Abn. Day 60: number analyzed (Participants) | 59 | 57 | 60 | 64 | 59
  EOS Nor. Day 0 - Abn. Day 60 | 8 | 8 | 8 | 14 | 8
  EOS Nor. Day 0 - Nor. Day 60: number analyzed (Participants) | 59 | 57 | 60 | 64 | 59
  EOS Nor. Day 0 - Nor. Day 60 | 51 | 49 | 52 | 50 | 51
  LYM Abn. Day 0 - Abn. Day 60: number analyzed (Participants) | 8 | 10 | 7 | 14 | 11
  LYM Abn. Day 0 - Abn. Day 60 | 5 | 4 | 6 | 9 | 7
  LYM Abn. Day 0 - Nor. Day 60: number analyzed (Participants) | 8 | 10 | 7 | 14 | 11
  LYM Abn. Day 0 - Nor. Day 60 | 3 | 6 | 1 | 5 | 4
  LYM Nor. Day 0 - Abn. Day 60: number analyzed (Participants) | 60 | 56 | 58 | 56 | 55
  LYM Nor. Day 0 - Abn. Day 60 | 10 | 10 | 13 | 6 | 12
  LYM Nor. Day 0 - Nor. Day 60: number analyzed (Participants) | 60 | 56 | 58 | 56 | 55
  LYM Nor. Day 0 - Nor. Day 60 | 50 | 46 | 45 | 50 | 43
  MON Abn. Day 0 - Abn. Day 60: number analyzed (Participants) | 4 | 3 | 3 | 4 | 3
  MON Abn. Day 0 - Abn. Day 60 | 0 | 2 | 3 | 2 | 2
  MON Abn. Day 0 - Nor. Day 60: number analyzed (Participants) | 4 | 3 | 3 | 4 | 3
  MON Abn. Day 0 - Nor. Day 60 | 4 | 1 | 0 | 2 | 1
  MON Nor. Day 0 - Abn. Day 60: number analyzed (Participants) | 64 | 63 | 62 | 66 | 63
  MON Nor. Day 0 - Abn. Day 60 | 8 | 9 | 9 | 4 | 6
  MON Nor. Day 0 - Nor. Day 60: number analyzed (Participants) | 64 | 63 | 62 | 66 | 63
  MON Nor. Day 0 - Nor. Day 60 | 56 | 54 | 53 | 62 | 57
  NEU Abn. Day 0 - Abn. Day 60: number analyzed (Participants) | 5 | 8 | 6 | 6 | 8
  NEU Abn. Day 0 - Abn. Day 60 | 3 | 4 | 3 | 3 | 5
  NEU Abn. Day 0 - Nor. Day 60: number analyzed (Participants) | 5 | 8 | 6 | 6 | 8
  NEU Abn. Day 0 - Nor. Day 60 | 2 | 4 | 3 | 3 | 3
  NEU Nor. Day 0 - Abn. Day 60: number analyzed (Participants) | 63 | 58 | 59 | 64 | 58
  NEU Nor. Day 0 - Abn. Day 60 | 9 | 12 | 17 | 13 | 5
  NEU Nor. Day 0 - Nor. Day 60: number analyzed (Participants) | 63 | 58 | 59 | 64 | 58
  NEU Nor. Day 0 - Nor. Day 60 | 54 | 46 | 42 | 51 | 53
  WBC Abn. Day 0 - Abn. Day 60: number analyzed (Participants) | 7 | 10 | 9 | 12 | 9
  WBC Abn. Day 0 - Abn. Day 60 | 5 | 7 | 5 | 11 | 8
  WBC Abn. Day 0 - Nor. Day 60: number analyzed (Participants) | 7 | 10 | 9 | 12 | 9
  WBC Abn. Day 0 - Nor. Day 60 | 2 | 3 | 4 | 1 | 1
  WBC Nor. Day 0 - Abn. Day 60: number analyzed (Participants) | 61 | 57 | 56 | 58 | 57
  WBC Nor. Day 0 - Abn. Day 60 | 7 | 7 | 7 | 10 | 6
  WBC Nor. Day 0 - Nor. Day 60: number analyzed (Participants) | 61 | 57 | 56 | 58 | 57
  WBC Nor. Day 0 - Nor. Day 60 | 54 | 50 | 49 | 48 | 51

29. Secondary Outcome: Number of Subjects Presenting Normal and Abnormal Levels of White Blood Cells, Neutrophils, Lymphocytes, Monocytes, Eosinophils, Basophils, C-reactive Protein, and Creatine Phosphokinase.
Description: Subjects were assessed with regard to their normal (Nor.) and abnormal (Abn.) levels for the above parameters of white blood cells (WBC), neutrophils (NEU), lymphocytes (LYM), monocytes (MON), eosinophils (EOS), basophils (BAS), C-reactive protein (CRP) and creatine phosphokinase (CPK) at the Day 0 baseline versus their status post vaccination (Day 180 or 360). Day 180 or 360 results were chosen based on assessment of grading of the abnormality observed, with results for higher grading being tabulated.
Time Frame: Post vaccination (up to Day 360)
Population: as for outcome 20
Measure: Number; unit: Subjects
Arm/Group | GSK223192A 1 Group | GSK223192A 2 Group | GSK223192A 3 Group | Fendrix Group | Engerix-B Group
Number analyzed (Participants) | 138 | 140 | 131 | 133 | 135
Subjects
  BAS Abn. | 12 | 13 | 13 | 11 | 12
  BAS Nor. | 126 | 127 | 118 | 122 | 123
  CPK Abn. | 35 | 25 | 36 | 38 | 37
  CPK Nor. | 103 | 115 | 95 | 95 | 98
  EOS Abn. | 13 | 20 | 20 | 19 | 10
  EOS Nor. | 125 | 120 | 111 | 114 | 125
  LYM Abn. | 19 | 22 | 19 | 22 | 25
  LYM Nor. | 119 | 118 | 112 | 111 | 110
  MON Abn. | 12 | 10 | 13 | 14 | 9
  MON Nor. | 126 | 130 | 118 | 119 | 126
  NEU Abn. | 14 | 18 | 24 | 16 | 15
  NEU Nor. | 124 | 122 | 107 | 117 | 120
  WBC Abn. | 20 | 18 | 25 | 14 | 20
  WBC Nor. | 118 | 122 | 106 | 119 | 115

30. Secondary Outcome: Number of Subjects Having Normal and Abnormal Levels of WBC, NEU, LYM, MON, EOS, BAS, CRP, and CPK.
Description: Subjects were assessed with regard to their normal (Nor.) and abnormal (Abn.) levels for the above parameters of white blood cells (WBC), neutrophils (NEU), lymphocytes (LYM), monocytes (MON), eosinophils (EOS), basophils (BAS), C-reactive protein (CRP) and creatine phosphokinase (CPK) at the Day 360 baseline versus their status post vaccination (Day 390). This outcome measure concerns solely subjects part of the HLA Subsets 1 & 2 who received the Day 360 booster dose of HBsAg.
Time Frame: At Days 360 and 390.
Population: Analysis was done on the Booster Total Vaccinated cohort which included all HLA Subsets 1 and 2 subjects who received the booster dose of HBsAg.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK223192A 1 - HLA Subsets Group | GSK223192A 2 - HLA Subsets Group | GSK223192A 3 - HLA Subsets Group | Fendrix - HLA Subsets Group | Engerix-B - HLA Subsets Group
Number analyzed (Participants) | 59 | 56 | 56 | 54 | 54
Participants
  BAS Abn. Day 360 - Abn. Day 390: number analyzed (Participants) | 3 | 4 | 2 | 1 | 2
  BAS Abn. Day 360 - Abn. Day 390 | 2 | 1 | 0 | 0 | 1
  BAS Abn. Day 360 - Nor. Day 390: number analyzed (Participants) | 3 | 4 | 2 | 1 | 2
  BAS Abn. Day 360 - Nor. Day 390 | 1 | 3 | 2 | 1 | 1
  BAS Nor. Day 360 - Abn. Day 390: number analyzed (Participants) | 56 | 52 | 54 | 53 | 52
  BAS Nor. Day 360 - Abn. Day 390 | 1 | 1 | 4 | 1 | 2
  BAS Nor. Day 360 - Nor. Day 390: number analyzed (Participants) | 56 | 52 | 54 | 53 | 52
  BAS Nor. Day 360 - Nor. Day 390 | 55 | 51 | 50 | 52 | 50
  CPK Abn. Day 360 - Abn. Day 390: number analyzed (Participants) | 15 | 4 | 11 | 6 | 6
  CPK Abn. Day 360 - Abn. Day 390 | 10 | 0 | 4 | 3 | 5
  CPK Abn. Day 360 - Nor. Day 390: number analyzed (Participants) | 15 | 4 | 11 | 6 | 6
  CPK Abn. Day 360 - Nor. Day 390 | 5 | 4 | 7 | 3 | 1
  CPK Nor. Day 360 - Abn. Day 390: number analyzed (Participants) | 44 | 52 | 45 | 49 | 47
  CPK Nor. Day 360 - Abn. Day 390 | 5 | 2 | 7 | 10 | 1
  CPK Nor. Day 360 - Nor. Day 390: number analyzed (Participants) | 44 | 52 | 45 | 49 | 47
  CPK Nor. Day 360 - Nor. Day 390 | 39 | 50 | 38 | 39 | 46
  EOS Abn. Day 360 - Abn. Day 390: number analyzed (Participants) | 2 | 2 | 2 | 4 | 0
  EOS Abn. Day 360 - Abn. Day 390 | 0 | 1 | 1 | 3 | 0
  EOS Abn. Day 360 - Nor. Day 390: number analyzed (Participants) | 2 | 2 | 2 | 4 | 0
  EOS Abn. Day 360 - Nor. Day 390 | 2 | 1 | 1 | 1 | 0
  EOS Nor. Day 360 - Abn. Day 390: number analyzed (Participants) | 57 | 54 | 54 | 50 | 54
  EOS Nor. Day 360 - Abn. Day 390 | 1 | 3 | 1 | 0 | 1
  EOS Nor. Day 360 - Nor. Day 390: number analyzed (Participants) | 57 | 54 | 54 | 50 | 54
  EOS Nor. Day 360 - Nor. Day 390 | 56 | 51 | 53 | 50 | 53
  LYM Abn. Day 360 - Abn. Day 390: number analyzed (Participants) | 9 | 5 | 8 | 4 | 7
  LYM Abn. Day 360 - Abn. Day 390 | 5 | 2 | 5 | 4 | 5
  LYM Abn. Day 360 - Nor. Day 390: number analyzed (Participants) | 9 | 5 | 8 | 4 | 7
  LYM Abn. Day 360 - Nor. Day 390 | 4 | 3 | 3 | 0 | 2
  LYM Nor. Day 360 - Abn. Day 390: number analyzed (Participants) | 50 | 51 | 48 | 50 | 47
  LYM Nor. Day 360 - Abn. Day 390 | 3 | 3 | 1 | 3 | 1
  LYM Nor. Day 360 - Nor. Day 390: number analyzed (Participants) | 50 | 51 | 48 | 50 | 47
  LYM Nor. Day 360 - Nor. Day 390 | 47 | 48 | 47 | 47 | 46
  MON Abn. Day 360 - Abn. Day 390: number analyzed (Participants) | 1 | 1 | 3 | 3 | 1
  MON Abn. Day 360 - Abn. Day 390 | 0 | 1 | 1 | 2 | 0
  MON Abn. Day 360 - Nor. Day 390: number analyzed (Participants) | 1 | 1 | 3 | 3 | 1
  MON Abn. Day 360 - Nor. Day 390 | 1 | 0 | 2 | 1 | 1
  MON Nor. Day 360 - Abn. Day 390: number analyzed (Participants) | 58 | 55 | 53 | 51 | 53
  MON Nor. Day 360 - Abn. Day 390 | 2 | 1 | 1 | 2 | 0
  MON Nor. Day 360 - Nor. Day 390: number analyzed (Participants) | 58 | 55 | 53 | 51 | 53
  MON Nor. Day 360 - Nor. Day 390 | 56 | 54 | 52 | 49 | 53
  NEU Abn. Day 360 - Abn. Day 390: number analyzed (Participants) | 8 | 4 | 5 | 4 | 3
  NEU Abn. Day 360 - Abn. Day 390 | 4 | 0 | 2 | 2 | 0
  NEU Abn. Day 360 - Nor. Day 390: number analyzed (Participants) | 8 | 4 | 5 | 4 | 3
  NEU Abn. Day 360 - Nor. Day 390 | 4 | 4 | 3 | 2 | 3
  NEU Nor. Day 360 - Abn. Day 390: number analyzed (Participants) | 51 | 52 | 51 | 50 | 51
  NEU Nor. Day 360 - Abn. Day 390 | 4 | 2 | 0 | 3 | 2
  NEU Nor. Day 360 - Nor. Day 390: number analyzed (Participants) | 51 | 52 | 51 | 50 | 51
  NEU Nor. Day 360 - Nor. Day 390 | 47 | 50 | 51 | 47 | 49
  WBC Abn. Day 360 - Abn. Day 390: number analyzed (Participants) | 9 | 3 | 8 | 2 | 5
  WBC Abn. Day 360 - Abn. Day 390 | 3 | 1 | 4 | 1 | 2
  WBC Abn. Day 360 - Nor. Day 390: number analyzed (Participants) | 9 | 3 | 8 | 2 | 5
  WBC Abn. Day 360 - Nor. Day 390 | 6 | 2 | 4 | 1 | 3
  WBC Nor. Day 360 - Abn. Day 390: number analyzed (Participants) | 50 | 53 | 48 | 52 | 49
  WBC Nor. Day 360 - Abn. Day 390 | 6 | 2 | 2 | 2 | 2
  WBC Nor. Day 360 - Nor. Day 390: number analyzed (Participants) | 50 | 53 | 48 | 52 | 49
  WBC Nor. Day 360 - Nor. Day 390 | 44 | 51 | 46 | 50 | 47

31. Secondary Outcome: Number of Subjects With Normal and Abnormal Levels of Red Blood Cells, Platelets, Haemoglobin, Alanine Aminotransferase, Aspartate Aminotransferase, Serum Creatinine, Urea and Lactate Dehydrogenase
Description: Subjects were assessed with regard to their normal (Nor.) and abnormal (Abn.) levels for the above parameters of red blood cells (RBC), platelets (PLA), haemoglobin (HGB), alanine aminotransferase (ALT), aspartate aminotransferase (AST), serum creatinine (S-CREA), urea and lactate dehydrogenase (LDH) at the Day 0 baseline versus their status post vaccination (Day 60).
Time Frame: At Day 0 and up to Day 60.
Population: as for outcome 20
Measure: Count of Participants; unit: Participants
Arm/Group | GSK223192A 1 Group | GSK223192A 2 Group | GSK223192A 3 Group | Fendrix Group | Engerix-B Group
Number analyzed (Participants) | 141 | 141 | 138 | 141 | 139
Participants
  ALT Abn. Day 0 - Abn. Day 60: number analyzed (Participants) | 16 | 14 | 13 | 13 | 17
  ALT Abn. Day 0 - Abn. Day 60 | 15 | 10 | 9 | 6 | 12
  ALT Abn. Day 0 - Nor. Day 60: number analyzed (Participants) | 16 | 14 | 13 | 13 | 17
  ALT Abn. Day 0 - Nor. Day 60 | 1 | 4 | 4 | 7 | 5
  ALT Nor. Day 0 - Abn. Day 60: number analyzed (Participants) | 125 | 127 | 125 | 128 | 122
  ALT Nor. Day 0 - Abn. Day 60 | 12 | 5 | 10 | 8 | 9
  ALT Nor. Day 0 - Nor. Day 60: number analyzed (Participants) | 125 | 127 | 125 | 128 | 122
  ALT Nor. Day 0 - Nor. Day 60 | 113 | 122 | 115 | 120 | 113
  AST Abn. Day 0 - Abn. Day 60: number analyzed (Participants) | 4 | 4 | 3 | 4 | 5
  AST Abn. Day 0 - Abn. Day 60 | 4 | 3 | 1 | 1 | 3
  AST Abn. Day 0 - Nor. Day 60: number analyzed (Participants) | 4 | 4 | 3 | 4 | 5
  AST Abn. Day 0 - Nor. Day 60 | 0 | 1 | 2 | 3 | 2
  AST Nor. Day 0 - Abn. Day 60: number analyzed (Participants) | 137 | 137 | 135 | 137 | 134
  AST Nor. Day 0 - Abn. Day 60 | 12 | 1 | 7 | 8 | 6
  AST Nor. Day 0 - Nor. Day 60: number analyzed (Participants) | 137 | 137 | 135 | 137 | 134
  AST Nor. Day 0 - Nor. Day 60 | 125 | 136 | 128 | 129 | 128
  HGB Abn. Day 0 - Abn. Day 60: number analyzed (Participants) | 19 | 15 | 12 | 13 | 13
  HGB Abn. Day 0 - Abn. Day 60 | 15 | 9 | 8 | 11 | 9
  HGB Abn. Day 0 - Nor. Day 60: number analyzed (Participants) | 19 | 15 | 12 | 13 | 13
  HGB Abn. Day 0 - Nor. Day 60 | 4 | 6 | 4 | 2 | 4
  HGB Nor. Day 0 - Abn. Day 60: number analyzed (Participants) | 122 | 126 | 126 | 128 | 126
  HGB Nor. Day 0 - Abn. Day 60 | 10 | 13 | 11 | 9 | 16
  HGB Nor. Day 0 - Nor. Day 60: number analyzed (Participants) | 122 | 126 | 126 | 128 | 126
  HGB Nor. Day 0 - Nor. Day 60 | 112 | 113 | 115 | 119 | 110
  LDH Abn. Day 0 - Abn. Day 60: number analyzed (Participants) | 11 | 8 | 6 | 8 | 9
  LDH Abn. Day 0 - Abn. Day 60 | 10 | 7 | 5 | 2 | 8
  LDH Abn. Day 0 - Nor. Day 60: number analyzed (Participants) | 11 | 8 | 6 | 8 | 9
  LDH Abn. Day 0 - Nor. Day 60 | 1 | 1 | 1 | 6 | 1
  LDH Nor. Day 0 - Abn. Day 60: number analyzed (Participants) | 130 | 132 | 132 | 133 | 130
  LDH Nor. Day 0 - Abn. Day 60 | 11 | 9 | 6 | 9 | 9
  LDH Nor. Day 0 - Nor. Day 60: number analyzed (Participants) | 130 | 132 | 132 | 133 | 130
  LDH Nor. Day 0 - Nor. Day 60 | 119 | 123 | 126 | 124 | 121
  PLA Abn. Day 0 - Abn. Day 60: number analyzed (Participants) | 10 | 8 | 6 | 11 | 8
  PLA Abn. Day 0 - Abn. Day 60 | 9 | 8 | 6 | 8 | 7
  PLA Abn. Day 0 - Nor. Day 60: number analyzed (Participants) | 10 | 8 | 6 | 11 | 8
  PLA Abn. Day 0 - Nor. Day 60 | 1 | 0 | 0 | 3 | 1
  PLA Nor. Day 0 - Abn. Day 60: number analyzed (Participants) | 131 | 133 | 132 | 130 | 131
  PLA Nor. Day 0 - Abn. Day 60 | 9 | 11 | 10 | 8 | 5
  PLA Nor. Day 0 - Nor. Day 60: number analyzed (Participants) | 131 | 133 | 132 | 130 | 131
  PLA Nor. Day 0 - Nor. Day 60 | 122 | 122 | 122 | 122 | 126
  RBC Abn. Day 0 - Abn. Day 60: number analyzed (Participants) | 7 | 13 | 8 | 6 | 9
  RBC Abn. Day 0 - Abn. Day 60 | 5 | 9 | 2 | 2 | 4
  RBC Abn. Day 0 - Nor. Day 60: number analyzed (Participants) | 7 | 13 | 8 | 6 | 9
  RBC Abn. Day 0 - Nor. Day 60 | 2 | 4 | 6 | 4 | 5
  RBC Nor. Day 0 - Abn. Day 60: number analyzed (Participants) | 134 | 128 | 130 | 135 | 130
  RBC Nor. Day 0 - Abn. Day 60 | 7 | 12 | 17 | 14 | 6
  RBC Nor. Day 0 - Nor. Day 60: number analyzed (Participants) | 134 | 128 | 130 | 135 | 130
  RBC Nor. Day 0 - Nor. Day 60 | 127 | 116 | 113 | 121 | 124
  S-CREA Abn. Day 0 - Abn. Day 60: number analyzed (Participants) | 5 | 6 | 7 | 7 | 15
  S-CREA Abn. Day 0 - Abn. Day 60 | 4 | 3 | 4 | 6 | 12
  S-CREA Abn. Day 0 - Nor. Day 60: number analyzed (Participants) | 5 | 6 | 7 | 7 | 15
  S-CREA Abn. Day 0 - Nor. Day 60 | 1 | 3 | 3 | 1 | 3
  S-CREA Nor. Day 0 - Abn. Day 60: number analyzed (Participants) | 136 | 135 | 131 | 134 | 124
  S-CREA Nor. Day 0 - Abn. Day 60 | 8 | 8 | 7 | 12 | 5
  S-CREA Nor. Day 0 - Nor. Day 60: number analyzed (Participants) | 136 | 135 | 131 | 134 | 124
  S-CREA Nor. Day 0 - Nor. Day 60 | 128 | 127 | 124 | 122 | 119
  UREA Abn. Day 0 - Abn. Day 60: number analyzed (Participants) | 6 | 3 | 9 | 11 | 6
  UREA Abn. Day 0 - Abn. Day 60 | 2 | 2 | 4 | 8 | 3
  UREA Abn. Day 0 - Nor. Day 60: number analyzed (Participants) | 6 | 3 | 9 | 11 | 6
  UREA Abn. Day 0 - Nor. Day 60 | 4 | 1 | 5 | 3 | 3
  UREA Nor. Day 0 - Abn. Day 60: number analyzed (Participants) | 135 | 138 | 129 | 130 | 133
  UREA Nor. Day 0 - Abn. Day 60 | 18 | 11 | 16 | 14 | 8
  UREA Nor. Day 0 - Nor. Day 60: number analyzed (Participants) | 135 | 138 | 129 | 130 | 133
  UREA Nor. Day 0 - Nor. Day 60 | 117 | 127 | 113 | 116 | 125

32. Secondary Outcome: Number of Subjects With Normal and Abnormal Levels of RBC, PLA, HGB, ALT, AST, S-CREA, Urea and LDH
Description: Subjects were assessed with regard to their normal (Nor.) and abnormal (Abn.) levels for the above parameters of red blood cells (RBC), platelets (PLA), haemoglobin (HGB), alanine aminotransferase (ALT), aspartate aminotransferase (AST), serum creatinine (S-CREA), urea and lactate dehydrogenase (LDH) at the Day 0 baseline versus their status post vaccination (Day 180 or 360). Day 180 or 360 results were chosen based on assessment of grading of the abnormality observed, with results for higher grading being tabulated.
Time Frame: post vaccination (up to Day 360).
Population: as for outcome 20
Measure: Count of Participants; unit: Participants
Arm/Group | GSK223192A 1 Group | GSK223192A 2 Group | GSK223192A 3 Group | Fendrix Group | Engerix-B Group
Number analyzed (Participants) | 138 | 140 | 131 | 133 | 135
Participants
  ALT Abn. | 26 | 17 | 18 | 23 | 17
  ALT Nor. | 112 | 123 | 113 | 110 | 118
  AST Abn. | 11 | 5 | 9 | 5 | 9
  AST Nor. | 127 | 135 | 122 | 128 | 126
  HGB Abn. | 24 | 13 | 12 | 17 | 15
  HGB Nor. | 114 | 127 | 119 | 116 | 120
  LDH Abn. | 10 | 14 | 10 | 4 | 11
  LDH Nor. | 128 | 126 | 121 | 129 | 124
  PLA Abn. | 11 | 9 | 7 | 13 | 10
  PLA Nor. | 127 | 131 | 124 | 120 | 125
  RBC Abn. | 15 | 20 | 16 | 7 | 12
  RBC Nor. | 123 | 120 | 115 | 126 | 123
  S-CREA Abn. | 11 | 11 | 12 | 9 | 18
  S-CREA Nor. | 127 | 129 | 119 | 124 | 117
  UREA Abn. | 11 | 14 | 19 | 17 | 8
  UREA Nor. | 127 | 126 | 112 | 116 | 127

33. Secondary Outcome: Number of Subjects Presenting Normal and Abnormal Levels of Red Blood Cells, Platelets, Haemoglobin, Alanine Aminotransferase, Aspartate Aminotransferase, Serum Creatinine, Urea and Lactate Dehydrogenase
Description: Subjects were assessed with regard to their normal (Nor.) and abnormal (Abn.) levels for the above parameters of red blood cells (RBC), platelets (PLA), haemoglobin (HGB), alanine aminotransferase (ALT), aspartate aminotransferase (AST), serum creatinine (S-CREA), urea and lactate dehydrogenase (LDH) at the Day 360 baseline versus their status post vaccination (Day 390). This outcome measure concerns solely subjects part of the HLA Subsets 1 & 2 who received the Day 360 booster dose of HBsAg.
Time Frame: At Days 360 and 390.
Population: as for outcome 30
Measure: Count of Participants; unit: Participants
Arm/Group | GSK223192A 1 - HLA Subsets Group | GSK223192A 2 - HLA Subsets Group | GSK223192A 3 - HLA Subsets Group | Fendrix - HLA Subsets Group | Engerix-B - HLA Subsets Group
Number analyzed (Participants) | 59 | 56 | 54 | 55 | 53
Participants
  ALT Abn. Day 360 - Abn. Day 390: number analyzed (Participants) | 7 | 3 | 10 | 5 | 4
  ALT Abn. Day 360 - Abn. Day 390 | 4 | 2 | 6 | 3 | 3
  ALT Abn. Day 360 - Nor. Day 390: number analyzed (Participants) | 7 | 3 | 10 | 5 | 4
  ALT Abn. Day 360 - Nor. Day 390 | 3 | 1 | 4 | 2 | 1
  ALT Nor. Day 360 - Abn. Day 390: number analyzed (Participants) | 52 | 53 | 46 | 50 | 49
  ALT Nor. Day 360 - Abn. Day 390 | 1 | 2 | 0 | 5 | 0
  ALT Nor. Day 360 - Nor. Day 390: number analyzed (Participants) | 52 | 53 | 46 | 50 | 49
  ALT Nor. Day 360 - Nor. Day 390 | 51 | 51 | 46 | 45 | 49
  AST Abn. Day 360 - Abn. Day 390: number analyzed (Participants) | 4 | 0 | 4 | 0 | 1
  AST Abn. Day 360 - Abn. Day 390 | 2 | 0 | 1 | 0 | 0
  AST Abn. Day 360 - Nor. Day 390: number analyzed (Participants) | 4 | 0 | 4 | 0 | 1
  AST Abn. Day 360 - Nor. Day 390 | 2 | 0 | 3 | 0 | 1
  AST Nor. Day 360 - Abn. Day 390: number analyzed (Participants) | 55 | 56 | 52 | 55 | 52
  AST Nor. Day 360 - Abn. Day 390 | 3 | 2 | 1 | 4 | 1
  AST Nor. Day 360 - Nor. Day 390: number analyzed (Participants) | 55 | 56 | 52 | 55 | 52
  AST Nor. Day 360 - Nor. Day 390 | 52 | 54 | 51 | 51 | 51
  HGB Abn. Day 360 - Abn. Day 390: number analyzed (Participants) | 4 | 3 | 2 | 4 | 5
  HGB Abn. Day 360 - Abn. Day 390 | 2 | 2 | 2 | 3 | 4
  HGB Abn. Day 360 - Nor. Day 390: number analyzed (Participants) | 4 | 3 | 2 | 4 | 5
  HGB Abn. Day 360 - Nor. Day 390 | 2 | 1 | 0 | 1 | 1
  HGB Nor. Day 360 - Abn. Day 390: number analyzed (Participants) | 55 | 53 | 54 | 50 | 49
  HGB Nor. Day 360 - Abn. Day 390 | 2 | 0 | 1 | 2 | 2
  HGB Nor. Day 360 - Nor. Day 390: number analyzed (Participants) | 55 | 53 | 54 | 50 | 49
  HGB Nor. Day 360 - Nor. Day 390 | 53 | 53 | 53 | 48 | 47
  LDH Abn. Day 360 - Abn. Day 390: number analyzed (Participants) | 4 | 1 | 3 | 0 | 2
  LDH Abn. Day 360 - Abn. Day 390 | 2 | 1 | 0 | 0 | 1
  LDH Abn. Day 360 - Nor. Day 390: number analyzed (Participants) | 4 | 1 | 3 | 0 | 2
  LDH Abn. Day 360 - Nor. Day 390 | 2 | 0 | 3 | 0 | 1
  LDH Nor. Day 360 - Abn. Day 390: number analyzed (Participants) | 55 | 55 | 53 | 55 | 51
  LDH Nor. Day 360 - Abn. Day 390 | 1 | 0 | 2 | 3 | 0
  LDH Nor. Day 360 - Nor. Day 390: number analyzed (Participants) | 55 | 55 | 53 | 55 | 51
  LDH Nor. Day 360 - Nor. Day 390 | 54 | 55 | 51 | 52 | 51
  PLA Abn. Day 360 - Abn. Day 390: number analyzed (Participants) | 4 | 1 | 2 | 5 | 4
  PLA Abn. Day 360 - Abn. Day 390 | 3 | 0 | 0 | 3 | 4
  PLA Abn. Day 360 - Nor. Day 390: number analyzed (Participants) | 4 | 1 | 2 | 5 | 4
  PLA Abn. Day 360 - Nor. Day 390 | 1 | 1 | 2 | 2 | 0
  PLA Nor. Day 360 - Abn. Day 390: number analyzed (Participants) | 55 | 55 | 54 | 49 | 50
  PLA Nor. Day 360 - Abn. Day 390 | 3 | 0 | 1 | 1 | 0
  PLA Nor. Day 360 - Nor. Day 390: number analyzed (Participants) | 55 | 55 | 54 | 49 | 50
  PLA Nor. Day 360 - Nor. Day 390 | 52 | 55 | 53 | 48 | 50
  RBC Abn. Day 360 - Abn. Day 390: number analyzed (Participants) | 2 | 4 | 3 | 3 | 4
  RBC Abn. Day 360 - Abn. Day 390 | 1 | 2 | 1 | 1 | 4
  RBC Abn. Day 360 - Nor. Day 390: number analyzed (Participants) | 2 | 4 | 3 | 3 | 4
  RBC Abn. Day 360 - Nor. Day 390 | 1 | 2 | 2 | 2 | 0
  RBC Nor. Day 360 - Abn. Day 390: number analyzed (Participants) | 57 | 52 | 53 | 51 | 50
  RBC Nor. Day 360 - Abn. Day 390 | 2 | 1 | 3 | 3 | 0
  RBC Nor. Day 360 - Nor. Day 390: number analyzed (Participants) | 57 | 52 | 53 | 51 | 50
  RBC Nor. Day 360 - Nor. Day 390 | 55 | 51 | 50 | 48 | 50
  S-CREA Abn. Day 360 - Abn. Day 390: number analyzed (Participants) | 0 | 0 | 3 | 2 | 4
  S-CREA Abn. Day 360 - Abn. Day 390 | 0 | 0 | 2 | 1 | 3
  S-CREA Abn. Day 360 - Nor. Day 390: number analyzed (Participants) | 0 | 0 | 3 | 2 | 4
  S-CREA Abn. Day 360 - Nor. Day 390 | 0 | 0 | 1 | 1 | 1
  S-CREA Nor. Day 360 - Abn. Day 390: number analyzed (Participants) | 59 | 56 | 53 | 53 | 49
  S-CREA Nor. Day 360 - Abn. Day 390 | 1 | 0 | 0 | 3 | 2
  S-CREA Nor. Day 360 - Nor. Day 390: number analyzed (Participants) | 59 | 56 | 53 | 53 | 49
  S-CREA Nor. Day 360 - Nor. Day 390 | 58 | 56 | 53 | 50 | 47
  UREA Abn. Day 360 - Abn. Day 390: number analyzed (Participants) | 3 | 4 | 7 | 5 | 4
  UREA Abn. Day 360 - Abn. Day 390 | 2 | 0 | 2 | 1 | 1
  UREA Abn. Day 360 - Nor. Day 390: number analyzed (Participants) | 3 | 4 | 7 | 5 | 4
  UREA Abn. Day 360 - Nor. Day 390 | 1 | 4 | 5 | 4 | 3
  UREA Nor. Day 360 - Abn. Day 390: number analyzed (Participants) | 56 | 52 | 49 | 50 | 49
  UREA Nor. Day 360 - Abn. Day 390 | 1 | 4 | 2 | 0 | 1
  UREA Nor. Day 360 - Nor. Day 390: number analyzed (Participants) | 56 | 52 | 49 | 50 | 49
  UREA Nor. Day 360 - Nor. Day 390 | 55 | 48 | 47 | 50 | 48

34. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Solicited Local Symptoms Following Primary Vaccination.
Description: Solicited local symptoms assessed were pain, redness and swelling. All solicited local symptoms were considered as related to study vaccination. Any = occurrence of any local symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling above (>) 50 millimeters (mm). Occurrence of a solicited local symptoms collected post-vaccination was a priori considered as related to vaccination.
Time Frame: Within the 14-day (Days 0-13) follow up period following primary vaccination with the GSK223192A, Fendrix™ or Engerix-B™ vaccines.
Population: Analysis was done on the Total Vaccinated cohort which included all vaccinated subjects, with analysis performed solely on subjects with results from post-primary vaccination available.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK223192A 1 Group | GSK223192A 2 Group | GSK223192A 3 Group | Fendrix Group | Engerix-B Group
Number analyzed (Participants) | 142 | 140 | 138 | 143 | 139
Participants
  Any Pain | 134 | 129 | 123 | 128 | 70
  Grade 3 Pain | 9 | 5 | 2 | 6 | 0
  Any Redness | 71 | 39 | 35 | 53 | 23
  Redness > 50 mm | 11 | 2 | 0 | 0 | 0
  Any Swelling | 46 | 36 | 34 | 43 | 16
  Swelling > 50 mm | 9 | 3 | 2 | 2 | 0

35. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Solicited General Symptoms Following Primary Vaccination.
Description: Solicited general symptoms assessed were Fatigue, Fever - oral temperature equal to or above (>=) 37.5 degrees Celsius (°C) -, Gastrointestinal symptoms (Gastr.), Headache, Malaise and Myalgia. Any = occurrence of a general symptom regardless of its intensity grade or relationship to vaccination. Related = occurrence of a general symptom assessed by the investigator to be causally related to vaccination. Grade 3 fever = oral temperature above (>) 39.0 °C. Grade 3 for Gastr., Headache, Malaise and Myalgia = occurrence of the specified solicited general symptom which prevented normal activity.
Time Frame: Within the 14-day (Days 0-13) follow up period following primary vaccination with the GSK223192A, Fendrix™ or Engerix-B™ vaccine.
Population: as for outcome 34
Measure: Count of Participants; unit: Participants
Arm/Group | GSK223192A 1 Group | GSK223192A 2 Group | GSK223192A 3 Group | Fendrix Group | Engerix-B Group
Number analyzed (Participants) | 142 | 140 | 138 | 144 | 139
Participants
  Any Fatigue | 91 | 76 | 67 | 70 | 62
  Grade 3 Fatigue | 5 | 5 | 5 | 4 | 3
  Related Fatigue | 83 | 67 | 57 | 55 | 42
  Any Fever | 45 | 23 | 24 | 12 | 17
  Grade 3 Fever | 1 | 0 | 1 | 0 | 1
  Related Fever | 42 | 17 | 17 | 6 | 5
  Any Gastr. | 30 | 27 | 29 | 36 | 35
  Grade 3 Gastr. | 2 | 5 | 5 | 4 | 7
  Related Gastr. | 21 | 13 | 19 | 20 | 19
  Any Headache | 90 | 67 | 66 | 62 | 59
  Grade 3 Headache | 8 | 6 | 8 | 3 | 5
  Related Headache | 74 | 52 | 46 | 41 | 35
  Any Malaise | 60 | 44 | 39 | 35 | 28
  Grade 3 Malaise | 9 | 5 | 4 | 4 | 2
  Related Malaise | 53 | 36 | 30 | 27 | 16
  Any Myalgia | 85 | 57 | 55 | 58 | 34
  Grade 3 Myalgia | 10 | 4 | 3 | 2 | 2
  Related Myalgia | 79 | 49 | 47 | 50 | 22

36. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Solicited Local Symptoms Following Booster Vaccination.
Description: Solicited local symptoms assessed were pain, redness and swelling. All solicited local symptoms were considered as related to study vaccination. Any = occurrence of any local symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling above (>) 50 millimeters (mm). Occurrence of a solicited local symptoms collected post-vaccination was a priori considered as related to vaccination. This outcome measure concerns solely subjects part of the HLA Subsets 1 & 2 who received the Day 360 booster dose of HBsAg.
Time Frame: Within the 7-day (Days 0-6) follow up period following booster vaccination with HBsAg antigens
Population: Analysis was done on the Booster Total Vaccinated cohort which included all HLA Subsets 1 and 2 subjects who received the booster dose of HBsAg, on subjects for whom results were available for the timepoint/outcome analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK223192A 1 - HLA Subsets Group | GSK223192A 2 - HLA Subsets Group | GSK223192A 3 - HLA Subsets Group | Fendrix - HLA Subsets Group | Engerix-B - HLA Subsets Group
Number analyzed (Participants) | 59 | 56 | 56 | 56 | 54
Participants
  Any Pain | 19 | 19 | 13 | 16 | 10
  Grade 3 Pain | 0 | 0 | 1 | 0 | 0
  Any Redness | 6 | 3 | 8 | 6 | 2
  Redness > 50 mm | 1 | 0 | 0 | 0 | 0
  Any Swelling | 3 | 4 | 2 | 5 | 1
  Swelling > 50 mm | 1 | 0 | 0 | 0 | 0

37. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Solicited General Symptoms Following Booster Vaccination.
Description: Solicited general symptoms assessed were Fatigue, Fever - oral temperature equal to or above (>=) 37.5 degrees Celsius (°C) -, Gastrointestinal symptoms (Gastr.), Headache, Malaise and Myalgia. Any = occurrence of a general symptom regardless of its intensity grade or relationship to vaccination. Related = occurrence of a general symptom assessed by the investigator to be causally related to vaccination. Grade 3 fever = oral temperature above (>) 39.0 °C. Grade 3 for Gastr., Headache, Malaise and Myalgia = occurrence of the specified solicited general symptom which prevented normal activity. This outcome measure concerns solely subjects part of the HLA Subsets 1 & 2 who received the Day 360 booster dose of HBsAg.
Time Frame: Within the 7-day (Days 0-6) follow up period following booster vaccination with HBsAg antigens
Population: as for outcome 36
Measure: Count of Participants; unit: Participants
Arm/Group | GSK223192A 1 - HLA Subsets Group | GSK223192A 2 - HLA Subsets Group | GSK223192A 3 - HLA Subsets Group | Fendrix - HLA Subsets Group | Engerix-B - HLA Subsets Group
Number analyzed (Participants) | 59 | 56 | 56 | 56 | 54
Participants
  Any Fatigue | 15 | 14 | 7 | 15 | 12
  Grade 3 Fatigue | 0 | 0 | 0 | 0 | 1
  Related Fatigue | 15 | 12 | 5 | 13 | 10
  Any Fever | 3 | 1 | 0 | 3 | 1
  Grade 3 Fever | 0 | 0 | 0 | 0 | 0
  Related Fever | 1 | 1 | 0 | 2 | 1
  Any Gastr. | 4 | 5 | 4 | 3 | 5
  Grade 3 Gastr. | 0 | 0 | 0 | 0 | 0
  Related Gastr. | 4 | 5 | 2 | 2 | 3
  Any Headache | 15 | 7 | 7 | 8 | 14
  Grade 3 Headache | 0 | 0 | 0 | 1 | 0
  Related Headache | 13 | 5 | 6 | 7 | 9
  Any Malaise | 6 | 5 | 2 | 4 | 4
  Grade 3 Malaise | 0 | 0 | 0 | 0 | 0
  Related Malaise | 6 | 4 | 2 | 4 | 4
  Any Myalgia | 4 | 3 | 2 | 5 | 1
  Grade 3 Myalgia | 0 | 0 | 0 | 0 | 1
  Related Myalgia | 4 | 2 | 2 | 5 | 1

38. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and/or Related Unsolicited Adverse Events (AEs) Following Primary Vaccination
Description: An unsolicited AE was defined as an untoward medical occurrence in a patient or clinical investigation subject, temporally associated with use of a medicinal product, whether or not considered related to the medicinal product reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any = occurrence of an AE regardless of intensity grade or relationship to study vaccination. Grade 3 = occurrence of an AE that prevented normal activity. Related = occurrence of an AE assessed by the investigators as causally related to the study vaccine.
Time Frame: Within the 31-day (Days 0-30) follow up period following primary vaccination with the GSK223192A, Fendrix™ or Engerix-B™ vaccine
Population: Analysis was done on the Total Vaccinated cohort which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK223192A 1 Group | GSK223192A 2 Group | GSK223192A 3 Group | Fendrix Group | Engerix-B Group
Number analyzed (Participants) | 143 | 142 | 141 | 145 | 142
Participants
  Subjects with any AE(s) | 80 | 73 | 76 | 67 | 71
  Subjects with Grade 3 AE(s) | 17 | 11 | 12 | 19 | 15
  Subjects with related AE(s) | 32 | 19 | 27 | 21 | 19
  Subjects with Grade 3 and related AE(s) | 7 | 1 | 2 | 1 | 2

39. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and/or Related Unsolicited Adverse Events (AEs) Following Booster Vaccination
Description: An unsolicited AE was defined as an untoward medical occurrence in a patient or clinical investigation subject, temporally associated with use of a medicinal product, whether or not considered related to the medicinal product reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any = occurrence of an AE regardless of intensity grade or relationship to study vaccination. Grade 3 = occurrence of an AE that prevented normal activity. Related = occurrence of an AE assessed by the investigators as causally related to the study vaccine. This outcome measure concerns solely subjects part of the HLA Subsets 1 & 2 who received the Day 360 booster dose of HBsAg.
Time Frame: Within the 31-day (Days 0-30) follow up period following booster vaccination with HBsAg antigens
Population: as for outcome 30
Measure: Count of Participants; unit: Participants
Arm/Group | GSK223192A 1 - HLA Subsets Group | GSK223192A 2 - HLA Subsets Group | GSK223192A 3 - HLA Subsets Group | Fendrix - HLA Subsets Group | Engerix-B - HLA Subsets Group
Number analyzed (Participants) | 59 | 56 | 56 | 56 | 54
Participants
  Subjects with any AE(s) | 12 | 8 | 9 | 14 | 10
  Subjects with any grade 3 AE(s) | 2 | 2 | 2 | 4 | 1
  Subjects with related AE(s) | 3 | 1 | 0 | 2 | 2
  Subjects with Grade 3 and related AE(s) | 0 | 0 | 0 | 0 | 0

40. Secondary Outcome: Number of Subjects Reporting Any and Related Adverse Events of Specific Interest (AESIs)
Description: AESIs included Autoimmune Disease (AID), neurological/demyelinating events, rheumatic and connective diseases, autoimmune endocrine diseases, inflammatory bowel diseases, autoimmune blood disorders, inflammatory skin disorders, and other autoimmune/inflammatory events. Any AESI(s) = occurrence of any AESI(s) in a subject regardless of assessment of relationship to study vaccination. Related AESI(s) = Occurrence of AESI(s) in a subject assessed by the investigator as causally related to the study vaccination.
Time Frame: During the entire study period, from Day 0 to study end, at Day 360 for subjects not in Subsets 1 & 2 and at Day 390 for subjects in Subsets 1 & 2.
Population: Analysis was done on the Total Vaccinated cohort which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK223192A 1 Group | GSK223192A 2 Group | GSK223192A 3 Group | Fendrix Group | Engerix-B Group
Number analyzed (Participants) | 143 | 142 | 141 | 145 | 142
Participants
  Any AESI(s) | 0 | 1 | 0 | 0 | 0
  Related AESI(s) | 0 | 0 | 0 | 0 | 0

41. Secondary Outcome: Number of Subjects Reporting Any Serious Adverse Events (SAEs) and SAEs Related to Study Vaccination
Description: A SAE was defined as a medical occurrence that resulted in death, was life-threatening, required hospitalization or prolongation of hospitalization, resulted in disability/incapacity or was a congenital anomaly/birth defect in the offspring of a study subject. Any SAE(s) = occurrence of SAE(s) in a subject regardless of assessment of relationship to study vaccination. Related SAE(s) = occurrence of occurrence of SAE(s) in a subject assessed by the investigators as causally related to the study vaccination.
Time Frame: as for outcome 40
Population: Analysis was done on the Total Vaccinated cohort which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK223192A 1 Group | GSK223192A 2 Group | GSK223192A 3 Group | Fendrix Group | Engerix-B Group
Number analyzed (Participants) | 143 | 142 | 141 | 145 | 142
Participants
  Any SAE(s) | 7 | 4 | 10 | 7 | 7
  Related SAE(s) | 0 | 0 | 0 | 0 | 0

42. Secondary Outcome: Levels of Messenger Ribonucleic Acid (mRNA) as Measured by Quantitative Polymerase Chain Reaction (qPCR)
Description: The analysis of the mRNA levels of 14 target genes was performed using whole blood, in the first 140 subjects from the 2 subsets recruited at the Immune Health (IH) centre in La Louvière, Belgium, by microarray/ Polymerase Chain Reaction (PCR) array/ quantitative PCR. Among the target genes were Tumor Necrosis Factor (TNF), Tumor Necrosis Factor Receptor Superfamily (TNFRSF9).
Time Frame: At Days 0, 1, 14, 30, 31, 33 and 37
Population: The ATP cohort for innate immunogenicity up to Day 60 included all evaluable subjects, who complied with the vaccination schedule, for whom data concerning immunogenicity outcome measures were available and for whom innate immunogenicity data were available for at least one post-vaccination time point.
Measure: Median (Full Range); unit: copies
Arm/Group | GSK223192A 1 Group | GSK223192A 2 Group | GSK223192A 3 Group | Fendrix Group | Engerix-B Group
Number analyzed (Participants) | 18 | 23 | 28 | 22 | 21
copies
  TNF.mRNA, Day 0: number analyzed (Participants) | 17 | 23 | 28 | 21 | 21
  TNF.mRNA, Day 0 | 1.18 [0.55 to 2.66] | 1.09 [0.78 to 1.75] | 1.24 [0.84 to 2.64] | 1.18 [0.78 to 3.18] | 1.18 [0.76 to 2.89]
  TNF.mRNA, Day 1: number analyzed (Participants) | 17 | 23 | 27 | 21 | 21
  TNF.mRNA, Day 1 | 1.33 [0.71 to 2.48] | 1.08 [0.44 to 3.01] | 1.1 [0.4 to 2.58] | 1 [0.56 to 2.39] | 1.06 [0.63 to 2.09]
  TNF.mRNA, Day 14: number analyzed (Participants) | 16 | 23 | 27 | 21 | 21
  TNF.mRNA, Day 14 | 0.95 [0.63 to 2.14] | 1.07 [0.57 to 1.8] | 1 [0.63 to 2.96] | 1.03 [0.62 to 1.58] | 1.13 [0.52 to 1.67]
  TNF.mRNA, Day 30: number analyzed (Participants) | 17 | 22 | 28 | 19 | 21
  TNF.mRNA, Day 30 | 1.03 [0.74 to 1.63] | 1.21 [0.55 to 2.56] | 1.25 [0.58 to 2.89] | 1.19 [0.64 to 2] | 1.09 [0.48 to 2.97]
  TNF.mRNA, Day 31: number analyzed (Participants) | 16 | 22 | 28 | 19 | 21
  TNF.mRNA, Day 31 | 1.31 [0.66 to 2.2] | 1.26 [0.58 to 2.13] | 1.41 [0.5 to 3.42] | 1.15 [0.46 to 2.59] | 1.1 [0.49 to 2.24]
  TNF.mRNA, Day 33: number analyzed (Participants) | 17 | 21 | 28 | 19 | 21
  TNF.mRNA, Day 33 | 0.99 [0.44 to 2.47] | 1.04 [0.67 to 2.1] | 1.12 [0.54 to 2.99] | 1.18 [0.47 to 2.27] | 0.97 [0.57 to 2.48]
  TNF.mRNA, Day 37: number analyzed (Participants) | 17 | 21 | 28 | 17 | 21
  TNF.mRNA, Day 37 | 0.82 [0.36 to 1.56] | 1.04 [0.32 to 1.69] | 1 [0.39 to 2.39] | 1.07 [0.42 to 1.99] | 1.06 [0.38 to 3.39]
  TNFRSF9.mRNA, Day 0: number analyzed (Participants) | 17 | 23 | 28 | 22 | 21
  TNFRSF9.mRNA, Day 0 | 1.04 [0.81 to 2.17] | 1.11 [0.74 to 1.52] | 1.14 [0.7 to 2.64] | 1.14 [0.86 to 2.11] | 1.11 [0.8 to 1.98]
  TNFRSF9.mRNA, Day 1: number analyzed (Participants) | 18 | 23 | 27 | 22 | 21
  TNFRSF9.mRNA, Day 1 | 1.14 [0.74 to 1.67] | 1.14 [0.59 to 2.5] | 1.24 [0.72 to 2.13] | 1.24 [0.73 to 3.19] | 1.01 [0.55 to 1.53]
  TNFRSF9.mRNA, Day 14: number analyzed (Participants) | 18 | 23 | 28 | 21 | 21
  TNFRSF9.mRNA, Day 14 | 0.98 [0.52 to 1.74] | 1.02 [0.52 to 1.97] | 1.19 [0.63 to 3.31] | 1.15 [0.59 to 2.13] | 1.02 [0.46 to 1.69]
  TNFRSF9.mRNA, Day 30: number analyzed (Participants) | 18 | 23 | 28 | 19 | 21
  TNFRSF9.mRNA, Day 30 | 1.06 [0.67 to 1.51] | 1.02 [0.73 to 1.61] | 1.08 [0.78 to 1.89] | 1.03 [0.72 to 1.42] | 1.14 [0.66 to 1.65]
  TNFRSF9.mRNA, Day 31: number analyzed (Participants) | 18 | 23 | 28 | 19 | 20
  TNFRSF9.mRNA, Day 31 | 1.14 [0.8 to 1.98] | 1.09 [0.55 to 1.49] | 1 [0.57 to 1.8] | 0.97 [0.73 to 2.01] | 1.07 [0.68 to 1.75]
  TNFRSF9.mRNA, Day 33: number analyzed (Participants) | 18 | 22 | 28 | 19 | 20
  TNFRSF9.mRNA, Day 33 | 0.67 [0.46 to 2.76] | 0.7 [0.32 to 1.45] | 0.73 [0.49 to 1.7] | 1.12 [0.84 to 1.95] | 1.07 [0.67 to 1.86]
  TNFRSF9.mRNA, Day 37: number analyzed (Participants) | 18 | 22 | 28 | 17 | 21
  TNFRSF9.mRNA, Day 37 | 0.77 [0.41 to 3.06] | 1.01 [0.6 to 1.61] | 0.91 [0.55 to 3.2] | 1.01 [0.59 to 1.78] | 1.14 [0.55 to 2.01]

43. Secondary Outcome: mRNA Levels as Measured by qPCR
Description: The analysis of the mRNA levels of 14 target genes was performed using whole blood, in the first 140 subjects from the 2 subsets recruited at the Immune Health (IH) centre in La Louvière, Belgium, by microarray/ Polymerase Chain Reaction (PCR) array/ quantitative PCR. Among the target genes were Fas associated factor 1 (FAF1), Signal Transducer And Activator Of Transcription 1(STAT1).
Time Frame: At Days 0, 1, 14, 30, 31, 33 and 37
Population: as for outcome 42
Measure: Median (Full Range); unit: copies
Arm/Group | GSK223192A 1 Group | GSK223192A 2 Group | GSK223192A 3 Group | Fendrix Group | Engerix-B Group
Number analyzed (Participants) | 18 | 23 | 28 | 22 | 21
copies
  FAF1.mRNA, Day 0 | 1.08 [0.66 to 1.54] | 1.02 [0.74 to 1.34] | 1.06 [0.72 to 1.39] | 1.06 [0.68 to 1.61] | 1.07 [0.85 to 1.39]
  FAF1.mRNA, Day 1: number analyzed (Participants) | 18 | 23 | 27 | 22 | 21
  FAF1.mRNA, Day 1 | 0.83 [0.66 to 1.04] | 0.88 [0.62 to 1.63] | 0.89 [0.57 to 1.28] | 0.93 [0.71 to 1.29] | 1.08 [0.72 to 1.44]
  FAF1.mRNA, Day 14 | 1.05 [0.69 to 1.32] | 1.06 [0.7 to 1.68] | 0.97 [0.7 to 1.48] | 1 [0.65 to 1.26] | 1.01 [0.75 to 1.3]
  FAF1.mRNA, Day 30: number analyzed (Participants) | 18 | 23 | 28 | 19 | 21
  FAF1.mRNA, Day 30 | 0.93 [0.73 to 1.29] | 1.03 [0.77 to 1.79] | 1.03 [0.77 to 1.58] | 0.99 [0.8 to 1.25] | 1.02 [0.7 to 1.54]
  FAF1.mRNA, Day 31: number analyzed (Participants) | 18 | 23 | 28 | 19 | 21
  FAF1.mRNA, Day 31 | 0.6 [0.46 to 1.09] | 0.67 [0.49 to 1.35] | 0.83 [0.4 to 1.43] | 0.9 [0.66 to 1.46] | 1.02 [0.79 to 1.72]
  FAF1.mRNA, Day 33: number analyzed (Participants) | 18 | 22 | 28 | 19 | 21
  FAF1.mRNA, Day 33 | 0.85 [0.65 to 1.37] | 0.95 [0.72 to 1.23] | 0.94 [0.71 to 1.38] | 1.01 [0.7 to 1.34] | 0.98 [0.54 to 1.89]
  FAF1.mRNA, Day 37: number analyzed (Participants) | 18 | 22 | 28 | 17 | 21
  FAF1.mRNA, Day 37 | 0.93 [0.63 to 1.38] | 0.97 [0.79 to 1.73] | 0.97 [0.77 to 1.65] | 0.97 [0.73 to 1.54] | 1.07 [0.71 to 1.95]
  STAT1.mRNA, Day 0 | 0.92 [0.7 to 1.21] | 0.99 [0.79 to 1.3] | 0.97 [0.77 to 1.41] | 0.96 [0.6 to 1.25] | 0.95 [0.8 to 1.19]
  STAT1.mRNA, Day 1: number analyzed (Participants) | 18 | 23 | 27 | 22 | 21
  STAT1.mRNA, Day 1 | 2.31 [0.71 to 5.23] | 2.88 [0.24 to 6.32] | 1.31 [0.54 to 6.66] | 0.92 [0.66 to 1.36] | 0.95 [0.56 to 1.97]
  STAT1.mRNA, Day 14 | 1.02 [0.15 to 2.84] | 0.96 [0.18 to 1.93] | 0.98 [0.2 to 2.41] | 1.04 [0.74 to 5.74] | 0.96 [0.42 to 2.44]
  STAT1.mRNA, Day 30: number analyzed (Participants) | 18 | 23 | 28 | 19 | 21
  STAT1.mRNA, Day 30 | 0.96 [0.63 to 1.2] | 0.88 [0.6 to 1.17] | 0.96 [0.73 to 1.45] | 0.89 [0.6 to 1.22] | 0.96 [0.71 to 1.21]
  STAT1.mRNA, Day 31: number analyzed (Participants) | 18 | 23 | 28 | 19 | 21
  STAT1.mRNA, Day 31 | 4.95 [1.5 to 7.8] | 3.83 [1.61 to 7.2] | 3.13 [1.06 to 7.93] | 0.88 [0.26 to 1.29] | 0.96 [0.19 to 1.25]
  STAT1.mRNA, Day 33: number analyzed (Participants) | 18 | 22 | 28 | 19 | 21
  STAT1.mRNA, Day 33 | 2.03 [0.82 to 4.86] | 1.25 [0.49 to 4.19] | 1.12 [0.42 to 2.95] | 1.01 [0.21 to 1.55] | 1 [0.25 to 1.54]
  STAT1.mRNA, Day 37: number analyzed (Participants) | 18 | 22 | 28 | 17 | 21
  STAT1.mRNA, Day 37 | 0.87 [0.63 to 1.45] | 0.89 [0.35 to 1.45] | 0.86 [0.23 to 1.37] | 0.95 [0.16 to 1.43] | 1.02 [0.19 to 1.81]

44. Secondary Outcome: mRNA Levels as Measured by Quantitative Polymerase Chain Reaction (qPCR)
Description: The analysis of the mRNA levels of 14 target genes was performed using whole blood, in the first 140 subjects from the 2 subsets recruited at the Immune Health (IH) centre in La Louvière, Belgium, by microarray/ Polymerase Chain Reaction (PCR) array/ quantitative PCR. Among the target genes were Interferon Regulatory Factor 1 (IRF1), MX Dynamin-Like GTPase 1(MX1).
Time Frame: At Days 0, 1, 14, 30, 31, 33 and 37
Population: as for outcome 42
Measure: Median (Full Range); unit: copies
Arm/Group | GSK223192A 1 Group | GSK223192A 2 Group | GSK223192A 3 Group | Fendrix Group | Engerix-B Group
Number analyzed (Participants) | 18 | 23 | 28 | 22 | 21
copies
  IRF1.mRNA, Day 0 | 0.96 [0.61 to 1.53] | 0.99 [0.65 to 1.83] | 0.95 [0.65 to 1.42] | 1.03 [0.84 to 1.69] | 1 [0.87 to 1.25]
  IRF1.mRNA, Day 1: number analyzed (Participants) | 18 | 23 | 27 | 22 | 20
  IRF1.mRNA, Day 1 | 1.51 [0.8 to 2.98] | 1.59 [0.44 to 3.23] | 1.24 [0.54 to 2.81] | 1.08 [0.76 to 1.45] | 0.95 [0.7 to 1.34]
  IRF1.mRNA, Day 14: number analyzed (Participants) | 18 | 23 | 28 | 21 | 21
  IRF1.mRNA, Day 14 | 1.02 [0.25 to 1.79] | 1.01 [0.49 to 1.93] | 1.02 [0.4 to 1.87] | 1.14 [0.82 to 4.12] | 0.97 [0.6 to 2]
  IRF1.mRNA, Day 30: number analyzed (Participants) | 18 | 23 | 28 | 19 | 21
  IRF1.mRNA, Day 30 | 1 [0.59 to 1.82] | 0.93 [0.69 to 1.62] | 0.92 [0.71 to 1.45] | 0.96 [0.71 to 1.2] | 0.99 [0.65 to 1.67]
  IRF1.mRNA, Day 31: number analyzed (Participants) | 18 | 23 | 28 | 19 | 21
  IRF1.mRNA, Day 31 | 3.14 [1.12 to 8.06] | 2.63 [1.32 to 3.95] | 1.73 [0.8 to 5.63] | 1.05 [0.35 to 1.5] | 0.99 [0.45 to 1.47]
  IRF1.mRNA, Day 33: number analyzed (Participants) | 18 | 22 | 28 | 19 | 21
  IRF1.mRNA, Day 33 | 1.33 [0.78 to 2.63] | 1.03 [0.62 to 1.72] | 0.9 [0.54 to 1.6] | 1.11 [0.43 to 1.59] | 1.05 [0.52 to 1.62]
  IRF1.mRNA, Day 37: number analyzed (Participants) | 18 | 22 | 28 | 17 | 21
  IRF1.mRNA, Day 37 | 0.99 [0.42 to 2.24] | 0.93 [0.59 to 1.3] | 0.9 [0.35 to 1.63] | 0.97 [0.27 to 1.38] | 1 [0.54 to 1.78]
  MX1.mRNA, Day 0 | 1 [0.77 to 1.21] | 1.01 [0.77 to 1.38] | 0.98 [0.7 to 1.32] | 1.01 [0.82 to 2.02] | 0.98 [0.66 to 1.29]
  MX1.mRNA, Day 1: number analyzed (Participants) | 18 | 23 | 27 | 22 | 21
  MX1.mRNA, Day 1 | 1.61 [0.96 to 3.42] | 1.59 [0.14 to 3.29] | 1.18 [0.45 to 4.98] | 1.01 [0.48 to 1.4] | 0.9 [0.58 to 1.35]
  MX1.mRNA, Day 14 | 0.95 [0.05 to 8.35] | 1.03 [0.08 to 4.12] | 0.91 [0.06 to 5.32] | 1.11 [0.4 to 9.7] | 1.08 [0.26 to 3.54]
  MX1.mRNA, Day 30: number analyzed (Participants) | 18 | 23 | 28 | 19 | 21
  MX1.mRNA, Day 30 | 0.96 [0.41 to 1.46] | 0.92 [0.74 to 2.02] | 0.92 [0.69 to 1.51] | 0.96 [0.55 to 1.26] | 0.94 [0.58 to 1.5]
  MX1.mRNA, Day 31: number analyzed (Participants) | 18 | 23 | 28 | 19 | 21
  MX1.mRNA, Day 31 | 3.06 [0.69 to 6.38] | 2.19 [1.18 to 9.95] | 2.06 [0.84 to 6.64] | 0.96 [0.28 to 1.22] | 0.92 [0.17 to 1.69]
  MX1.mRNA, Day 33: number analyzed (Participants) | 18 | 22 | 27 | 19 | 21
  MX1.mRNA, Day 33 | 2.92 [0.6 to 8.49] | 1.83 [0.32 to 7.39] | 1.87 [0.38 to 5.45] | 1.07 [0.16 to 1.35] | 0.98 [0.12 to 1.54]
  MX1.mRNA, Day 37: number analyzed (Participants) | 18 | 22 | 28 | 17 | 21
  MX1.mRNA, Day 37 | 0.93 [0.63 to 5.86] | 0.9 [0.19 to 1.75] | 0.86 [0.1 to 1.74] | 1.07 [0.06 to 2.17] | 1.08 [0.08 to 4.66]

45. Secondary Outcome: Messenger Ribonucleic Acid (mRNA) Levels as Measured by Quantitative Polymerase Chain Reaction (qPCR)
Description: The analysis of the mRNA levels of 14 target genes was performed using whole blood, in the first 140 subjects from the 2 subsets recruited at the Immune Health (IH) centre in La Louvière, Belgium, by microarray/ Polymerase Chain Reaction (PCR) array/ quantitative PCR. Among the target genes were Interleukin-12A (IL-12A), Marker Of Proliferation Ki-67 (MKI67).
Time Frame: At Days 0, 1, 14, 30, 31, 33 and 37
Population: as for outcome 42
Measure: Median (Full Range); unit: copies
Arm/Group | GSK223192A 1 Group | GSK223192A 2 Group | GSK223192A 3 Group | Fendrix Group | Engerix-B Group
Number analyzed (Participants) | 18 | 23 | 28 | 22 | 21
copies
  IL-12A.mRNA, Day 0: number analyzed (Participants) | 18 | 23 | 28 | 21 | 21
  IL-12A.mRNA, Day 0 | 1.01 [0.53 to 2.3] | 0.97 [0.54 to 1.36] | 0.95 [0.53 to 1.88] | 0.9 [0.31 to 1.73] | 1.07 [0.55 to 1.69]
  IL-12A.mRNA, Day 1: number analyzed (Participants) | 18 | 23 | 27 | 21 | 20
  IL-12A.mRNA, Day 1 | 1.04 [0.5 to 2.68] | 1.01 [0.56 to 2.97] | 1.04 [0.45 to 2.23] | 0.94 [0.39 to 1.71] | 1.06 [0.44 to 2.56]
  IL-12A.mRNA, Day 14: number analyzed (Participants) | 18 | 23 | 28 | 21 | 21
  IL-12A.mRNA, Day 14 | 0.97 [0.6 to 1.73] | 0.97 [0.42 to 2.64] | 1.09 [0.36 to 2.06] | 0.77 [0.57 to 1.72] | 0.96 [0.5 to 2.1]
  IL-12A.mRNA, Day 30: number analyzed (Participants) | 18 | 23 | 28 | 18 | 21
  IL-12A.mRNA, Day 30 | 1.01 [0.5 to 1.61] | 1 [0.44 to 5.85] | 0.87 [0.46 to 1.8] | 1.1 [0.39 to 2.52] | 1.03 [0.38 to 1.76]
  IL-12A.mRNA, Day 31: number analyzed (Participants) | 18 | 22 | 28 | 19 | 21
  IL-12A.mRNA, Day 31 | 1.32 [0.68 to 3.55] | 1.2 [0.61 to 2.61] | 1.04 [0.47 to 2.35] | 0.9 [0.36 to 1.41] | 1.01 [0.43 to 2.22]
  IL-12A.mRNA, Day 33: number analyzed (Participants) | 18 | 21 | 28 | 19 | 21
  IL-12A.mRNA, Day 33 | 0.94 [0.61 to 2.92] | 0.85 [0.44 to 1.64] | 0.86 [0.41 to 1.78] | 0.89 [0.46 to 1.52] | 1.05 [0.37 to 2.72]
  IL-12A.mRNA, Day 37: number analyzed (Participants) | 18 | 22 | 27 | 17 | 21
  IL-12A.mRNA, Day 37 | 1.14 [0.56 to 1.73] | 1.08 [0.42 to 2.75] | 0.95 [0.47 to 2.45] | 1.09 [0.33 to 3.13] | 1.22 [0.61 to 1.78]
  MKI67.mRNA, Day 0: number analyzed (Participants) | 18 | 23 | 28 | 22 | 20
  MKI67.mRNA, Day 0 | 0.91 [0.23 to 1.63] | 0.89 [0.45 to 2.72] | 0.98 [0.45 to 1.74] | 0.83 [0.51 to 2.12] | 1.03 [0.61 to 2.51]
  MKI67.mRNA, Day 1: number analyzed (Participants) | 18 | 23 | 27 | 22 | 21
  MKI67.mRNA, Day 1 | 0.89 [0.33 to 1.7] | 0.9 [0.46 to 2.63] | 0.99 [0.55 to 1.48] | 0.94 [0.37 to 1.85] | 1.03 [0.48 to 1.79]
  MKI67.mRNA, Day 14: number analyzed (Participants) | 18 | 23 | 27 | 22 | 20
  MKI67.mRNA, Day 14 | 1.06 [0.57 to 2.83] | 1.14 [0.39 to 3.17] | 1.18 [0.32 to 2.74] | 0.99 [0.6 to 2.75] | 1.07 [0.4 to 3.71]
  MKI67.mRNA, Day 30: number analyzed (Participants) | 18 | 23 | 27 | 19 | 21
  MKI67.mRNA, Day 30 | 1 [0.56 to 1.61] | 0.92 [0.68 to 1.56] | 1.1 [0.48 to 1.77] | 0.98 [0.42 to 1.8] | 0.97 [0.5 to 1.7]
  MKI67.mRNA, Day 31: number analyzed (Participants) | 18 | 23 | 28 | 19 | 21
  MKI67.mRNA, Day 31 | 0.84 [0.45 to 1.57] | 0.83 [0.5 to 1.87] | 0.97 [0.42 to 2.44] | 0.95 [0.3 to 1.52] | 1.12 [0.52 to 4.01]
  MKI67.mRNA, Day 33: number analyzed (Participants) | 18 | 22 | 28 | 18 | 21
  MKI67.mRNA, Day 33 | 0.96 [0.44 to 2.13] | 1.02 [0.5 to 2.72] | 1.14 [0.38 to 2.52] | 0.89 [0.28 to 1.42] | 1.03 [0.55 to 8.12]
  MKI67.mRNA, Day 37: number analyzed (Participants) | 18 | 22 | 28 | 17 | 21
  MKI67.mRNA, Day 37 | 1.52 [0.38 to 3.28] | 1.56 [0.58 to 4.01] | 1.38 [0.37 to 3.94] | 1.06 [0.58 to 2.01] | 1.08 [0.35 to 1.76]

46. Secondary Outcome: Levels of mRNA as Measured by qPCR
Description: The analysis of the mRNA levels of 14 target genes was performed using whole blood, in the first 140 subjects from the 2 subsets recruited at the Immune Health (IH) centre in La Louvière, Belgium, by microarray/ Polymerase Chain Reaction (PCR) array/ quantitative PCR. Among the target genes were Chemokine Ligand 10 (CXCL10), Interleukin-1B (IL-1B).
Time Frame: At Days 0, 1, 14, 30, 31, 33 and 37
Population: as for outcome 42
Measure: Median (Full Range); unit: copies
Arm/Group | GSK223192A 1 Group | GSK223192A 2 Group | GSK223192A 3 Group | Fendrix Group | Engerix-B Group
Number analyzed (Participants) | 18 | 23 | 28 | 22 | 21
copies
  IL-1B.mRNA, Day 0 | 1.04 [0.41 to 1.54] | 1.12 [0.6 to 2.33] | 1.02 [0.51 to 2.24] | 1.04 [0.59 to 2.21] | 0.96 [0.53 to 1.35]
  IL-1B.mRNA, Day 1: number analyzed (Participants) | 18 | 23 | 27 | 22 | 21
  IL-1B.mRNA, Day 1 | 1.56 [0.56 to 2.8] | 1.31 [0.67 to 2.1] | 1.21 [0.55 to 2.58] | 1.24 [0.82 to 2.68] | 0.92 [0.4 to 1.48]
  IL-1B.mRNA, Day 14 | 0.94 [0.24 to 1.95] | 0.93 [0.43 to 3.61] | 0.97 [0.34 to 2.24] | 1.23 [0.72 to 3.1] | 1 [0.52 to 1.78]
  IL-1B.mRNA, Day 30: number analyzed (Participants) | 18 | 23 | 28 | 19 | 21
  IL-1B.mRNA, Day 30 | 1.2 [0.43 to 2.08] | 0.98 [0.55 to 1.51] | 1.04 [0.68 to 1.51] | 0.94 [0.58 to 1.48] | 1.05 [0.57 to 1.86]
  IL-1B.mRNA, Day 31: number analyzed (Participants) | 18 | 23 | 28 | 19 | 21
  IL-1B.mRNA, Day 31 | 2.02 [1.38 to 5.6] | 1.47 [0.78 to 2.2] | 1.23 [0.64 to 2.87] | 1.14 [0.47 to 1.92] | 1.06 [0.44 to 1.54]
  IL-1B.mRNA, Day 33: number analyzed (Participants) | 18 | 22 | 28 | 19 | 21
  IL-1B.mRNA, Day 33 | 1.31 [0.81 to 6.05] | 1.07 [0.54 to 1.76] | 0.93 [0.58 to 1.59] | 1.02 [0.72 to 1.95] | 1.01 [0.49 to 2.16]
  IL-1B.mRNA, Day 37: number analyzed (Participants) | 18 | 22 | 28 | 17 | 21
  IL-1B.mRNA, Day 37 | 0.97 [0.38 to 2.6] | 0.87 [0.36 to 1.83] | 0.85 [0.29 to 1.8] | 0.83 [0.35 to 1.52] | 1.01 [0.45 to 2.01]
  CXCL10.mRNA, Day 0: number analyzed (Participants) | 17 | 23 | 28 | 22 | 21
  CXCL10.mRNA, Day 0 | 0.92 [0.55 to 1.36] | 0.97 [0.52 to 1.79] | 0.92 [0.37 to 1.97] | 0.97 [0.31 to 1.73] | 1.07 [0.55 to 1.99]
  CXCL10.mRNA, Day 1: number analyzed (Participants) | 18 | 23 | 27 | 22 | 21
  CXCL10.mRNA, Day 1 | 0.96 [0.28 to 4.43] | 1.14 [0.27 to 9.62] | 1.06 [0.12 to 12.97] | 0.97 [0.39 to 1.91] | 0.96 [0.44 to 2.56]
  CXCL10.mRNA, Day 14 | 0.88 [0.16 to 1.99] | 0.95 [0.13 to 2.64] | 1.06 [0.06 to 2.92] | 0.9 [0.39 to 48.74] | 0.97 [0.6 to 3.39]
  CXCL10.mRNA, Day 30: number analyzed (Participants) | 18 | 23 | 28 | 19 | 21
  CXCL10.mRNA, Day 30 | 1.08 [0.64 to 2.04] | 1.03 [0.61 to 5.85] | 0.88 [0.46 to 2.62] | 1.1 [0.33 to 1.81] | 0.92 [0.43 to 1.76]
  CXCL10.mRNA, Day 31: number analyzed (Participants) | 18 | 23 | 28 | 19 | 21
  CXCL10.mRNA, Day 31 | 6.25 [0.68 to 32.91] | 2.93 [0.75 to 16.09] | 1.59 [0.47 to 16.85] | 0.95 [0.04 to 1.44] | 1.18 [0.29 to 1.54]
  CXCL10.mRNA, Day 33: number analyzed (Participants) | 18 | 22 | 28 | 19 | 21
  CXCL10.mRNA, Day 33 | 1.35 [0.61 to 5.9] | 1.06 [0.6 to 2.73] | 0.86 [0.38 to 2.6] | 1.13 [0.02 to 1.94] | 1.05 [0.31 to 2.48]
  CXCL10.mRNA, Day 37: number analyzed (Participants) | 18 | 22 | 28 | 17 | 21
  CXCL10.mRNA, Day 37 | 0.91 [0.51 to 5.33] | 1.02 [0.53 to 2.75] | 0.94 [0.35 to 2.45] | 1.03 [0.02 to 2.06] | 1.09 [0.51 to 2.37]

47. Secondary Outcome: Levels of Messenger Ribonucleic Acid (mRNA) as Measured by qPCR
Description: The analysis of the mRNA levels of 14 target genes was performed using whole blood, in the first 140 subjects from the 2 subsets recruited at the Immune Health (IH) centre in La Louvière, Belgium, by microarray/ Polymerase Chain Reaction (PCR) array/ quantitative PCR. Among the target genes were Prostaglandin-Endoperoxide Synthase 2 (PTGS2), Dual Specificity Phosphatase 1 (DUSP1).
Time Frame: At Days 0, 1, 14, 30, 31, 33 and 37
Population: as for outcome 42
Measure: Median (Full Range); unit: copies
Arm/Group | GSK223192A 1 Group | GSK223192A 2 Group | GSK223192A 3 Group | Fendrix Group | Engerix-B Group
Number analyzed (Participants) | 18 | 23 | 28 | 22 | 21
copies
  PTGS2.mRNA, Day 0 | 1.06 [0.63 to 1.59] | 1.01 [0.67 to 1.66] | 1.07 [0.64 to 1.73] | 1.06 [0.77 to 1.76] | 1.04 [0.63 to 1.28]
  PTGS2.mRNA, Day 1: number analyzed (Participants) | 18 | 23 | 27 | 22 | 21
  PTGS2.mRNA, Day 1 | 1.25 [0.74 to 1.74] | 1.15 [0.69 to 2.55] | 1.16 [0.77 to 2.13] | 1.05 [0.73 to 1.47] | 0.95 [0.71 to 1.32]
  PTGS2.mRNA, Day 14 | 1.07 [0.65 to 1.69] | 0.92 [0.7 to 1.66] | 1.01 [0.4 to 2.08] | 1.06 [0.67 to 2.4] | 1.13 [0.49 to 1.29]
  PTGS2.mRNA, Day 30: number analyzed (Participants) | 18 | 23 | 28 | 19 | 21
  PTGS2.mRNA, Day 30 | 1.14 [0.58 to 1.5] | 0.94 [0.67 to 1.38] | 1.02 [0.69 to 1.51] | 0.98 [0.58 to 1.22] | 1.09 [0.67 to 1.56]
  PTGS2.mRNA, Day 31: number analyzed (Participants) | 18 | 23 | 28 | 19 | 21
  PTGS2.mRNA, Day 31 | 1.66 [1.17 to 2.83] | 1.33 [0.97 to 2.4] | 1.11 [0.74 to 1.99] | 1.08 [0.72 to 1.63] | 1.04 [0.63 to 1.43]
  PTGS2.mRNA, Day 33: number analyzed (Participants) | 18 | 22 | 28 | 19 | 21
  PTGS2.mRNA, Day 33 | 0.97 [0.66 to 3.53] | 0.85 [0.52 to 1.22] | 0.82 [0.57 to 1.64] | 1.07 [0.77 to 2.73] | 1.01 [0.6 to 2.03]
  PTGS2.mRNA, Day 37: number analyzed (Participants) | 18 | 22 | 28 | 17 | 21
  PTGS2.mRNA, Day 37 | 0.87 [0.33 to 3.76] | 0.94 [0.59 to 1.65] | 0.91 [0.57 to 2.15] | 0.96 [0.62 to 1.35] | 1.15 [0.55 to 1.68]
  DUSP1.mRNA, Day 0 | 0.84 [0.45 to 1.52] | 0.96 [0.52 to 1.8] | 1.02 [0.58 to 2.27] | 0.89 [0.55 to 1.96] | 0.9 [0.5 to 1.27]
  DUSP1.mRNA, Day 1: number analyzed (Participants) | 18 | 23 | 27 | 22 | 21
  DUSP1.mRNA, Day 1 | 1.09 [0.67 to 1.95] | 1.1 [0.52 to 2.03] | 1.12 [0.68 to 2.46] | 1.14 [0.6 to 1.99] | 0.85 [0.53 to 1.81]
  DUSP1.mRNA, Day 14 | 0.95 [0.6 to 1.81] | 0.85 [0.63 to 1.91] | 1.2 [0.32 to 2.45] | 1.07 [0.81 to 1.86] | 1 [0.45 to 1.55]
  DUSP1.mRNA, Day 30: number analyzed (Participants) | 18 | 23 | 28 | 19 | 21
  DUSP1.mRNA, Day 30 | 1.03 [0.44 to 2.14] | 0.81 [0.48 to 1.46] | 0.92 [0.55 to 2.04] | 0.86 [0.63 to 1.28] | 0.96 [0.53 to 1.8]
  DUSP1.mRNA, Day 31: number analyzed (Participants) | 18 | 23 | 28 | 19 | 21
  DUSP1.mRNA, Day 31 | 1.34 [0.8 to 3.56] | 1.3 [0.64 to 1.95] | 1.05 [0.63 to 1.67] | 1.31 [0.76 to 1.97] | 0.94 [0.57 to 1.85]
  DUSP1.mRNA, Day 33: number analyzed (Participants) | 18 | 22 | 28 | 19 | 21
  DUSP1.mRNA, Day 33 | 0.97 [0.58 to 5.29] | 0.84 [0.43 to 1.42] | 0.81 [0.52 to 1.56] | 1.18 [0.78 to 2.69] | 0.99 [0.42 to 1.91]
  DUSP1.mRNA, Day 37: number analyzed (Participants) | 18 | 22 | 28 | 17 | 21
  DUSP1.mRNA, Day 37 | 0.91 [0.27 to 4.05] | 0.94 [0.34 to 1.57] | 0.95 [0.51 to 1.61] | 0.94 [0.68 to 1.53] | 1 [0.45 to 2.3]

48. Secondary Outcome: Levels of mRNA as Measured by Quantitative Polymerase Chain Reaction (qPCR)
Description: The analysis of the mRNA levels of 14 target genes was performed using whole blood, in the first 140 subjects from the 2 subsets recruited at the Immune Health (IH) centre in La Louvière, Belgium, by microarray/ Polymerase Chain Reaction (PCR) array/ quantitative PCR. Among the target genes were Nuclear Factor Of Activated T-Cells, Cytoplasmic, Calcineurin-Dependent 2 (NFATC2) and Interferon-gamma (IFN-γ).
Time Frame: At Days 0, 1, 14, 30, 31, 33 and 37
Population: as for outcome 42
Measure: Median (Full Range); unit: copies
Arm/Group | GSK223192A 1 Group | GSK223192A 2 Group | GSK223192A 3 Group | Fendrix Group | Engerix-B Group
Number analyzed (Participants) | 18 | 23 | 28 | 22 | 21
copies
  NFATC2.mRNA, Day 0 | 0.98 [0.52 to 1.25] | 0.94 [0.64 to 1.64] | 1.03 [0.74 to 1.91] | 0.93 [0.51 to 1.56] | 1.11 [0.64 to 1.5]
  NFATC2.mRNA, Day 1: number analyzed (Participants) | 18 | 23 | 27 | 22 | 21
  NFATC2.mRNA, Day 1 | 0.66 [0.48 to 1.06] | 0.73 [0.43 to 2.55] | 0.83 [0.47 to 1.56] | 0.83 [0.6 to 1.23] | 1.04 [0.73 to 1.57]
  NFATC2.mRNA, Day 14 | 1 [0.48 to 1.69] | 0.98 [0.42 to 2.12] | 1.09 [0.61 to 1.78] | 0.89 [0.53 to 1.39] | 1.1 [0.64 to 1.59]
  NFATC2.mRNA, Day 30: number analyzed (Participants) | 18 | 23 | 28 | 19 | 21
  NFATC2.mRNA, Day 30 | 0.92 [0.7 to 1.64] | 0.99 [0.72 to 1.37] | 1 [0.78 to 1.57] | 1.05 [0.82 to 1.5] | 1.08 [0.79 to 1.44]
  NFATC2.mRNA, Day 31: number analyzed (Participants) | 18 | 23 | 28 | 19 | 21
  NFATC2.mRNA, Day 31 | 0.46 [0.32 to 1.06] | 0.58 [0.34 to 1.15] | 0.78 [0.33 to 1.46] | 0.87 [0.69 to 1.78] | 1.1 [0.83 to 1.33]
  NFATC2.mRNA, Day 33: number analyzed (Participants) | 18 | 23 | 28 | 19 | 21
  NFATC2.mRNA, Day 33 | 0.79 [0.59 to 1.36] | 0.9 [0.56 to 1.79] | 0.87 [0.63 to 1.55] | 1.05 [0.63 to 1.43] | 1.05 [0.75 to 1.62]
  NFATC2.mRNA, Day 37: number analyzed (Participants) | 18 | 22 | 28 | 17 | 21
  NFATC2.mRNA, Day 37 | 1.03 [0.74 to 1.22] | 1.03 [0.66 to 1.59] | 0.98 [0.72 to 1.99] | 1.16 [0.83 to 1.56] | 1.11 [0.69 to 1.91]
  IFN-γ.mRNA, Day 0 | 0.97 [0.55 to 1.36] | 0.97 [0.54 to 1.79] | 0.94 [0.59 to 1.97] | 0.97 [0.31 to 1.73] | 1.07 [0.55 to 1.99]
  IFN-γ.mRNA, Day 1: number analyzed (Participants) | 18 | 23 | 27 | 22 | 21
  IFN-γ.mRNA, Day 1 | 0.89 [0.5 to 1.74] | 1.01 [0.6 to 2.97] | 1.03 [0.45 to 1.94] | 0.97 [0.39 to 1.91] | 0.96 [0.44 to 2.56]
  IFN-γ.mRNA, Day 14 | 0.88 [0.55 to 1.99] | 0.97 [0.44 to 2.64] | 1.11 [0.48 to 2.08] | 0.82 [0.39 to 1.72] | 0.96 [0.6 to 2.1]
  IFN-γ.mRNA, Day 30: number analyzed (Participants) | 18 | 23 | 28 | 19 | 21
  IFN-γ.mRNA, Day 30 | 1.08 [0.64 to 2.04] | 1.03 [0.61 to 5.85] | 0.88 [0.46 to 3.19] | 1.13 [0.47 to 1.81] | 0.92 [0.48 to 1.76]
  IFN-γ.mRNA, Day 31: number analyzed (Participants) | 18 | 23 | 28 | 19 | 21
  IFN-γ.mRNA, Day 31 | 0.91 [0.61 to 2.46] | 0.86 [0.44 to 2.61] | 0.89 [0.4 to 1.53] | 0.96 [0.41 to 1.89] | 1.18 [0.45 to 1.54]
  IFN-γ.mRNA, Day 33: number analyzed (Participants) | 18 | 22 | 28 | 19 | 21
  IFN-γ.mRNA, Day 33 | 0.9 [0.61 to 4.25] | 0.92 [0.6 to 2.04] | 0.83 [0.38 to 2.6] | 1.13 [0.47 to 1.94] | 1.05 [0.53 to 2.48]
  IFN-γ.mRNA, Day 37: number analyzed (Participants) | 18 | 22 | 28 | 17 | 21
  IFN-γ.mRNA, Day 37 | 0.89 [0.51 to 5.33] | 1.02 [0.53 to 2.75] | 0.94 [0.47 to 2.45] | 1.09 [0.6 to 2.06] | 1.09 [0.71 to 2.37]

ADVERSE EVENTS:
Time Frame: Solicited symptoms post primary/booster vaccination: 14/7-day follow-up period after vaccination; Unsolicited adverse events (AEs): 31-day follow-up period after vaccination; Serious AEs: From Day 0 to Day 360 (non-Subsets 1 & 2)/390 (Subsets 1 & 2)
Description: Solicited symptoms data below result from analyses on the Total Vaccinated cohort, inclusive of all vaccinated subjects, and on the Booster Total Vaccinated cohort, inclusive of all vaccinated subjects from Subsets 1and 2 vaccinated with HBsAg antigens at Day 360, performed solely on subjects from whose symptom sheets were collected.
Arm/Group | GSK223192A 1 Group | GSK223192A 2 Group | GSK223192A 3 Group | Fendrix Group | Engerix-B Group
All-Cause Mortality (participants affected / at risk) | 0/143 | 0/142 | 0/141 | 0/145 | 0/142
Serious Adverse Events (participants affected / at risk) | 7/143 | 4/142 | 10/141 | 7/145 | 7/142
Other Adverse Events (participants affected / at risk) | 137/143 | 135/142 | 131/141 | 141/145 | 114/142
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GSK223192A 1 Group (N=143) | GSK223192A 2 Group (N=142) | GSK223192A 3 Group (N=141) | Fendrix Group (N=145) | Engerix-B Group (N=142)
Depression (Psychiatric disorders) | 0 | 0 | 0 | 2 | 1
Appendicitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0
Abdominal injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Acute stress disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Anxiety disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Chondropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Cluster headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Epicondylitis (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Ovarian cyst torsion (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Paranasal cyst (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Post-traumatic stress disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Somatisation disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Varicocele (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | GSK223192A 1 Group (N=143) | GSK223192A 2 Group (N=142) | GSK223192A 3 Group (N=141) | Fendrix Group (N=145) | Engerix-B Group (N=142)
Nasopharyngitis (Infections and infestations) | 11 | 8 | 7 | 4 | 7 — Unsolicited AE reported post vaccination with the GSK223192A, Fendrix™ or Engerix-B™ vaccine
Nasopharyngitis (Infections and infestations) | 3/59 | 0/56 | 1/56 | 0/56 | 0/54 — Unsolicited AE reported post vaccination with HBsAg antigens.
Headache (Nervous system disorders) | 3 | 2 | 4 | 3 | 8 — Unsolicited AE reported post vaccination with the GSK223192A, Fendrix™ or Engerix-B™ vaccine.
Pain (General disorders) | 134/142 | 129/140 | 123/138 | 128/143 | 70/139 — Solicited symptom reported post vaccination with the GSK223192A, Fendrix™ or Engerix-B™ vaccine.
Redness (General disorders) | 71/142 | 39/140 | 35/138 | 53/143 | 23/139 — Solicited symptom reported post vaccination with the GSK223192A, Fendrix™ or Engerix-B™ vaccine.
Swelling (General disorders) | 46/142 | 36/140 | 34/138 | 43/143 | 16/139 — Solicited symptom reported post vaccination with the GSK223192A, Fendrix™ or Engerix-B™ vaccine.
Pain (General disorders) | 19/59 | 19/56 | 13/56 | 16/56 | 10/54 — Solicited symptom reported post vaccination with HBsAg antigens.
Redness (General disorders) | 6/59 | 3/56 | 8/56 | 6/56 | 2/54 — Solicited symptom reported post vaccination with HBsAg antigens.
Swelling (General disorders) | 3/59 | 4/56 | 2/56 | 5/56 | 1/54 — Solicited symptom reported post vaccination with HBsAg antigens.
Fatigue (General disorders) | 91/142 | 76/140 | 67/138 | 70/144 | 62/139 — Solicited symptom reported post vaccination with the GSK223192A, Fendrix™ or Engerix-B™ vaccine.
Fever (Oral temperature >= 37.5°C) (General disorders) | 45/142 | 23/140 | 24/138 | 12/144 | 17/139 — Solicited symptom reported post vaccination with the GSK223192A, Fendrix™ or Engerix-B™ vaccine.
Gastrointestinal symptoms (General disorders) | 30/142 | 27/140 | 29/138 | 36/144 | 35/139 — Solicited symptom reported post vaccination with the GSK223192A, Fendrix™ or Engerix-B™ vaccine.
Headache (General disorders) | 90/142 | 67/140 | 66/138 | 62/144 | 59/139 — Solicited symptom reported post vaccination with the GSK223192A, Fendrix™ or Engerix-B™ vaccine.
Malaise (General disorders) | 60/142 | 44/140 | 39/138 | 35/144 | 28/139 — Solicited symptom reported post vaccination with the GSK223192A, Fendrix™ or Engerix-B™ vaccine.
Myalgia (General disorders) | 85/142 | 57/140 | 55/138 | 58/144 | 34/139 — Solicited symptom reported post vaccination with the GSK223192A, Fendrix™ or Engerix-B™ vaccine.
Fatigue (General disorders) | 15/59 | 14/56 | 7/56 | 15/56 | 12/54 — Solicited symptom reported post vaccination with HBsAg antigens.
Fever (Oral temperature > = 37.5°C) (General disorders) | 3/59 | 1/56 | 0/56 | 3/56 | 1/54 — Solicited symptom reported post vaccination with HBsAg antigens.
Gastrointestinal symptoms (General disorders) | 4/59 | 5/56 | 4/56 | 3/56 | 5/54 — Solicited symptom reported post vaccination with HBsAg antigens.
Headache (General disorders) | 15/59 | 7/56 | 7/56 | 8/56 | 14/54 — Solicited symptom reported post vaccination with HBsAg antigens.
Malaise (General disorders) | 6/59 | 5/56 | 2/56 | 4/56 | 4/54 — Solicited symptom reported post vaccination with HBsAg antigens.
Myalgia (General disorders) | 4/59 | 3/56 | 2/56 | 5/56 | 1/54 — Solicited symptom reported post vaccination with HBsAg antigens.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.